CLINICAL TRIAL: NCT04955626
Title: A PHASE 3 MASTER PROTOCOL TO EVALUATE ADDITIONAL DOSE(S) OF BNT162B2 IN HEALTHY INDIVIDUALS PREVIOUSLY VACCINATED WITH BNT162B2
Brief Title: To Evaluate the Safety, Tolerability, Efficacy and Immunogenicity of BNT162b2 Boosting Strategies Against COVID-19 in Participants ≥12 Years of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4591031; 2021-005197-25 (EudraCT Number)
Record Dates: First submitted 2021-06-09; First posted 2021-07-09 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: COVID-19; Coronavirus; Vaccine; SARS-CoV-2; RNA Vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10 µg dose (Experimental): 1 dose
  Interventions: Biological: BNT162b2
- Placebo (Placebo Comparator): 1 dose
  Interventions: Other: Placebo
- 30 µg dose (Experimental): 1 dose
  Interventions: Biological: BNT162b2; Biological: BNT162b2 OMI; Biological: Combination BNT162b2 and BNT162b2 OMI; Biological: Combination (Bivalent) BNT162b2 and BNT162b2 OMI
- 60 µg dose (Experimental): 1 dose
  Interventions: Biological: BNT162b2; Biological: BNT162b2 OMI; Biological: Combination BNT162b2 and BNT162b2 OMI; Biological: Combination (Bivalent) BNT162b2 and BNT162b2 OMI

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular Injection
  Arms: 10 µg dose; 30 µg dose; 60 µg dose
Other: Placebo — Intramuscular Injection
  Arms: Placebo
Biological: BNT162b2 OMI — Intramuscular Injection
  Arms: 30 µg dose; 60 µg dose
Biological: Combination BNT162b2 and BNT162b2 OMI — 30-µg (15-µg each) or 60-µg (30-µg each)
  Site prepared dosing suspension from 1 vial each of diluted BNT162b2 and BNT162b2 OMI
  Intramuscular Injection
  Arms: 30 µg dose; 60 µg dose
Biological: Combination (Bivalent) BNT162b2 and BNT162b2 OMI — 30-µg (15-µg each) or 60-µg (30-µg each)
  Preformulated bivalent mixture (no dilution required) presented in a single vial
  Intramuscular Injection
  Arms: 30 µg dose; 60 µg dose

SUMMARY:
Substudy A: The study will evaluate the safety, tolerability, and efficacy of a booster dose of BNT162b2 when administered to participants having previously received 2 doses of BNT162b2 at least 6 months prior to randomization.

The study is designed to describe vaccine efficacy of a booster dose of BNT162b2 over time against COVID-19

* At a dose of 30µg (as studied in the Phase 2/3 study C4591001)
* In healthy adults 16 years of age and older
* The duration of the study for each participant will be up to approximately 12 months.
* The study will be conducted in the United States, Brazil and South Africa

Substudy B: The study will assess the safety and tolerability of a single dose of BNT162b2 as compared to placebo control, through the potential analysis of serum troponin levels, in participants ≥12 and ≤30 years of age who have received 2 or 3 prior doses of BNT162b2 (30-µg doses) with their last dose at least 4 months (120 days) prior to randomization.

* Blood samples will be collected for troponin testing
* The duration of the study for each participant will be up to approximately 2 months.
* The study will be conducted in the United States, Germany, Poland and South Africa

Substudy C: The study will assess the safety, tolerability, and immunogenicity of a booster (third) dose of BNT162b2 at doses of 10 µg or 30 µg in participants who have completed a 2-dose primary series of BNT162b2 (30 µg doses) at least 5 months (150 days) prior to randomization.

* In healthy adults 12 years of age and older
* The duration of the study for each participant will be up to approximately 12 months.
* The study will be conducted in the United States, Germany and South Africa

Substudy D: The study will assess the safety, tolerability, and immunogenicity of a 2-dose primary series of BNT162b2 OMI, and as a booster (third, fourth or fifth) dose

* Participants in Cohort 1 will have completed a 2-dose primary series of BNT162b2 (30-µg doses), with their last dose 90 to 240 days prior to enrolment
* Participants in Cohort 2 will be enrolled from Study C4591001 and C4591031 Substudy A and will have completed a 2-dose primary series and received a single booster (third) dose of BNT162b2, with their last dose 90 to 180 days prior to randomization
* Participants in Cohort 3 who are COVID-19 vaccine-naïve and have not experienced COVID-19 will be enrolled to receive 2 doses (primary series) of BNT162b2 OMI, 3 weeks apart, with a dose of BNT162b2 approximately 5 months (150 days) later. If participants do not consent to receive BNT162b2 as a third dose, they will not receive a third dose. No participants should receive BNT162b2 OMI as a third dose.

  * In healthy adults 18 to 55 years of age
  * The duration of the study for each participant will be up to approximately 12 months.
  * The study will be conducted in the United States and South Africa

Substudy E: This study will assess the safety, tolerability, and immunogenicity of high-dose BNT162b2 (60 µg), high-dose BNT162b2 OMI (60 µg), and a high-dose combination of BNT162b2 and BNT162b2 OMI at 60 µg (30 µg each), given as a single dose

* In healthy adults 18 years of age and older who have received 3 prior doses of BNT162b2 (30 µg) with the most recent dose being 5 to 12 months (150 to 360 days) prior to randomization
* The duration of the study for each participant will be approximately 6 months.
* The study will be conducted in the United States

Substudy F: This study will assess the safety, tolerability, and immunogenicity of high-dose BNT162b2 (60 µg), high-dose BNT162b2 OMI (60 µg), and a high-dose combination of BNT162b2 and BNT162b2 OMI at 60 µg (30 µg each), given as a single dose.

* In healthy adults 60 years of age and older who have received 3 prior doses of BNT162b2 (30 µg) with the most recent dose being ≥4 months prior to randomization
* The duration of the study for each participant will be approximately 6 months.
* The study will be conducted in Israel

ELIGIBILITY:
Substudy A

Inclusion Criteria:

* Male or female participants ≥16 years of age at Visit 1 (Day 1) who participated in C4591001.
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving signed informed consent.
* Participants who have received 2 prior doses of 30 µg BNT162b2 19-42 days apart, with the second dose being at least 175 days before Visit 1 (Day 1).

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before study intervention administration, or planned receipt throughout the study.
* Prior receipt of any COVID-19 vaccine other than BNT162b2.
* Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Receipt of medications intended to prevent COVID-19.
* Prior receipt of more than 2 doses of BNT162b2 30 µg.
* Participation in other studies involving study intervention within 28 days prior to study entry, other than C4591001, and/or within 28 days of confirmed receipt of BNT162b2 within the study.

Substudy B

Inclusion Criteria:

* Male or female participants 12 to 30 years of age, inclusive, who have received 2 prior doses of 30 µg BNT162b2 19 to 60 days apart, with the second dose being at least at least 4 months (120 days) before Visit 1 (Day 1)
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behaviour or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before study intervention administration, or planned receipt throughout the study.
* Prior receipt of any COVID-19 vaccine other than BNT162b2.
* Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Receipt of medications intended to prevent COVID-19.
* Prior receipt of more than 3 doses of BNT162b2 30 µg.
* Participation in other studies involving study intervention within 28 days prior to study entry through and including 28 days after the last dose of study intervention, with the exception of non-Pfizer interventional studies for prevention of COVID-19, which are prohibited throughout study participation.

Substudy C

Inclusion Criteria:

* Male or female participants ≥12 years of age, inclusive, who have received 2 prior doses of 30 µg BNT162b2 19 to 60 days apart, with the second dose being at least 150 days before Visit 301 (Day 1)
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behaviour or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before study intervention administration, or planned receipt throughout the study.
* Prior receipt of any COVID-19 vaccine other than BNT162b2.
* Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Receipt of medications intended to prevent COVID-19.
* Prior receipt of more than 2 doses of BNT162b2 30 µg.
* Participation in other studies involving study intervention within 28 days prior to study entry through and including 28 days after the last dose of study intervention, with the exception of non-Pfizer interventional studies for prevention of COVID-19, which are prohibited throughout study participation.

Substudy D

Inclusion Criteria:

* Male or female participants 18 to 55 years of age inclusive
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Cohort 2: Participants who provided a serum sample at Visit 3 in Study C4591001, with Visit 3 occurring within the protocol-specified window.
* Capable of giving signed informed consent
* Cohort 1: Participants who have received 2 prior doses of 30 µg BNT162b2, with the second dose being 90 to 240 days before Visit 401 (Day 1) or Cohort 2: Participants who have received 3 prior doses of 30 µg BNT162b2, with the third dose being 90 to 180 days before Visit 401 (Day 1).

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before study intervention administration, or planned receipt throughout the study.
* Cohorts 1 and 2: prior receipt of any COVID-19 vaccine other than BNT162b2.
* Cohort 3 only: prior receipt of any COVID-19 vaccine.
* Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Receipt of medications intended to prevent COVID 19.
* Participation in other studies involving study intervention within 28 days prior to study entry through and including 28 days after the last dose of study intervention, with the exception of non-Pfizer interventional studies for prevention of COVID-19, which are prohibited throughout study participation.

Substudy E

Inclusion Criteria:

* Groups 1-6: Male or female participants >55 years of age
* Groups 7-9: Male or female participants 18 to 55 years of age
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving signed informed consent.
* Participants who have received 3 prior doses of 30 µg BNT162b2, with the third dose being 5 to 12 months (150 to 360 days) before Visit 601 (Day 1).
* Groups 7 to 9 (sentinel participants): Screening troponin levels must be within normal range prior to randomization.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before study intervention administration, or planned receipt throughout the study.
* Prior receipt of any COVID-19 vaccine other than BNT162b2.
* Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Receipt of medications intended to prevent COVID-19.
* Participation in other studies involving study intervention within 28 days prior to study entry through and including 28 days after the last dose of study intervention, with the exception of non-Pfizer interventional studies for prevention of COVID-19, which are prohibited throughout study participation.

Substudy F

Inclusion Criteria:

* Male or female participants ≥60 years of age
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving signed informed consent.
* Participants who have received 3 prior doses of 30 µg BNT162b2, with the third dose being ≥4 months before Visit 701 (Day 1).

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before study intervention administration, or planned receipt throughout the study.
* Prior receipt of any COVID-19 vaccine other than BNT162b2.
* Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Receipt of medications intended to prevent COVID-19.
* Participation in other studies involving study intervention within 28 days prior to study entry through and including 28 days after the last dose of study intervention, with the exception of non-Pfizer interventional studies for prevention of COVID-19, which are prohibited throughout study participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16372 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (153):
- United States (138):
  - North Alabama Research Center, Athens, Alabama
  - Accel Research Sites - Birmingham Clinical Research Unit, Birmingham, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - AMR Clinical, Mobile, Alabama
  - Johns Hopkins Center for American Indian Health, Chinle, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Johns Hopkins Center for American Indian Health, Whiteriver, Arizona
  - Whiteriver Indian Hospital- Garrett Building, Whiteriver, Arizona
  - Whiteriver Indian Hospital, Whiteriver, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permenente Medical Center Infectious Disease, Los Angeles, California
  - Velocity Clinical Research, Los Angeles, Los Angeles, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Kaiser Permanente Oakland, Oakland, California
  - Paradigm Clinical Research Centers, Inc, Redding, California
  - UC Davis Medical Center, Sacramento, California
  - California Research Foundation, San Diego, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Bayview Research Group, LLC, Valley Village, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Clinical Research Consulting, Milford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - IACT Health, Columbus, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - University of Iowa, Iowa City, Iowa
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - AMR Clinical, Newton, Kansas
  - AMR Clinical, Wichita, Kansas
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Michigan Center of Medical Research (MICHMER), Farmington Hills, Michigan
  - Velocity Clinical Research, Covington, Gulfport, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Bozeman Health Deaconess Hospital d/b/a Bozeman Health Clinical Research, Bozeman, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Methodist Physicians Clinic/CCT Research, Fremont, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Wake Research - Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Gallup Indian Medical Center, Gallup, New Mexico
  - Johns Hopkins Center for American Indian Health, Gallup, New Mexico
  - Johns Hopkins Center for American Indian Health, Shiprock, New Mexico
  - Northern Navajo Medical Center, Shiprock, New Mexico
  - Meridian Clinical Research LLC, Binghamton, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - University of Rochester Medical Center- Kari Steinmetz, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Velocity Clinical Research, Vestal, Vestal, New York
  - Accellacare, Cary, North Carolina
  - Accellacare, Charlotte, North Carolina
  - Duke University - Main Hospital and Clinics, Durham, North Carolina
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - Accellacare, Hickory, North Carolina
  - Accellacare, Raleigh, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Accellacare - Salisbury, Salisbury, North Carolina
  - Accellacare (formerly PMG Research of Wilmington, LLC), Wilmington, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Accellacare, Winston-Salem, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Meridian Clinical Research, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - VA Northeast Ohio Healthcare System, Cleveland, Ohio
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - PriMED Clinical Research, Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Lehigh Valley Health Network/Network Office of Research and Innovation, Allentown, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Main Street Physician's Care, Little River, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Alliance for Multispecialty Research - Weisgarber Medical Park, Knoxville, Tennessee
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Trinity Clinical Research, Tullahoma, Tennessee
  - Benchmark Research, Austin, Texas
  - Innovo Research - Austin Regional Clinic, Austin, Texas
  - Tekton Research, Inc, Austin, Texas
  - North Texas Infectious Diseases Consultants, P.A, Dallas, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Benchmark Research, Fort Worth, Texas
  - HG Pediatrics, Houston, Texas
  - Renu Garg, MD Pediatrics, Houston, Texas
  - Van Tran Family Practice, Houston, Texas
  - Ventavia Research Group, LLC, Houston, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - SCR of Texas, LLC, Keller, Texas
  - SMS Clinical Research, Mesquite, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - DM Clinical Research - Kool Kids Pediatrics, Tomball, Texas
  - DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Clinical Alliance for Research & Education - Infectious Diseases (CARE-ID), Annandale, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Research Building, Wenatchee, Washington
  - Wenatchee Valley Hospital, Wenatchee, Washington
- Brazil (2):
  - Obras Sociais Irma Dulce, Salvador, Estado de Bahia
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Germany (2):
  - Studienzentrum Dr. Keller, Frankfurt
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
- Sheba Medical Center, Ramat Gan, Central District, Israel
- South Africa (10):
  - Synergy Biomed Research Institute, East London, Eastern Cape
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Clinresco Centres, Kempton Park, Gauteng
  - Dr A Jacovides & Partners Inc., Midrand, Gauteng
  - Botho Ke Bontle Health Services PTY LTD, Pretoria, Gauteng
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - TREAD Research, Cape Town, Parow
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Jongaie Research, Pretoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winokur P, Diya O, Fitz-Patrick D, Dever M, Gayed J, Lockhart S, Xu X, Zhang Y, Bangad V, Wadsworth LT, Cannon K, Cardona JF, Usdan L, Ginis J, Mensa FJ, Zou J, Xie X, Lu C, Buitrago S, Scully IL, Cooper D, Koury K, Jansen KU, Tureci Ӧ, Sahin U, Swanson KA, Gruber WC, Kitchin N. Safety and Immunogenicity of a Fourth Dose of Omicron-BA.1-Adapted BNT162b2 COVID-19 Vaccines in Adults 18-55 Years Old. Clin Infect Dis. 2026 Jan 21:ciag026. doi: 10.1093/cid/ciag026. Online ahead of print. PMID 41560517
- [Derived] Muik A, Lui BG, Quandt J, Diao H, Fu Y, Bacher M, Gordon J, Toker A, Grosser J, Ozhelvaci O, Grikscheit K, Hoehl S, Kohmer N, Lustig Y, Regev-Yochay G, Ciesek S, Beguir K, Poran A, Vogler I, Tureci O, Sahin U. Progressive loss of conserved spike protein neutralizing antibody sites in Omicron sublineages is balanced by preserved T cell immunity. Cell Rep. 2023 Aug 29;42(8):112888. doi: 10.1016/j.celrep.2023.112888. Epub 2023 Jul 31. PMID 37527039
- [Derived] Winokur P, Gayed J, Fitz-Patrick D, Thomas SJ, Diya O, Lockhart S, Xu X, Zhang Y, Bangad V, Schwartz HI, Denham D, Cardona JF, Usdan L, Ginis J, Mensa FJ, Zou J, Xie X, Shi PY, Lu C, Buitrago S, Scully IL, Cooper D, Koury K, Jansen KU, Tureci O, Sahin U, Swanson KA, Gruber WC, Kitchin N; C4591031 Clinical Trial Group. Bivalent Omicron BA.1-Adapted BNT162b2 Booster in Adults Older than 55 Years. N Engl J Med. 2023 Jan 19;388(3):214-227. doi: 10.1056/NEJMoa2213082. PMID 36652353
- [Derived] Moreira ED Jr, Kitchin N, Xu X, Dychter SS, Lockhart S, Gurtman A, Perez JL, Zerbini C, Dever ME, Jennings TW, Brandon DM, Cannon KD, Koren MJ, Denham DS, Berhe M, Fitz-Patrick D, Hammitt LL, Klein NP, Nell H, Keep G, Wang X, Koury K, Swanson KA, Cooper D, Lu C, Tureci O, Lagkadinou E, Tresnan DB, Dormitzer PR, Sahin U, Gruber WC, Jansen KU; C4591031 Clinical Trial Group. Safety and Efficacy of a Third Dose of BNT162b2 Covid-19 Vaccine. N Engl J Med. 2022 May 19;386(20):1910-1921. doi: 10.1056/NEJMoa2200674. Epub 2022 Mar 23. PMID 35320659
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 6 parts: sub-study A (SSA), sub-study B (SSB), sub-study C (SSC), sub-study D (SSD), sub-study E (SSE) and sub-study F (SSF).
Pre-assignment Details: SSA: 10133 participants randomized, 10121 vaccinated and evaluated. SSB: 1487 participants randomized,1485 vaccinated and evaluated. SSC: 140 participants randomized, vaccinated, evaluated. SSD: 1469 participants randomized 1467 vaccinated, 1465vaccinated with 30 mcg BNT162b2 and BNT162b2 OMI and evaluated. SSE: 3020 participants randomized, 3014 vaccinated, 3010 vaccinated with 30 and 60 mcg BNT162b2 and BNT162b2 OMI and evaluated. SSF: 123 participants randomized,122 vaccinated and evaluated.
Groups:
- SSA: BNT162b2 30 mcg: Blinded and Open Label Period: Participants received one dose (30 microgram) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
- SSA: Placebo: Blinded Period, Then BNT162b2 30 mcg Open-Label Period: Participants received placebo (normal saline solution of 0.9 percent [%] sodium chloride) intramuscularly during the Double-Blinded period. Then, they could have received BNT162b2 30 mcg in the Open-Label Period.
- SSB: BNT162b2 30 mcg Then Placebo: Participants received one dose (30 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm on Day 1 and received placebo (normal saline solution of 0.9 % sodium chloride) intramuscularly on Day 28.
- SSB: Placebo Then BNT162b2 30 mcg: Participants received placebo (normal saline solution of 0.9 % sodium chloride) intramuscularly on Day 1 and one dose (30 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm on Day 28.
- SSC: BNT162b2 10 mcg: Participants who previously received two booster doses of BNT162b2 prior to enrollment in SSC, received one booster dose (10 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
- SSC: BNT162b2 30 mcg: Participants who previously received two booster doses of BNT162b2 prior to enrollment in SSC, received one booster dose (30 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
- SSD: Cohort 1: Group 1; SSF: BNT162b2 OMI 30 mcg: Participants received one dose (30 mcg) of BNT162b2 Omicron (OMI) intramuscularly in the deltoid muscle of the non-dominant arm.
- SSD: Cohort 1: Group 2: Participants received two doses (30 mcg) of BNT162b2 Omicron (OMI) intramuscularly 4 weeks apart in the deltoid muscle of the non-dominant arm.
- SSD: Cohort 1: Group 2b; SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg; SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg; SSF: BNT162b2 30 mcg: Participants received one dose (30 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
- SSD: Cohort 2: Group 3: Participants received one dose (30 mcg) of BNT162b2 Omicron (OMI) intramuscularly in the deltoid muscle of the non-dominant arm. After 3 months, participants upon their consent received optional additional one dose (30 mcg) of BNT162b2 OMI.
- SSD: Cohort 2: Group 4: Participants received one dose (30 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm. After 3 months, participants upon their consent received optional additional one dose (30 mcg) of BNT162b2 OMI.
- SSD: Cohort 3: Group 5: Participants received two doses (30 mcg) of BNT162b2 Omicron (OMI) 3 weeks apart intramuscularly in the deltoid muscle of the non-dominant arm. Participants upon their consent received one dose (30 mcg) of BNT162b2 5 months after second dose of BNT162b2 OMI vaccination.
- SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg; SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg; SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg; SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg; SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg: Participants received a total of 60 mcg bivalent BNT162b2 (30 mcg BNT162b2 and 30 mcg BNT162b2 OMI) as a single dose intramuscularly in the deltoid muscle of the non-dominant arm.
- SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg; SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg; SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg; SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg; SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg: Participants received a total of 30 mcg bivalent BNT162b2 (15 mcg BNT162b2 and 15 mcg BNT162b2 OMI) as a single dose intramuscularly in the deltoid muscle of the non-dominant arm.
- SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg: Participants received one dose (60 mcg) of BNT162b2 OMI intramuscularly in the deltoid muscle of the non-dominant arm.
- SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg; SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg; SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg; SSF: BNT162b2 OMI 60 mcg: Participants received one dose (60 mcg) of BNT162b2 Omicron (OMI) intramuscularly in the deltoid muscle of the non-dominant arm.
- SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg; SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg; SSF: BNT162b2 60 mcg: Participants received one dose (60 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
- SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg; SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg: Participants received one dose (30 mcg) of BNT162b2 OMI intramuscularly in the deltoid muscle of the non-dominant arm.
Period: Blinded Period
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period, Then BNT162b2 30 mcg Open-Label Period | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4 | SSD: Cohort 3: Group 5 | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Started | 5080 (Vaccinated with booster dose) | 5041 (Vaccinated with booster dose) | 753 (Vaccinated with booster dose) | 732 (Vaccinated with booster dose) | 75 (Vaccinated with booster dose) | 65 (Vaccinated with booster dose) | 216 (Vaccinated with booster dose) | 197 (Vaccinated with booster dose) | 204 (Vaccinated with booster dose) | 315 (Vaccinated with booster dose) | 325 (Vaccinated with booster dose) | 210 (Vaccinated with booster dose) | 30 (Vaccinated with booster dose) | 30 (Vaccinated with booster dose) | 30 (Vaccinated with booster dose) | 482 (Vaccinated with booster dose) | 159 (Vaccinated with booster dose) | 321 (Vaccinated with booster dose) | 20 (Vaccinated with booster dose) | 20 (Vaccinated with booster dose) | 20 (Vaccinated with booster dose) | 20 (Vaccinated with booster dose) | 20 (Vaccinated with booster dose) | 20 (Vaccinated with booster dose) | 305 (Vaccinated with booster dose) | 302 (Vaccinated with booster dose) | 307 (Vaccinated with booster dose) | 307 (Vaccinated with booster dose) | 308 (Vaccinated with booster dose) | 313 (Vaccinated with booster dose) | 21 (Vaccinated with booster dose) | 19 (Vaccinated with booster dose) | 21 (Vaccinated with booster dose) | 20 (Vaccinated with booster dose) | 20 (Vaccinated with booster dose) | 21 (Vaccinated with booster dose)
Safety Analysis Set | 5080 | 5041 | 753 | 732 | 75 | 65 | 216 | 197 | 204 | 315 | 323 | 210 | 30 | 30 | 30 | 482 | 159 | 321 | 20 | 20 | 20 | 20 | 20 | 20 | 305 | 302 | 307 | 307 | 308 | 313 | 21 | 19 | 21 | 20 | 20 | 21
Completed | 421 | 22 | 726 | 693 | 69 | 58 | 197 | 183 | 193 | 286 | 293 | 159 | 28 | 30 | 27 | 450 | 151 | 302 | 19 | 19 | 19 | 19 | 20 | 19 | 292 | 294 | 291 | 299 | 294 | 307 | 21 | 19 | 21 | 20 | 20 | 21
Not Completed | 4659 | 5019 | 27 | 39 | 6 | 7 | 19 | 14 | 11 | 29 | 32 | 51 | 2 | 0 | 3 | 32 | 8 | 19 | 1 | 1 | 1 | 1 | 0 | 1 | 13 | 8 | 16 | 8 | 14 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 28 | 28 | 7 | 14 | 3 | 2 | 6 | 4 | 5 | 8 | 10 | 32 | 0 | 0 | 0 | 12 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 14 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 4 | 6 | 1 | 0 | 0 | 2 | 6 | 4 | 6 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 6 | 5 | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer meets eligibility criteria | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 54 | 3 | 4 | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 26 | 62 | 14 | 16 | 1 | 2 | 9 | 5 | 3 | 15 | 11 | 7 | 2 | 0 | 1 | 11 | 2 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 1 | 5 | 1 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Refused further study procedures | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participants entered open label period | 4544 | 4906 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Medication error | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Period
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period, Then BNT162b2 30 mcg Open-Label Period | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4 | SSD: Cohort 3: Group 5 | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Started | 4544 (Participants received BNT162b2 30 mcg in blinded period then entered open label period.) | 4906 (Participants who received placebo in blinded period then either received BNT162b2 30 mcg in open label period or discontinued or completed the study without BNT162b2 administration.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Open-label BNT162b2 30 mcg | 4544 | 4430 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3272 | 3878 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1272 | 1028 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 109 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 377 | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer meets eligibility criteria | 20 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 621 | 429 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 135 | 25 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Refused further study procedures | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by parent/guardian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive Open-label BNT162b2 30 mcg | 0 | 476 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention.
Groups:
- SSA: Placebo: Blinded Period: Participants received placebo (normal saline solution of 0.9 percent [%] sodium chloride) intramuscularly.
- Total: Total of all reporting groups
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4 | SSD: Cohort 3: Group 5 | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg | Total
Number analyzed (Participants) | 5080 | 5041 | 753 | 732 | 75 | 65 | 216 | 197 | 204 | 315 | 323 | 210 | 30 | 30 | 30 | 482 | 159 | 321 | 20 | 20 | 20 | 20 | 20 | 20 | 305 | 302 | 307 | 307 | 308 | 313 | 21 | 19 | 21 | 20 | 20 | 21 | 16347
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 46 | 44 | 233 | 228 | 75 | 65 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 691
  Adults (18-64 years) | 3859 | 3811 | 520 | 504 | 0 | 0 | 216 | 197 | 204 | 315 | 323 | 210 | 30 | 30 | 30 | 482 | 159 | 321 | 6 | 5 | 5 | 7 | 5 | 9 | 126 | 105 | 121 | 123 | 112 | 109 | 6 | 7 | 6 | 8 | 9 | 9 | 11989
  From 65-84 years | 1166 | 1174 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 15 | 13 | 15 | 10 | 176 | 196 | 186 | 183 | 194 | 199 | 15 | 12 | 15 | 12 | 11 | 12 | 3633
  85 years and over | 9 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2624 | 2526 | 434 | 447 | 37 | 33 | 137 | 119 | 121 | 152 | 156 | 106 | 14 | 17 | 15 | 269 | 89 | 180 | 8 | 9 | 14 | 12 | 7 | 11 | 160 | 157 | 153 | 154 | 144 | 162 | 9 | 9 | 13 | 10 | 8 | 12 | 8528
  Male | 2456 | 2515 | 319 | 285 | 38 | 32 | 79 | 78 | 83 | 163 | 167 | 104 | 16 | 13 | 15 | 213 | 70 | 141 | 12 | 11 | 6 | 8 | 13 | 9 | 145 | 145 | 154 | 153 | 164 | 151 | 12 | 10 | 8 | 10 | 12 | 9 | 7819
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3998 | 4002 | 491 | 493 | 55 | 50 | 16 | 8 | 9 | 237 | 224 | 31 | 25 | 24 | 26 | 389 | 124 | 250 | 16 | 19 | 15 | 17 | 14 | 16 | 268 | 254 | 261 | 262 | 277 | 272 | 21 | 19 | 21 | 20 | 20 | 21 | 12265
  Black or African American | 470 | 457 | 159 | 155 | 11 | 9 | 176 | 172 | 178 | 21 | 34 | 155 | 2 | 3 | 1 | 34 | 10 | 32 | 1 | 0 | 2 | 2 | 2 | 1 | 19 | 22 | 23 | 20 | 13 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 2203
  American Indian or Alaska Native | 86 | 92 | 4 | 6 | 0 | 0 | 1 | 0 | 2 | 1 | 4 | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 206
  Asian | 288 | 269 | 61 | 58 | 7 | 5 | 4 | 2 | 1 | 42 | 45 | 1 | 2 | 3 | 3 | 42 | 20 | 25 | 3 | 1 | 2 | 1 | 4 | 3 | 13 | 20 | 16 | 20 | 16 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 994
  Native Hawaiian or other Pacific Islander | 7 | 11 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 34
  Multiracial | 209 | 197 | 24 | 12 | 1 | 0 | 10 | 11 | 6 | 10 | 12 | 22 | 1 | 0 | 0 | 12 | 2 | 8 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 5 | 6 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 559
  Not reported | 22 | 13 | 13 | 7 | 1 | 0 | 9 | 4 | 8 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 759 | 750 | 152 | 150 | 15 | 11 | 6 | 0 | 4 | 48 | 46 | 7 | 3 | 4 | 3 | 66 | 17 | 39 | 1 | 1 | 4 | 3 | 2 | 4 | 57 | 38 | 44 | 46 | 45 | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 2369
  Non-Hispanic/non-Latino | 4309 | 4283 | 595 | 577 | 59 | 53 | 209 | 196 | 200 | 266 | 277 | 202 | 27 | 26 | 27 | 413 | 142 | 282 | 19 | 19 | 16 | 17 | 18 | 16 | 248 | 264 | 263 | 261 | 263 | 269 | 21 | 19 | 21 | 20 | 19 | 21 | 13937
  Not reported | 12 | 8 | 6 | 5 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 41

OUTCOME MEASURES:

1. Primary Outcome: SSA: Occurrence of First COVID-19 Infection After Booster Dose Per 1000 Person-Years of Blinded Follow-up Without Evidence of Past SARS-CoV-2 Infection at Interim Analysis: Evaluable Efficacy Population
Description: Occurrences (number of cases) of first COVID-19 infection in participants after booster dose per 1000 person-year, without past SARS-CoV-2 infection at interim analysis were reported in this outcome measure.
Time Frame: From 7 Days after booster vaccination to end of surveillance period, total surveillance time (in 1000 person-year [PY]) for BNT162b2 was 0.823 and for Placebo was 0.792
Population: SSA evaluable efficacy population included all eligible randomized participants who received the booster vaccination as randomized and had no other important protocol deviations as determined by the clinician. Human Immunodeficiency Virus (HIV) positive participants were excluded from this analysis. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Number of first Covid-19 cases/1000 PY
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 4659 | 4614
Number of first Covid-19 cases/1000 PY | 7.290 | 155.303
Statistical Analysis 1: Comparison: SSA: BNT162b2 30 mcg: Blinded and Open Label Period vs SSA: Placebo: Blinded Period; 2-Sided CI for Relative vaccine efficacy (RVE) is derived based on the Clopper and Pearson method adjusted for surveillance time; Test type: Other; Adjusted Surveillance Time = 95.3, 95% CI 2-sided [89.5 to 98.3]

2. Primary Outcome: SSA: Occurrence of First COVID-19 Infection After Booster Dose Per 1000 Person-Years of Blinded Follow-up With and Without Evidence of Past SARS-CoV-2 Infection at Interim Analysis: Evaluable Efficacy Population
Description: Occurrences (number of cases) of first COVID-19 infection in participants after booster dose with and without past SARS-CoV-2 infection at interim analysis were reported in this outcome measure.
Time Frame: From 7 Days after booster vaccination to end of surveillance period, total surveillance time (in 1000 person-year) for BNT162b2 was 0.871 and for Placebo was 0.835
Population: SSA evaluable efficacy population included all eligible randomized participants who received the booster vaccination as randomized and had no other important protocol deviations as determined by the clinician. HIV positive participants were excluded from this analysis. Here, 'Number of Subjects Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Number of first Covid-19 cases/1000 PY
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 4934 | 4863
Number of first Covid-19 cases/1000 PY | 8.037 | 148.503
Statistical Analysis 1: Comparison: SSA: BNT162b2 30 mcg: Blinded and Open Label Period vs SSA: Placebo: Blinded Period; 2-Sided CI for RVE is derived based on the Clopper and Pearson method adjusted for surveillance time; Test type: Other; Adjusted Surveillance Time = 94.6, 95% CI 2-sided [88.5 to 97.9]

3. Primary Outcome: SSA: Occurrence of First COVID-19 Infection After Booster Dose Per 1000 Person-Years of Blinded Follow-up Without Evidence of Past SARS-CoV-2 Infection at Final Analysis: Evaluable Efficacy Population
Description: Occurrences (number of cases) of first COVID-19 infection in participants after booster dose without past SARS-CoV-2 infection at final analysis were reported in this outcome measure.
Time Frame: From 7 Days after booster vaccination to end of surveillance period, total surveillance time (in 1000 person-year) for BNT162b2 was 1.098 and for Placebo was 0.932
Population: SSA evaluable efficacy population included all eligible randomized participants who received the booster vaccination as randomized and had no other important protocol deviations as determined by the clinician. HIV positive participants were excluded from this analysis. Here, 'Number of participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Number of first Covid-19 cases/1000 PY
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 4639 | 4601
Number of first Covid-19 cases/1000 PY | 57.377 | 158.798
Statistical Analysis 1: Comparison: SSA: BNT162b2 30 mcg: Blinded and Open Label Period vs SSA: Placebo: Blinded Period; [analysis description as in outcome 1, analysis 1]; Test type: Other; Adjusted Surveillance Time = 63.9, 95% CI 2-sided [51.1 to 73.5]

4. Primary Outcome: SSA: Occurrence of First COVID-19 Infection After Booster Dose Per 1000 Person-Years of Blinded Follow-up With and Without Evidence of Past SARS-CoV-2 Infection at Final Analysis: Evaluable Efficacy Population
Description: Occurrences (number of cases) of first COVID-19 infection in participants after booster dose with and without past SARS-CoV-2 infection at final analysis were reported in this outcome measure.
Time Frame: From 7 Days after booster vaccination to end of surveillance period, total surveillance time (in 1000 person-year) for BNT162b2 was 1.173 and for Placebo was 0.989
Population: as for outcome 3
Measure: Number; unit: Number of first Covid-19 cases/1000 PY
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 4903 | 4846
Number of first Covid-19 cases/1000 PY | 57.118 | 151.668
Statistical Analysis 1: Comparison: SSA: BNT162b2 30 mcg: Blinded and Open Label Period vs SSA: Placebo: Blinded Period; 2-Sided CI for RVE is derived based on the Clopper and Pearson method adjusted for surveillance time; Test type: Other; Adjusted Surveillance Time = 62.4, 95% CI 2-sided [49.5 to 72.2]

5. Primary Outcome: SSA: Percentage of Participants Reporting Adverse Events
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: From booster dose (Day 1) to 1 month after booster dose
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention. HIV positive participants were excluded from this analysis. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 5054 | 5016
Percentage of participants | 26.3 [25.0 to 27.5] | 7.1 [6.4 to 7.8]

6. Primary Outcome: SSA: Percentage of Participants Reporting Serious Adverse Events (SAE)
Description: An SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect; or that was considered as an important medical event.
Time Frame: BNT162b2 30 mcg, Placebo then BNT162b2 30 mcg: From BNT162b2 dose to 6 months after BNT162b2 dose; Placebo: From placebo dose to unblinding for original placebo participants. Median blinded follow-up period for Placebo group=2.8 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSA: Original Placebo/BNT162b2 30 mcg: Open Label Period: Participants received placebo (normal saline solution of 0.9 percent [%] sodium chloride) intramuscularly and then one dose (30 microgram) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period | SSA: Original Placebo/BNT162b2 30 mcg: Open Label Period
Number analyzed (Participants) | 5054 | 5016 | 4405
Percentage of participants | 1.4 [1.1 to 1.8] | 0.8 [0.6 to 1.1] | 1.0 [0.7 to 1.3]

7. Primary Outcome: SSB: Percentage of Participants With Elevated Troponin I Level Pre-Dose; Vaccination 1
Description: Percentage of participants with elevated troponin I levels before administration of Vaccination 1 were reported in this outcome measure.
Time Frame: Pre-dose on Day 1 (Vaccination 1)
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 751 | 730
Percentage of participants | 0.7 [0.2 to 1.5] | 0.5 [0.1 to 1.4]

8. Primary Outcome: SSB: Percentage of Participants With Elevated Troponin I Level Within 5 Days After Vaccination 1
Description: Percentage of participants with elevated troponin I levels within 5 days after administration of Vaccination 1 were reported in this outcome measure.
Time Frame: Within 5 days after Vaccination 1
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 719 | 693
Percentage of participants | 1.0 [0.4 to 2.0] | 0.6 [0.2 to 1.5]

9. Primary Outcome: SSB: Percentage of Participants With Elevated Troponin I Level Pre-Vaccination 2 (1 Month After Vaccination 1)
Description: Percentage of participants with elevated troponin I levels pre vaccination 2 were reported in this outcome measure.
Time Frame: Pre-Vaccination 2 (1 month after Vaccination 1)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 628 | 600
Percentage of participants | 1.1 [0.4 to 2.3] | 0.3 [0.0 to 1.2]

10. Primary Outcome: SSB: Percentage of Participants With Elevated Troponin I Level Within 5 Days After Vaccination 2
Description: Percentage of participants with elevated troponin I levels within 5 days after administration of Vaccination 2 were reported in this outcome measure.
Time Frame: Within 5 days after vaccination 2
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure and received two doses of study vaccination for SSB.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 667 | 634
Percentage of participants | 1.5 [0.7 to 2.7] | 0.3 [0.0 to 1.1]

11. Primary Outcome: SSB: Percentage of Participants With Elevated Troponin I Level 1 Month After Vaccination 2
Description: Percentage of participants with elevated troponin I levels within 1 month after administration of Vaccination 2 were reported in this outcome measure.
Time Frame: 1 month after Vaccination 2
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 676 | 645
Percentage of participants | 0.7 [0.2 to 1.7] | 0.3 [0.0 to 1.1]

12. Primary Outcome: SSB: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions were recorded by participants in e-diary. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu =0.5 centimeter (cm) and were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Percentage of participants reporting local reactions after Vaccination 1 and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented.
Time Frame: Day 1 up to Day 7 after Vaccination 1
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'Number of Participants Analyzed' (N) signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 747 | 728
Percentage of participants
  Redness: Any | 5.8 [4.2 to 7.7] | 0.5 [0.1 to 1.4]
  Redness: Mild | 4.4 [3.1 to 6.1] | 0.4 [0.1 to 1.2]
  Redness: Moderate | 1.1 [0.5 to 2.1] | 0.1 [0.0 to 0.8]
  Redness: Severe | 0.3 [0.0 to 1.0] | 0 [0.0 to 0.5]
  Redness: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Swelling: Any | 6.6 [4.9 to 8.6] | 0.5 [0.1 to 1.4]
  Swelling: Mild | 5.0 [3.5 to 6.8] | 0.4 [0.1 to 1.2]
  Swelling: Moderate | 1.5 [0.7 to 2.6] | 0 [0.0 to 0.5]
  Swelling: Severe | 0.1 [0.0 to 0.7] | 0.1 [0.0 to 0.8]
  Swelling: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Pain at injection site: Any | 74.4 [71.1 to 77.5] | 13.9 [11.4 to 16.6]
  Pain at injection site: Mild | 48.7 [45.1 to 52.4] | 12.2 [9.9 to 14.8]
  Pain at injection site: Moderate | 25.4 [22.3 to 28.7] | 1.6 [0.9 to 2.9]
  Pain at injection site: Severe | 0.3 [0.0 to 1.0] | 0 [0.0 to 0.5]
  Pain at injection site: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]

13. Primary Outcome: SSB: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions were recorded by participants in e-diary. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu =0.5 centimeter (cm) and were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Percentage of participants reporting local reactions after Vaccination 2 and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented.
Time Frame: Day 1 up to Day 7 after Vaccination 2
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'Number of Participants Analyzed' (N) signifies participants evaluable for this outcome measure and received two doses of study vaccination for SSB.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 706 | 672
Percentage of participants
  Redness: Any | 0.7 [0.2 to 1.6] | 4.6 [3.2 to 6.5]
  Redness: Mild | 0.3 [0.0 to 1.0] | 2.8 [1.7 to 4.4]
  Redness: Moderate | 0.4 [0.1 to 1.2] | 1.5 [0.7 to 2.7]
  Redness: Severe | 0 [0.0 to 0.5] | 0.3 [0.0 to 1.1]
  Redness: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Swelling: Any | 0.4 [0.1 to 1.2] | 5.5 [3.9 to 7.5]
  Swelling: Mild | 0.4 [0.1 to 1.2] | 3.4 [2.2 to 5.1]
  Swelling: Moderate | 0 [0.0 to 0.5] | 1.9 [1.0 to 3.3]
  Swelling: Severe | 0 [0.0 to 0.5] | 0.1 [0.0 to 0.8]
  Swelling: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Pain at injection site: Any | 8.8 [6.8 to 11.1] | 71.7 [68.2 to 75.1]
  Pain at injection site: Mild | 6.7 [4.9 to 8.8] | 40.3 [36.6 to 44.1]
  Pain at injection site: Moderate | 2.1 [1.2 to 3.5] | 30.5 [27.0 to 34.1]
  Pain at injection site: Severe | 0 [0.0 to 0.5] | 0.9 [0.3 to 1.9]
  Pain at injection site: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]

14. Primary Outcome: SSB: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events were recorded in e-diary. Fever: oral temperature greater than or equal to (>=) 38.0 degree Celsius (deg C) and categorized as >=38.0-38.4 deg C, >38.4-38.9 deg C, >38.9-40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity) and Grade 4 (ER visit/hospitalization). Vomiting: mild: 1-2 times in 24 hours (h), moderate: >2 times in 24h, severe: required intravenous hydration and Grade 4: ER visit/hospitalization for hypotensive shock. Diarrhea: mild: 2-3 loose stools in 24h, moderate: 4-5 loose stools in 24h, severe: 6 or more loose stools in 24h and Grade 4: ER visit/hospitalization for severe diarrhea. Grade 4 were classified by investigator or medically qualified person. Exact 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 up to Day 7 after Vaccination 1
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 747 | 728
Percentage of participants
  Fever: >=38 deg C | 6.0 [4.4 to 8.0] | 1.9 [1.1 to 3.2]
  Fever: 38.0 to 38.4 deg C | 4.1 [2.8 to 5.8] | 1.4 [0.7 to 2.5]
  Fever: >38.4 to 38.9 deg C | 1.7 [0.9 to 3.0] | 0.3 [0.0 to 1.0]
  Fever: >38.9 to 40.0 deg C | 0.1 [0.0 to 0.7] | 0.3 [0.0 to 1.0]
  Fever: >40.0 deg C | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Fatigue: Any | 54.2 [50.6 to 57.8] | 31.9 [28.5 to 35.4]
  Fatigue: Mild | 27.4 [24.3 to 30.8] | 19.5 [16.7 to 22.6]
  Fatigue: Moderate | 25.3 [22.2 to 28.6] | 12.2 [9.9 to 14.8]
  Fatigue: Severe | 1.5 [0.7 to 2.6] | 0.1 [0.0 to 0.8]
  Fatigue: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Headache: Any | 42.6 [39.0 to 46.2] | 28.3 [25.0 to 31.7]
  Headache: Mild | 24.2 [21.2 to 27.5] | 18.0 [15.3 to 21.0]
  Headache: Moderate | 17.3 [14.6 to 20.2] | 10.0 [7.9 to 12.4]
  Headache: Severe | 1.1 [0.5 to 2.1] | 0.3 [0.0 to 1.0]
  Headache: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Chills: Any | 17.1 [14.5 to 20.0] | 5.9 [4.3 to 7.9]
  Chills: Mild | 10.6 [8.5 to 13.0] | 4.4 [3.0 to 6.1]
  Chills: Moderate | 6.3 [4.7 to 8.3] | 1.5 [0.8 to 2.7]
  Chills: Severe | 0.3 [0.0 to 1.0] | 0 [0.0 to 0.5]
  Chills: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Vomiting: Any | 3.2 [2.1 to 4.7] | 0.8 [0.3 to 1.8]
  Vomiting: Mild | 2.8 [1.7 to 4.3] | 0.7 [0.2 to 1.6]
  Vomiting: Moderate | 0.4 [0.1 to 1.2] | 0.1 [0.0 to 0.8]
  Vomiting: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Vomiting: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Diarrhea: Any | 7.4 [5.6 to 9.5] | 7.4 [5.6 to 9.6]
  Diarrhea: Mild | 6.4 [4.8 to 8.4] | 6.0 [4.4 to 8.0]
  Diarrhea: Moderate | 0.9 [0.4 to 1.9] | 1.4 [0.7 to 2.5]
  Diarrhea: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Diarrhea: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  New or worsened muscle pain: Any | 27.6 [24.4 to 30.9] | 7.7 [5.9 to 9.9]
  New or worsened muscle pain: Mild | 14.1 [11.6 to 16.8] | 5.1 [3.6 to 6.9]
  New or worsened muscle pain: Moderate | 13.3 [10.9 to 15.9] | 2.5 [1.5 to 3.9]
  New or worsened muscle pain: Severe | 0.3 [0.0 to 1.0] | 0.1 [0.0 to 0.8]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  New or worsened joint pain: Any | 12.9 [10.5 to 15.5] | 4.5 [3.1 to 6.3]
  New or worsened joint pain: Mild | 8.3 [6.4 to 10.5] | 3.0 [1.9 to 4.5]
  New or worsened joint pain: Moderate | 4.3 [2.9 to 6.0] | 1.5 [0.8 to 2.7]
  New or worsened joint pain: Severe | 0.3 [0.0 to 1.0] | 0 [0.0 to 0.5]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]

15. Primary Outcome: SSB: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2
Description: as for outcome 14
Time Frame: Day 1 up to Day 7 after Vaccination 2
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 706 | 672
Percentage of participants
  Fever: >=38 deg C | 0.4 [0.1 to 1.2] | 4.3 [2.9 to 6.1]
  Fever: 38.0 to 38.4 deg C | 0.3 [0.0 to 1.0] | 2.5 [1.5 to 4.0]
  Fever: >38.4 to 38.9 deg C | 0.1 [0.0 to 0.8] | 1.3 [0.6 to 2.5]
  Fever: >38.9 to 40.0 deg C | 0 [0.0 to 0.5] | 0.4 [0.1 to 1.3]
  Fever: >40.0 deg C | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Fatigue: Any | 17.6 [14.8 to 20.6] | 47.3 [43.5 to 51.2]
  Fatigue: Mild | 8.6 [6.7 to 11.0] | 18.8 [15.9 to 21.9]
  Fatigue: Moderate | 8.5 [6.5 to 10.8] | 27.1 [23.8 to 30.6]
  Fatigue: Severe | 0.4 [0.1 to 1.2] | 1.5 [0.7 to 2.7]
  Fatigue: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Headache: Any | 17.8 [15.1 to 20.9] | 39.7 [36.0 to 43.5]
  Headache: Mild | 10.3 [8.2 to 12.8] | 19.8 [16.8 to 23.0]
  Headache: Moderate | 7.2 [5.4 to 9.4] | 19.0 [16.1 to 22.2]
  Headache: Severe | 0.3 [0.0 to 1.0] | 0.9 [0.3 to 1.9]
  Headache: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Chills: Any | 3.7 [2.4 to 5.3] | 22.3 [19.2 to 25.7]
  Chills: Mild | 2.3 [1.3 to 3.7] | 13.2 [10.8 to 16.0]
  Chills: Moderate | 1.1 [0.5 to 2.2] | 8.8 [6.8 to 11.2]
  Chills: Severe | 0.3 [0.0 to 1.0] | 0.3 [0.0 to 1.1]
  Chills: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Vomiting: Any | 1.0 [0.4 to 2.0] | 1.9 [1.0 to 3.3]
  Vomiting: Mild | 0.7 [0.2 to 1.6] | 1.8 [0.9 to 3.1]
  Vomiting: Moderate | 0.3 [0.0 to 1.0] | 0.1 [0.0 to 0.8]
  Vomiting: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Vomiting: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Diarrhea: Any | 3.3 [2.1 to 4.8] | 8.0 [6.1 to 10.4]
  Diarrhea: Mild | 2.1 [1.2 to 3.5] | 6.5 [4.8 to 8.7]
  Diarrhea: Moderate | 1.1 [0.5 to 2.2] | 1.5 [0.7 to 2.7]
  Diarrhea: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Diarrhea: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  New or worsened muscle pain: Any | 4.5 [3.1 to 6.3] | 29.2 [25.8 to 32.8]
  New or worsened muscle pain: Mild | 2.3 [1.3 to 3.7] | 15.9 [13.2 to 18.9]
  New or worsened muscle pain: Moderate | 2.1 [1.2 to 3.5] | 12.9 [10.5 to 15.7]
  New or worsened muscle pain: Severe | 0.1 [0.0 to 0.8] | 0.3 [0.0 to 1.1]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  New or worsened joint pain: Any | 3.1 [2.0 to 4.7] | 12.2 [9.8 to 14.9]
  New or worsened joint pain: Mild | 1.6 [0.8 to 2.8] | 7.4 [5.6 to 9.7]
  New or worsened joint pain: Moderate | 1.6 [0.8 to 2.8] | 4.8 [3.3 to 6.7]
  New or worsened joint pain: Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]

16. Primary Outcome: SSB: Percentage of Participants Reporting Adverse Events (AEs) 1 Month After Vaccination 1
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs within 1 month after Vaccination 1 were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Vaccination 1 up to 1 Month After Vaccination 1
Population: Safety population included all participant who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 753 | 732
Percentage of participants | 9.4 [7.4 to 11.7] | 10.4 [8.3 to 12.8]

17. Primary Outcome: SSB: Percentage of Participants Reporting Adverse Events (AEs) 1 Month After Vaccination 2
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs within 1 month after Vaccination 2 were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Vaccination 2 up to 1 month after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of the study intervention. Participants who did not receive Vaccination 2 or who received an incorrect vaccine at Vaccination 2 were excluded from this analysis. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure and received two doses of study vaccination for SSB.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 731 | 700
Percentage of participants | 5.6 [4.1 to 7.5] | 7.4 [5.6 to 9.6]

18. Primary Outcome: SSB: Percentage of Participants Reporting Serious Adverse Events (SAEs) 1 Month After Vaccination 1
Description: An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening; resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required inpatient hospitalization or prolongation of existing hospitalization. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Vaccination 1 up to 1 month after Vaccination 1
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 753 | 732
Percentage of participants | 0.1 [0.0 to 0.7] | 0.3 [0.0 to 1.0]

19. Primary Outcome: SSB: Percentage of Participants Reporting Serious Adverse Events (SAEs) 1 Month After Vaccination 2
Description: as for outcome 18
Time Frame: Vaccination 2 up to 1 month after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, 'Number of Participants Analyzed' signifies participants evaluable for the specified outcome measure and received two doses of study vaccination for SSB.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: BNT162b2 30 mcg Then Placebo | SSB: Placebo Then BNT162b2 30 mcg
Number analyzed (Participants) | 731 | 700
Percentage of participants | 0 [0.0 to 0.5] | 0.1 [0.0 to 0.8]

20. Primary Outcome: SSC: Percentage of Participants With Local Reactions Within 7 Days After Booster Dose
Description: Local reactions were recorded by participants in e-diary. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu =0.5 cm and were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Percentage of participants reporting local reactions after the booster (third) dose and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented.
Time Frame: Day 1 up to Day 7 after the booster dose
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 75 | 64
Percentage of participants
  Redness: Any | 1.3 [0.0 to 7.2] | 6.3 [1.7 to 15.2]
  Redness: Mild | 1.3 [0.0 to 7.2] | 4.7 [1.0 to 13.1]
  Redness: Moderate | 0 [0.0 to 4.8] | 1.6 [0.0 to 8.4]
  Redness: Severe | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Redness: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Swelling: Any | 2.7 [0.3 to 9.3] | 9.4 [3.5 to 19.3]
  Swelling: Mild | 2.7 [0.3 to 9.3] | 6.3 [1.7 to 15.2]
  Swelling: Moderate | 0 [0.0 to 4.8] | 3.1 [0.4 to 10.8]
  Swelling: Severe | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Swelling: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Pain at the injection site: Any | 56.0 [44.1 to 67.5] | 78.1 [66.0 to 87.5]
  Pain at the injection site: Mild | 40.0 [28.9 to 52.0] | 46.9 [34.3 to 59.8]
  Pain at the injection site: Moderate | 16.0 [8.6 to 26.3] | 31.3 [20.2 to 44.1]
  Pain at the injection site: Severe | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Pain at the injection site: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]

21. Primary Outcome: SSC: Percentage of Participants With Systemic Events Within 7 Days After Booster Dose
Description: Systemic events were recorded in e-diary. Fever: oral temperature greater than or equal to (>=) 38.0 degree Celsius (deg C) and categorized as >=38.0-38.4 deg C, >38.4-38.9 deg C, >38.9-40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity) and Grade 4 (ER visit/hospitalization). Vomiting: mild: 1-2 times in 24 hours (h), moderate: >2 times in 24h, severe: required intravenous hydration and Grade 4: ER visit/hospitalization for hypotensive shock. Diarrhea: mild: 2-3 loose stools in 24 h, moderate: 4-5 loose stools in 24h, severe: 6 or more loose stools in 24h and Grade 4: ER visit/hospitalization for severe diarrhea. Grade 4 were classified by investigator or medically qualified person. Exact 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 up to Day 7 after the booster dose
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 75 | 64
Percentage of participants
  Fever: >=38.0 deg C | 4.0 [0.8 to 11.2] | 6.3 [1.7 to 15.2]
  Fever: >=38.0°C to 38.4 deg C | 2.7 [0.3 to 9.3] | 3.1 [0.4 to 10.8]
  Fever: >38.4°C to 38.9 deg C | 0 [0.0 to 4.8] | 1.6 [0.0 to 8.4]
  Fever: >38.9°C to 40.0 deg C | 1.3 [0.0 to 7.2] | 0 [0.0 to 5.6]
  Fever: >40.0 deg C | 0 [0.0 to 4.8] | 1.6 [0.0 to 8.4]
  Fatigue: Any | 49.3 [37.6 to 61.1] | 54.7 [41.7 to 67.2]
  Fatigue: Mild | 22.7 [13.8 to 33.8] | 25.0 [15.0 to 37.4]
  Fatigue: Moderate | 25.3 [16.0 to 36.7] | 26.6 [16.3 to 39.1]
  Fatigue: Severe | 1.3 [0.0 to 7.2] | 3.1 [0.4 to 10.8]
  Fatigue: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Headache: Any | 41.3 [30.1 to 53.3] | 53.1 [40.2 to 65.7]
  Headache: Mild | 21.3 [12.7 to 32.3] | 31.3 [20.2 to 44.1]
  Headache: Moderate | 20.0 [11.6 to 30.8] | 20.3 [11.3 to 32.2]
  Headache: Severe | 0 [0.0 to 4.8] | 1.6 [0.0 to 8.4]
  Headache: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Chills: Any | 13.3 [6.6 to 23.2] | 23.4 [13.8 to 35.7]
  Chills: Mild | 5.3 [1.5 to 13.1] | 12.5 [5.6 to 23.2]
  Chills: Moderate | 8.0 [3.0 to 16.6] | 10.9 [4.5 to 21.2]
  Chills: Severe | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Chills: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Vomiting: Any | 1.3 [0.0 to 7.2] | 3.1 [0.4 to 10.8]
  Vomiting: Mild | 0 [0.0 to 4.8] | 1.6 [0.0 to 8.4]
  Vomiting: Moderate | 1.3 [0.0 to 7.2] | 1.6 [0.0 to 8.4]
  Vomiting: Severe | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Vomiting: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Diarrhea: Any | 4.0 [0.8 to 11.2] | 9.4 [3.5 to 19.3]
  Diarrhea: Mild | 2.7 [0.3 to 9.3] | 9.4 [3.5 to 19.3]
  Diarrhea: Moderate | 1.3 [0.0 to 7.2] | 0 [0.0 to 5.6]
  Diarrhea: Severe | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  Diarrhea: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  New or worsened muscle pain: Any | 24.0 [14.9 to 35.3] | 37.5 [25.7 to 50.5]
  New or worsened muscle pain: Mild | 4.0 [0.8 to 11.2] | 20.3 [11.3 to 32.2]
  New or worsened muscle pain: Moderate | 20.0 [11.6 to 30.8] | 17.2 [8.9 to 28.7]
  New or worsened muscle pain: Severe | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  New or worsened joint pain: Any | 14.7 [7.6 to 24.7] | 15.6 [7.8 to 26.9]
  New or worsened joint pain: Mild | 5.3 [1.5 to 13.1] | 10.9 [4.5 to 21.2]
  New or worsened joint pain: Moderate | 9.3 [3.8 to 18.3] | 4.7 [1.0 to 13.1]
  New or worsened joint pain: Severe | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 4.8] | 0 [0.0 to 5.6]

22. Primary Outcome: SSC: Percentage of Participants Reporting Adverse Events From Booster Dose Through 1 Month After Booster Dose
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs from booster (third) dose up to 1 month after booster (third) dose were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From booster dose (Day 1) up to 1 month after booster dose
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 75 | 65
Percentage of participants | 4.0 [0.8 to 11.2] | 7.7 [2.5 to 17.0]

23. Primary Outcome: SSC: Percentage of Participants Reporting Serious Adverse Events From Booster Dose Through 6 Months After Booster Dose
Description: as for outcome 18
Time Frame: From booster dose (Day 1) up to 6 months after booster dose
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 75 | 65
Percentage of participants | 0 [0.0 to 4.8] | 1.5 [0.0 to 8.3]

24. Primary Outcome: SSC: Geometric Mean Titers (GMT) of SARS-CoV-2 Reference-Strain-Neutralizing Titers at Baseline
Description: GMT of SARS-CoV-2 reference-strain-neutralizing titers at baseline (before the booster dose) was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: At baseline (pre-dose)
Population: Evaluable immunogenicity population included all eligible randomized participants who received the study intervention to which they are randomized, have valid and determinate immunogenicity result for Visit 303 (1 month after booster dose), have blood sample collected within an appropriate window (within 28-42 days after booster dose), and have no other important protocol deviations as determined by clinician. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 65 | 54
Titer | 1337.2 [941.5 to 1899.2] | 1648.4 [1087.5 to 2498.6]

25. Primary Outcome: SSC: GMT of SARS-CoV-2 Reference-Strain-Neutralizing Titers at 1 Month After the Booster Dose
Description: GMT of SARS-CoV-2 reference-strain-neutralizing titers at 1 month after the booster dose was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: 1 month after the booster dose
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 67 | 54
Titer | 11672.4 [9754.8 to 13967.0] | 15680.7 [13308.9 to 18475.2]

26. Primary Outcome: SSC: Geometric Mean Fold-Rise (GMFR) of SARS-CoV-2 Reference-Strain-Neutralizing Titers From Baseline to 1 Month After the Booster Dose
Description: GMFR of SARS-CoV-2 reference-strain-neutralizing titers from baseline to 1 month after the booster dose received in this sub-study was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From baseline to 1 month after the booster dose
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 65 | 54
Fold rise | 8.6 [6.4 to 11.6] | 9.5 [6.5 to 13.9]

27. Primary Outcome: SSC: Percentage of Participants With Seroresponse to Reference-Strain at 1 Month After the Booster Dose
Description: Seroresponse was defined as achieving >= 4-fold rise from baseline (before the study vaccination). If the baseline measurement is below the lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse at 1 month after the booster dose was reported in this outcome measure.
Time Frame: 1 month after the booster dose
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 65 | 54
Percentage of participants | 67.7 [54.9 to 78.8] | 66.7 [52.5 to 78.9]

28. Primary Outcome: SSD: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions were recorded by participants in e-diary. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu=0.5 centimeter (cm) and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection (inj) site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (emergency room [ER] visit/hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Percentage of participants reporting local reactions after Vaccination 1 and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented.
Time Frame: Day 1 up to Day 7 after Vaccination 1
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'N' signifies participants who received Vaccination 1 and 'Number Analyzed (n)' signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4 | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 188
Percentage of participants
  Redness: Any: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Redness: Any | 3.4 [1.4 to 6.8] | 5.7 [2.9 to 10.0] | 2.5 [0.8 to 5.7] | 7.1 [4.5 to 10.7] | 4.3 [2.3 to 7.2] | 5.4 [2.6 to 9.7]
  Redness: Mild: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Redness: Mild | 1.0 [0.1 to 3.4] | 4.2 [1.8 to 8.0] | 1.0 [0.1 to 3.5] | 4.4 [2.4 to 7.4] | 3.9 [2.1 to 6.8] | 3.2 [1.2 to 6.9]
  Redness: Moderate: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Redness: Moderate | 1.4 [0.3 to 4.2] | 1.6 [0.3 to 4.5] | 1.5 [0.3 to 4.3] | 2.7 [1.2 to 5.3] | 0.3 [0.0 to 1.8] | 2.2 [0.6 to 5.4]
  Redness: Severe: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Redness: Severe | 1.0 [0.1 to 3.4] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Redness: Grade 4: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Redness: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Swelling: Any: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Swelling: Any | 8.2 [4.9 to 12.8] | 7.3 [4.0 to 11.9] | 5.5 [2.8 to 9.6] | 8.5 [5.6 to 12.3] | 8.9 [5.9 to 12.7] | 11.3 [7.1 to 16.7]
  Swelling: Mild: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Swelling: Mild | 4.3 [2.0 to 8.1] | 4.2 [1.8 to 8.0] | 4.5 [2.1 to 8.3] | 5.4 [3.1 to 8.7] | 6.9 [4.3 to 10.4] | 6.5 [3.4 to 11.0]
  Swelling: Moderate: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Swelling: Moderate | 3.9 [1.7 to 7.5] | 2.6 [0.9 to 6.0] | 1.0 [0.1 to 3.5] | 3.1 [1.4 to 5.7] | 2.0 [0.7 to 4.2] | 4.8 [2.2 to 9.0]
  Swelling: Severe: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Swelling: Severe | 0 [0.0 to 1.8] | 0.5 [0.0 to 2.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Swelling: Grade 4: number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
  Swelling: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Injection site pain: Any | 46.4 [39.4 to 53.4] | 42.7 [35.6 to 50.0] | 42.3 [35.4 to 49.4] | 78.2 [73.1 to 82.8] | 78.9 [73.9 to 83.4] | 54.3 [46.8 to 61.5]
  Injection site pain: Mild | 30.9 [24.7 to 37.7] | 27.1 [20.9 to 34.0] | 32.3 [25.9 to 39.3] | 59.2 [53.3 to 64.9] | 61.5 [55.8 to 67.0] | 27.7 [21.4 to 34.6]
  Injection site pain: Moderate | 15.0 [10.4 to 20.6] | 14.1 [9.5 to 19.8] | 9.5 [5.8 to 14.4] | 18.4 [14.1 to 23.3] | 16.4 [12.5 to 21.1] | 26.1 [19.9 to 33.0]
  Injection site pain: Severe | 0.5 [0.0 to 2.7] | 1.6 [0.3 to 4.5] | 0.5 [0.0 to 2.7] | 0.7 [0.1 to 2.4] | 1.0 [0.2 to 2.9] | 0.5 [0.0 to 2.9]
  Injection site pain: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.9]

29. Primary Outcome: SSD: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions were recorded by participants in e-diary. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu =0.5 centimeter (cm) and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Percentage of participants reporting local reactions after Vaccination 2 and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented.
Time Frame: Day 1 up to Day 7 after Vaccination 2
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'N' signifies participants who received Vaccination 2 and 'Number Analyzed (n)' signifies participants evaluable for specified rows and received two doses of study vaccination for SSD. Participants of SSD: Cohort 1: Group 1 did not receive Vaccination 2 and therefore were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 1: Group 2 | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4 | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 157 | 196 | 218 | 142
Percentage of participants
  Redness: Any: number analyzed (Participants) | 157 | 196 | 217 | 140
  Redness: Any | 5.7 [2.7 to 10.6] | 5.1 [2.5 to 9.2] | 4.1 [1.9 to 7.7] | 4.3 [1.6 to 9.1]
  Redness: Mild: number analyzed (Participants) | 157 | 196 | 217 | 140
  Redness: Mild | 4.5 [1.8 to 9.0] | 3.6 [1.4 to 7.2] | 4.1 [1.9 to 7.7] | 2.1 [0.4 to 6.1]
  Redness: Moderate: number analyzed (Participants) | 157 | 196 | 217 | 140
  Redness: Moderate | 1.3 [0.2 to 4.5] | 1.5 [0.3 to 4.4] | 0 [0.0 to 1.7] | 2.1 [0.4 to 6.1]
  Redness: Severe: number analyzed (Participants) | 157 | 196 | 217 | 140
  Redness: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Redness: Grade 4: number analyzed (Participants) | 157 | 196 | 217 | 140
  Redness: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Swelling: Any: number analyzed (Participants) | 157 | 196 | 217 | 141
  Swelling: Any | 8.9 [5.0 to 14.5] | 4.1 [1.8 to 7.9] | 6.5 [3.6 to 10.6] | 9.2 [5.0 to 15.3]
  Swelling: Mild: number analyzed (Participants) | 157 | 196 | 217 | 141
  Swelling: Mild | 7.0 [3.5 to 12.2] | 2.0 [0.6 to 5.1] | 5.5 [2.9 to 9.5] | 5.7 [2.5 to 10.9]
  Swelling: Moderate: number analyzed (Participants) | 157 | 196 | 217 | 141
  Swelling: Moderate | 1.3 [0.2 to 4.5] | 2.0 [0.6 to 5.1] | 0.9 [0.1 to 3.3] | 3.5 [1.2 to 8.1]
  Swelling: Severe: number analyzed (Participants) | 157 | 196 | 217 | 141
  Swelling: Severe | 0.6 [0.0 to 3.5] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Swelling: Grade 4: number analyzed (Participants) | 157 | 196 | 217 | 141
  Swelling: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Injection site pain: Any | 40.1 [32.4 to 48.2] | 74.5 [67.8 to 80.4] | 70.6 [64.1 to 76.6] | 34.5 [26.7 to 42.9]
  Injection site pain: Mild | 29.9 [22.9 to 37.8] | 55.6 [48.4 to 62.7] | 57.8 [50.9 to 64.4] | 21.1 [14.7 to 28.8]
  Injection site pain: Moderate | 10.2 [5.9 to 16.0] | 18.9 [13.7 to 25.1] | 12.4 [8.3 to 17.5] | 13.4 [8.3 to 20.1]
  Injection site pain: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0.5 [0.0 to 2.5] | 0 [0.0 to 2.6]
  Injection site pain | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]

30. Primary Outcome: SSD: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 3
Description: Local reactions were recorded by participants in e-diary. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu =0.5 centimeter (cm) and were graded as mild (> 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person. Percentage of participants reporting local reactions after Vaccination 3 and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented.
Time Frame: Day 1 up to Day 7 after Vaccination 3
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'N' signifies participants who received Vaccination 3. Participants of SSD: Cohort 1: Group 1, Group 2 and SSD Cohort 2: Group 3, Group 4 did not receive Vaccination 3 and therefore were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 154
Percentage of participants
  Redness: Any | 4.5 [1.8 to 9.1]
  Redness: Mild | 1.3 [0.2 to 4.6]
  Redness: Moderate | 3.2 [1.1 to 7.4]
  Redness: Severe | 0 [0.0 to 2.4]
  Redness: Grade 4 | 0 [0.0 to 2.4]
  Swelling: Any | 10.4 [6.1 to 16.3]
  Swelling: Mild | 3.2 [1.1 to 7.4]
  Swelling: Moderate | 7.1 [3.6 to 12.4]
  Swelling: Severe | 0 [0.0 to 2.4]
  Swelling: Grade 4 | 0 [0.0 to 2.4]
  Pain at the injection site: Any | 39.0 [31.2 to 47.1]
  Pain at the injection site: Mild | 19.5 [13.5 to 26.6]
  Pain at the injection site: Moderate | 18.8 [13.0 to 25.9]
  Pain at the injection site: Severe | 0.6 [0.0 to 3.6]
  Pain at the injection site: Grade 4 | 0 [0.0 to 2.4]

31. Primary Outcome: SSD: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events were recorded in e-diary. Fever: oral temperature >= 38.0 deg C, categorized as >=38.0-38.4 deg C, >38.4-38.9 deg C, >38.9-40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity) and Grade 4 (ER visit/hospitalization). Vomiting: mild: 1-2 times in 24 h, moderate: >2 times in 24h, severe: required intravenous hydration and Grade 4: ER visit/hospitalization for hypotensive shock. Diarrhea: mild: 2-3 loose stools in 24h, moderate: 4-5 loose stools in 24h, severe: 6 or more loose stools in 24h and Grade 4: ER visit/hospitalization for severe diarrhea. Grade 4 were classified by investigator or medically qualified person. Exact 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 up to Day 7 after Vaccination 1
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'N' signifies participants who received Vaccination 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4 | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 207 | 192 | 201 | 294 | 304 | 186
Percentage of participants
  Fever: Any | 5.8 [3.0 to 9.9] | 2.6 [0.9 to 6.0] | 5.0 [2.4 to 9.0] | 8.8 [5.9 to 12.7] | 7.2 [4.6 to 10.8] | 4.8 [2.2 to 9.0]
  Fever: >=38.0 deg C to 38.4 deg C | 4.3 [2.0 to 8.1] | 1.6 [0.3 to 4.5] | 2.5 [0.8 to 5.7] | 4.8 [2.6 to 7.9] | 3.9 [2.1 to 6.8] | 1.1 [0.1 to 3.8]
  Fever: >38.4 deg C to 38.9 deg C | 0.5 [0.0 to 2.7] | 0.5 [0.0 to 2.9] | 1.5 [0.3 to 4.3] | 3.4 [1.6 to 6.2] | 3.0 [1.4 to 5.5] | 2.7 [0.9 to 6.2]
  Fever: >38.9 deg C to 40.0 deg C | 1.0 [0.1 to 3.4] | 0.5 [0.0 to 2.9] | 1.0 [0.1 to 3.5] | 0.3 [0.0 to 1.9] | 0.3 [0.0 to 1.8] | 1.1 [0.1 to 3.8]
  Fever: >40.0 deg C | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Fever: Unknown | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0.3 [0.0 to 1.9] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Fatigue: Any | 32.4 [26.0 to 39.2] | 26.6 [20.5 to 33.4] | 28.4 [22.2 to 35.1] | 64.6 [58.9 to 70.1] | 60.5 [54.8 to 66.1] | 39.2 [32.2 to 46.7]
  Fatigue: Mild | 18.8 [13.8 to 24.8] | 14.6 [9.9 to 20.4] | 16.4 [11.6 to 22.3] | 26.5 [21.6 to 32.0] | 29.3 [24.2 to 34.7] | 16.7 [11.6 to 22.8]
  Fatigue: Moderate | 12.6 [8.4 to 17.9] | 12.0 [7.7 to 17.4] | 10.9 [7.0 to 16.1] | 34.7 [29.3 to 40.4] | 28.9 [23.9 to 34.4] | 22.0 [16.3 to 28.7]
  Fatigue: Severe | 1.0 [0.1 to 3.4] | 0 [0.0 to 1.9] | 1.0 [0.1 to 3.5] | 3.4 [1.6 to 6.2] | 2.3 [0.9 to 4.7] | 0.5 [0.0 to 3.0]
  Fatigue: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Headache: Any | 30.9 [24.7 to 37.7] | 27.1 [20.9 to 34.0] | 27.4 [21.3 to 34.1] | 47.6 [41.8 to 53.5] | 45.1 [39.4 to 50.8] | 27.4 [21.1 to 34.4]
  Headache: Mild | 20.3 [15.0 to 26.4] | 15.6 [10.8 to 21.5] | 16.4 [11.6 to 22.3] | 27.2 [22.2 to 32.7] | 25.7 [20.8 to 31.0] | 10.2 [6.3 to 15.5]
  Headache: Moderate | 10.1 [6.4 to 15.1] | 9.4 [5.7 to 14.4] | 10.4 [6.6 to 15.5] | 18.4 [14.1 to 23.3] | 17.4 [13.3 to 22.2] | 16.7 [11.6 to 22.8]
  Headache: Severe | 0.5 [0.0 to 2.7] | 2.1 [0.6 to 5.2] | 0.5 [0.0 to 2.7] | 2.0 [0.8 to 4.4] | 2.0 [0.7 to 4.2] | 0.5 [0.0 to 3.0]
  Headache: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Chills: Any | 15.0 [10.4 to 20.6] | 11.5 [7.3 to 16.8] | 10.4 [6.6 to 15.5] | 31.6 [26.4 to 37.3] | 26.3 [21.5 to 31.6] | 14.0 [9.3 to 19.8]
  Chills: Mild | 10.1 [6.4 to 15.1] | 6.8 [3.7 to 11.3] | 8.0 [4.6 to 12.6] | 13.3 [9.6 to 17.7] | 15.1 [11.3 to 19.7] | 7.0 [3.8 to 11.7]
  Chills: Moderate | 4.3 [2.0 to 8.1] | 4.7 [2.2 to 8.7] | 2.5 [0.8 to 5.7] | 17.0 [12.9 to 21.8] | 10.2 [7.0 to 14.2] | 7.0 [3.8 to 11.7]
  Chills: Severe | 0.5 [0.0 to 2.7] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 1.4 [0.4 to 3.4] | 1.0 [0.2 to 2.9] | 0 [0.0 to 2.0]
  Chills: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Vomiting: Any | 1.0 [0.1 to 3.4] | 2.1 [0.6 to 5.2] | 3.5 [1.4 to 7.0] | 2.7 [1.2 to 5.3] | 1.6 [0.5 to 3.8] | 2.2 [0.6 to 5.4]
  Vomiting: Mild | 1.0 [0.1 to 3.4] | 1.6 [0.3 to 4.5] | 2.5 [0.8 to 5.7] | 2.4 [1.0 to 4.8] | 1.6 [0.5 to 3.8] | 0.5 [0.0 to 3.0]
  Vomiting: Moderate | 0 [0.0 to 1.8] | 0.5 [0.0 to 2.9] | 1.0 [0.1 to 3.5] | 0.3 [0.0 to 1.9] | 0 [0.0 to 1.2] | 1.6 [0.3 to 4.6]
  Vomiting: Severe | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Vomiting: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  Diarrhea: Any | 9.2 [5.6 to 14.0] | 8.3 [4.8 to 13.2] | 6.5 [3.5 to 10.8] | 8.5 [5.6 to 12.3] | 11.5 [8.2 to 15.6] | 8.1 [4.6 to 13.0]
  Diarrhea: Mild | 8.2 [4.9 to 12.8] | 7.8 [4.4 to 12.6] | 5.0 [2.4 to 9.0] | 7.5 [4.7 to 11.1] | 9.2 [6.2 to 13.0] | 3.8 [1.5 to 7.6]
  Diarrhea: Moderate | 1.0 [0.1 to 3.4] | 0.5 [0.0 to 2.9] | 1.5 [0.3 to 4.3] | 1.0 [0.2 to 3.0] | 2.0 [0.7 to 4.2] | 3.8 [1.5 to 7.6]
  Diarrhea: Severe | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.8] | 0.5 [0.0 to 3.0]
  Diarrhea: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  New or worsened muscle pain: Any | 15.5 [10.8 to 21.1] | 16.1 [11.2 to 22.1] | 13.9 [9.5 to 19.5] | 34.0 [28.6 to 39.7] | 28.3 [23.3 to 33.7] | 19.9 [14.4 to 26.4]
  New or worsened muscle pain: Mild | 7.2 [4.1 to 11.7] | 6.8 [3.7 to 11.3] | 7.5 [4.2 to 12.0] | 14.6 [10.8 to 19.2] | 16.8 [12.8 to 21.5] | 6.5 [3.4 to 11.0]
  New or worsened muscle pain: Moderate | 8.2 [4.9 to 12.8] | 9.4 [5.7 to 14.4] | 6.5 [3.5 to 10.8] | 18.7 [14.4 to 23.6] | 10.5 [7.3 to 14.5] | 12.9 [8.4 to 18.6]
  New or worsened muscle pain: Severe | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0.7 [0.1 to 2.4] | 1.0 [0.2 to 2.9] | 0.5 [0.0 to 3.0]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  New or worsened joint pain: Any | 11.1 [7.2 to 16.2] | 13.5 [9.0 to 19.2] | 10.0 [6.2 to 14.9] | 23.5 [18.7 to 28.7] | 15.1 [11.3 to 19.7] | 12.4 [8.0 to 18.0]
  New or worsened joint pain: Mild | 5.3 [2.7 to 9.3] | 6.8 [3.7 to 11.3] | 4.5 [2.1 to 8.3] | 10.2 [7.0 to 14.2] | 7.9 [5.1 to 11.5] | 3.8 [1.5 to 7.6]
  New or worsened joint pain: Moderate | 5.3 [2.7 to 9.3] | 6.3 [3.3 to 10.7] | 5.5 [2.8 to 9.6] | 12.2 [8.7 to 16.5] | 7.2 [4.6 to 10.8] | 8.6 [5.0 to 13.6]
  New or worsened joint pain: Severe | 0.5 [0.0 to 2.7] | 0.5 [0.0 to 2.9] | 0 [0.0 to 1.8] | 1.0 [0.2 to 3.0] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 1.8] | 0 [0.0 to 1.9] | 0 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 2.0]

32. Primary Outcome: SSD: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2
Description: as for outcome 31
Time Frame: Day 1 up to Day 7 after Vaccination 2
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'N' signifies participants who received Vaccination 2 and 'n' signifies participants evaluable for specified rows and received two doses of study vaccination for SSD. Participants of SSD: Cohort 1: Group 1 did not receive Vaccination 2 and therefore were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 1: Group 2 | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4 | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 157 | 197 | 219 | 142
Percentage of participants
  Fever: Any: number analyzed (Participants) | 157 | 196 | 217 | 140
  Fever: Any | 1.3 [0.2 to 4.5] | 5.1 [2.5 to 9.2] | 6.0 [3.2 to 10.0] | 2.1 [0.4 to 6.1]
  Fever:>=38.0 deg C-38.4 deg C: number analyzed (Participants) | 157 | 196 | 217 | 140
  Fever:>=38.0 deg C-38.4 deg C | 0 [0.0 to 2.3] | 2.6 [0.8 to 5.9] | 3.7 [1.6 to 7.1] | 0.7 [0.0 to 3.9]
  Fever:>38.4 deg C-38.9 deg C: number analyzed (Participants) | 157 | 196 | 217 | 140
  Fever:>38.4 deg C-38.9 deg C | 1.3 [0.2 to 4.5] | 1.0 [0.1 to 3.6] | 1.8 [0.5 to 4.7] | 1.4 [0.2 to 5.1]
  Fever:>38.9 deg C-40.0 deg C: number analyzed (Participants) | 157 | 196 | 217 | 140
  Fever:>38.9 deg C-40.0 deg C | 0 [0.0 to 2.3] | 1.0 [0.1 to 3.6] | 0.5 [0.0 to 2.5] | 0 [0.0 to 2.6]
  Fever:>40.0 deg C: number analyzed (Participants) | 157 | 196 | 217 | 140
  Fever:>40.0 deg C | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Fever: Unknown: number analyzed (Participants) | 157 | 196 | 217 | 140
  Fever: Unknown | 0 [0.0 to 2.3] | 0.5 [0.0 to 2.8] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Fatigue: Any: number analyzed (Participants) | 157 | 197 | 219 | 141
  Fatigue: Any | 17.8 [12.2 to 24.7] | 60.9 [53.7 to 67.8] | 54.3 [47.5 to 61.1] | 27.0 [19.8 to 35.1]
  Fatigue: Mild: number analyzed (Participants) | 157 | 197 | 219 | 141
  Fatigue: Mild | 11.5 [6.9 to 17.5] | 27.9 [21.8 to 34.7] | 26.9 [21.2 to 33.3] | 13.5 [8.3 to 20.2]
  Fatigue: Moderate: number analyzed (Participants) | 157 | 197 | 219 | 141
  Fatigue: Moderate | 5.7 [2.7 to 10.6] | 32.0 [25.5 to 39.0] | 25.1 [19.5 to 31.4] | 12.1 [7.2 to 18.6]
  Fatigue: Severe: number analyzed (Participants) | 157 | 197 | 219 | 141
  Fatigue: Severe | 0.6 [0.0 to 3.5] | 1.0 [0.1 to 3.6] | 2.3 [0.7 to 5.2] | 1.4 [0.2 to 5.0]
  Fatigue: Grade 4: number analyzed (Participants) | 157 | 197 | 219 | 141
  Fatigue: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Headache: Any: number analyzed (Participants) | 157 | 196 | 217 | 142
  Headache: Any | 24.8 [18.3 to 32.4] | 39.8 [32.9 to 47.0] | 37.3 [30.9 to 44.1] | 19.7 [13.5 to 27.2]
  Headache: Mild: number analyzed (Participants) | 157 | 196 | 217 | 142
  Headache: Mild | 13.4 [8.5 to 19.7] | 26.5 [20.5 to 33.3] | 18.0 [13.1 to 23.7] | 10.6 [6.0 to 16.8]
  Headache: Moderate: number analyzed (Participants) | 157 | 196 | 217 | 142
  Headache: Moderate | 10.8 [6.4 to 16.8] | 13.3 [8.9 to 18.8] | 17.1 [12.3 to 22.7] | 9.2 [5.0 to 15.1]
  Headache: Severe: number analyzed (Participants) | 157 | 196 | 217 | 142
  Headache: Severe | 0.6 [0.0 to 3.5] | 0 [0.0 to 1.9] | 2.3 [0.8 to 5.3] | 0 [0.0 to 2.6]
  Headache: Grade 4: number analyzed (Participants) | 157 | 196 | 217 | 142
  Headache: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Chills: Any: number analyzed (Participants) | 157 | 197 | 217 | 140
  Chills: Any | 12.1 [7.4 to 18.3] | 21.8 [16.3 to 28.3] | 19.4 [14.3 to 25.2] | 7.1 [3.5 to 12.7]
  Chills: Mild: number analyzed (Participants) | 157 | 197 | 217 | 140
  Chills: Mild | 7.0 [3.5 to 12.2] | 10.7 [6.7 to 15.8] | 12.4 [8.4 to 17.6] | 2.1 [0.4 to 6.1]
  Chills: Moderate: number analyzed (Participants) | 157 | 197 | 217 | 140
  Chills: Moderate | 5.1 [2.2 to 9.8] | 10.7 [6.7 to 15.8] | 6.5 [3.6 to 10.6] | 5.0 [2.0 to 10.0]
  Chills: Severe: number analyzed (Participants) | 157 | 197 | 217 | 140
  Chills: Severe | 0 [0.0 to 2.3] | 0.5 [0.0 to 2.8] | 0.5 [0.0 to 2.5] | 0 [0.0 to 2.6]
  Chills: Grade 4: number analyzed (Participants) | 157 | 197 | 217 | 140
  Chills: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Vomiting: Any: number analyzed (Participants) | 157 | 196 | 217 | 140
  Vomiting: Any | 2.5 [0.7 to 6.4] | 0.5 [0.0 to 2.8] | 1.8 [0.5 to 4.7] | 2.1 [0.4 to 6.1]
  Vomiting: Mild: number analyzed (Participants) | 157 | 196 | 217 | 140
  Vomiting: Mild | 1.9 [0.4 to 5.5] | 0.5 [0.0 to 2.8] | 1.8 [0.5 to 4.7] | 2.1 [0.4 to 6.1]
  Vomiting: Moderate: number analyzed (Participants) | 157 | 196 | 217 | 140
  Vomiting: Moderate | 0.6 [0.0 to 3.5] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Vomiting: Severe: number analyzed (Participants) | 157 | 196 | 217 | 140
  Vomiting: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Vomiting: Grade 4: number analyzed (Participants) | 157 | 196 | 217 | 140
  Vomiting: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Diarrhea: Any: number analyzed (Participants) | 157 | 196 | 217 | 140
  Diarrhea: Any | 5.1 [2.2 to 9.8] | 9.7 [5.9 to 14.7] | 6.0 [3.2 to 10.0] | 6.4 [3.0 to 11.9]
  Diarrhea: Mild: number analyzed (Participants) | 157 | 196 | 217 | 140
  Diarrhea: Mild | 3.8 [1.4 to 8.1] | 8.2 [4.7 to 12.9] | 5.1 [2.6 to 8.9] | 4.3 [1.6 to 9.1]
  Diarrhea: Moderate: number analyzed (Participants) | 157 | 196 | 217 | 140
  Diarrhea: Moderate | 1.3 [0.2 to 4.5] | 1.5 [0.3 to 4.4] | 0.9 [0.1 to 3.3] | 2.1 [0.4 to 6.1]
  Diarrhea: Severe: number analyzed (Participants) | 157 | 196 | 217 | 140
  Diarrhea: Severe | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  Diarrhea: Grade 4: number analyzed (Participants) | 157 | 196 | 217 | 140
  Diarrhea: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  New or worsened muscle pain: Any: number analyzed (Participants) | 157 | 196 | 216 | 140
  New or worsened muscle pain: Any | 10.8 [6.4 to 16.8] | 27.6 [21.4 to 34.4] | 26.7 [21.0 to 33.1] | 8.6 [4.5 to 14.5]
  New or worsened muscle pain: Mild: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened muscle pain: Mild | 5.7 [2.7 to 10.6] | 17.9 [12.8 to 23.9] | 14.7 [10.3 to 20.2] | 4.3 [1.6 to 9.1]
  New or worsened muscle pain: Moderate: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened muscle pain: Moderate | 4.5 [1.8 to 9.0] | 9.7 [5.9 to 14.7] | 11.1 [7.2 to 16.0] | 4.3 [1.6 to 9.1]
  New or worsened muscle pain: Severe: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened muscle pain: Severe | 0.6 [0.0 to 3.5] | 0 [0.0 to 1.9] | 0.9 [0.1 to 3.3] | 0 [0.0 to 2.6]
  New or worsened muscle pain: Grade 4: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  New or worsened joint pain: Any: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened joint pain: Any | 7.6 [4.0 to 13.0] | 14.3 [9.7 to 20.0] | 12.0 [8.0 to 17.1] | 5.7 [2.5 to 10.9]
  New or worsened joint pain: Mild: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened joint pain: Mild | 3.2 [1.0 to 7.3] | 7.1 [4.0 to 11.7] | 6.5 [3.6 to 10.6] | 2.1 [0.4 to 6.1]
  New or worsened joint pain: Moderate: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened joint pain: Moderate | 4.5 [1.8 to 9.0] | 6.1 [3.2 to 10.5] | 5.5 [2.9 to 9.5] | 3.6 [1.2 to 8.1]
  New or worsened joint pain: Severe: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened joint pain: Severe | 0 [0.0 to 2.3] | 1.0 [0.1 to 3.6] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]
  New or worsened joint pain: Grade 4: number analyzed (Participants) | 157 | 196 | 217 | 140
  New or worsened joint pain: Grade 4 | 0 [0.0 to 2.3] | 0 [0.0 to 1.9] | 0 [0.0 to 1.7] | 0 [0.0 to 2.6]

33. Primary Outcome: SSD: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 3
Description: Systemic events were recorded in e-diary. Fever: oral temperature >= 38.0 deg C and categorized as >=38.0-38.4 deg C, >38.4-38.9 deg C, >38.9-40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity) and Grade 4 (ER visit/hospitalization). Vomiting: mild: 1-2 times in 24 hours (h), moderate: >2 times in 24h, severe: required intravenous hydration and Grade 4: ER visit/hospitalization for hypotensive shock. Diarrhea: mild: 2-3 loose stools in 24h, moderate: 4-5 loose stools in 24h, severe: 6 or more loose stools in 24h and Grade 4: ER visit/hospitalization for severe diarrhea. Grade 4 were classified by investigator or medically qualified person. Exact 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 up to Day 7 after Vaccination 3
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'N'= participants who received vaccination 3. Participants of SSD: Cohort 1: Group 1, Group 2 and SSD Cohort 2: Group 3, Group 4 did not receive Vaccination 3 and therefore were not analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 154
Percentage of participants
  Fever: Any | 2.6 [0.7 to 6.5]
  Fever: >=38.0 deg C to 38.4 deg C | 0.6 [0.0 to 3.6]
  Fever: >38.4 deg C to 38.9 deg C | 1.3 [0.2 to 4.6]
  Fever: >38.9 deg C to 40.0 deg C | 0.6 [0.0 to 3.6]
  Fever: >40.0 deg C | 0 [0.0 to 2.4]
  Fatigue: Any | 22.7 [16.4 to 30.2]
  Fatigue: Mild | 3.9 [1.4 to 8.3]
  Fatigue: Moderate | 18.2 [12.4 to 25.2]
  Fatigue: Severe | 0.6 [0.0 to 3.6]
  Fatigue: Grade 4 | 0 [0.0 to 2.4]
  Headache: Any | 25.3 [18.7 to 33.0]
  Headache: Mild | 9.1 [5.1 to 14.8]
  Headache: Moderate | 14.9 [9.7 to 21.6]
  Headache: Severe | 1.3 [0.2 to 4.6]
  Headache: Grade 4 | 0 [0.0 to 2.4]
  Chills: Any | 9.1 [5.1 to 14.8]
  Chills: Mild | 4.5 [1.8 to 9.1]
  Chills: Moderate | 3.2 [1.1 to 7.4]
  Chills: Severe | 1.3 [0.2 to 4.6]
  Chills: Grade 4 | 0 [0.0 to 2.4]
  Vomiting: Any | 2.6 [0.7 to 6.5]
  Vomiting: Mild | 1.3 [0.2 to 4.6]
  Vomiting: Moderate | 1.3 [0.2 to 4.6]
  Vomiting: Severe | 0 [0.0 to 2.4]
  Vomiting: Grade 4 | 0 [0.0 to 2.4]
  Diarrhea: Any | 1.9 [0.4 to 5.6]
  Diarrhea: Mild | 1.3 [0.2 to 4.6]
  Diarrhea: Moderate | 0.6 [0.0 to 3.6]
  Diarrhea: Severe | 0 [0.0 to 2.4]
  Diarrhea: Grade 4 | 0 [0.0 to 2.4]
  New or worsened muscle pain: Any | 14.9 [9.7 to 21.6]
  New or worsened muscle pain: Mild | 4.5 [1.8 to 9.1]
  New or worsened muscle pain: Moderate | 10.4 [6.1 to 16.3]
  New or worsened muscle pain: Severe | 0 [0.0 to 2.4]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 2.4]
  New or worsened joint pain: Any | 9.1 [5.1 to 14.8]
  New or worsened joint pain: Mild | 3.2 [1.1 to 7.4]
  New or worsened joint pain: Moderate | 5.2 [2.3 to 10.0]
  New or worsened joint pain: Severe | 0.6 [0.0 to 3.6]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 2.4]

34. Primary Outcome: SSD: Percentage of Participants Reporting Adverse Events (AEs) From First Study Vaccination (Day 1) Through 1 Month After Last Study Vaccination: Cohort 1
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs from first study vaccination (Day 1) up to 1 month after last study vaccination were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From Day 1 up to 1 month after last study vaccination
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b
Number analyzed (Participants) | 216 | 197 | 204
Percentage of participants | 3.2 [1.3 to 6.6] | 6.1 [3.2 to 10.4] | 2.0 [0.5 to 4.9]

35. Primary Outcome: SSD: Percentage of Participants Reporting Adverse Events (AEs) From First Study Vaccination (Day 1) Through 1 Month After Vaccination 1: Cohort 2
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs from first study vaccination (Day 1) up to 1 month after Vaccination 1 were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From first study vaccination (Day 1) up to 1 month after Vaccination 1
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4
Number analyzed (Participants) | 315 | 323
Percentage of participants | 4.1 [2.2 to 7.0] | 3.7 [1.9 to 6.4]

36. Primary Outcome: SSD: Percentage of Participants Reporting Adverse Events (AEs) From Second Study Vaccination Through 1 Month After Second Study Vaccination: Cohort 2
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs from Vaccination 2 up to 1 month after Vaccination 2 were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From Vaccination 2 up to 1 month after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure and received two doses of study vaccination for SSD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4
Number analyzed (Participants) | 213 | 238
Percentage of participants | 2.3 [0.8 to 5.4] | 3.8 [1.7 to 7.1]

37. Primary Outcome: SSD: Percentage of Participants Reporting Adverse Events (AEs) From First Study Vaccination (Day 1) Through 1 Month After Second Study Vaccination: Cohort 3
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs from first study vaccination (Day 1) up to 1 month after Vaccination 2 were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From first study vaccination (Day 1) up to 1 month after Vaccination 2
Population: as for outcome 36
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 210
Percentage of participants | 6.7 [3.7 to 10.9]

38. Primary Outcome: SSD: Percentage of Participants Reporting Adverse Events (AEs) From Third Study Vaccination Through 1 Month After Third Study Vaccination: Cohort 3
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs from Vaccination 3 up to 1 month after Vaccination 3 were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From Vaccination 3 up to 1 month after Vaccination 3
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure and received three doses of study vaccination for SSD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 172
Percentage of participants | 0.6 [0.0 to 3.2]

39. Primary Outcome: SSD: Percentage of Participants Reporting Serious Adverse Events (SAEs) From First Study Vaccination (Day 1) Through 6 Months After Last Study Vaccination: Cohort 1 and Cohort 3
Description: A SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening; resulted in persistent disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required inpatient hospitalization or prolongation of existing hospitalization. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: From first study vaccination (Day 1) up to 6 months after last study vaccination
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b | SSD: Cohort 3: Group 5
Number analyzed (Participants) | 216 | 197 | 204 | 210
Percentage of participants | 0.9 [0.1 to 3.3] | 1.5 [0.3 to 4.4] | 1.0 [0.1 to 3.5] | 3.8 [1.7 to 7.4]

40. Primary Outcome: SSD: Percentage of Participants Reporting SAEs From First Study Vaccination (Day 1) Through 6 Months After Vaccination 1 (For Participants Who Received 1 Dose Only) and up to Vaccination 2 (For Participants Who Received 2 Doses): Cohort 2
Description: as for outcome 39
Time Frame: From vaccination 1 (Day 1) up to 6 months after vaccination 1 (participants received 1 dose only); From vaccination 1 up to before vaccination 2 (participants received 2 doses)
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4
Number analyzed (Participants) | 315 | 323
Percentage of participants | 1.6 [0.5 to 3.7] | 0.6 [0.1 to 2.2]

41. Primary Outcome: SSD: Percentage of Participants Reporting Serious Adverse Events (SAEs) From First Study Vaccination Through 6 Months After Vaccination 2: Cohort 2
Description: as for outcome 39
Time Frame: From first study vaccination (Day 1) up to 6 months after vaccination 2
Population: as for outcome 36
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4
Number analyzed (Participants) | 213 | 238
Percentage of participants | 0.5 [0.0 to 2.6] | 1.3 [0.3 to 3.6]

42. Primary Outcome: SSD: GMR Based on Geometric Mean Titers of SARS-CoV-2 Omicron BA.1 Strain Neutralizing Titers 1 Month After First Study Vaccination: Comparison Between Cohort 2 Group 3 and Group 4
Description: GMR was calculated based on GMT levels of SSD: Cohort 2: Group 3 and SSD: Cohort 2: Group 4 and reported in statistical analysis section below. GMT of SARS-CoV-2 Omicron strain-neutralizing titers and reported in statistical analysis. GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers at 1 month after first study vaccination was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: 1 month after Vaccination 1
Population: Evaluable immunogenicity population (EIP) included all eligible randomized participants who received 1st study intervention to which they were randomized (Group 3, 4), had valid determinate immunogenicity result from blood sample collected within 28-42 days after 1st study vaccination (Group 3, 4), have no other important protocol deviations as determined by clinician. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4
Number analyzed (Participants) | 132 | 141
Titer | 1929.2 [1631.5 to 2281.1] | 1099.6 [932.0 to 1297.4]
Statistical Analysis 1: Comparison: SSD: Cohort 2: Group 3 vs SSD: Cohort 2: Group 4; GMRs and 2-sided 95% CIs were calculated by exponentiating the mean difference of the logarithms of the titers (BNT162b2 OMI [30 mcg] - BNT162b2 [30 μg]) and the corresponding CI (based on the student t distribution); Test type: Other; Geometric Mean Ration (GMR) = 1.75, 95% CI 2-sided [1.39 to 2.22]

43. Primary Outcome: SSD: Percentage of Participants With Seroresponse to the SARS-CoV-2 Omicron BA.1 Strain at 1 Month After First Study Vaccination: Comparison Between Cohort 2 Group 3 and Group 4
Description: Seroresponse: achieving >= 4-fold rise from baseline (before study vaccination). If baseline measurement is below the lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse 1 month after first study vaccination was reported in this outcome measure.
Time Frame: 1 month after Vaccination 1
Population: Evaluable immunogenicity population (EIP) included all eligible randomized participants who received 1st study intervention to which they were randomized (Group 3, 4), had valid determinate immunogenicity result from blood sample collected within 28-42 days after 1st study vaccination (Group 3, 4), had no other important protocol deviations as determined by clinician. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 2: Group 3 | SSD: Cohort 2: Group 4
Number analyzed (Participants) | 130 | 140
Percentage of participants | 62.3 [53.4 to 70.7] | 39.3 [31.1 to 47.9]
Statistical Analysis 1: Comparison: SSD: Cohort 2: Group 3 vs SSD: Cohort 2: Group 4; Difference in proportions, expressed as a percentage (BNT162b2 OMI [30 mcg] - BNT162b2 [30 mcg]). 2-Sided CI based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Other; Difference in Percentages = 23.0, 95% CI 2-sided [11.1 to 34.3]

44. Primary Outcome: SSD: GMR Based on Geometric Mean Titers of SARS-CoV-2 Omicron BA.1 Strain Neutralizing Titers 1 Month After First Study Vaccination: Comparison Between Cohort 1 Group 1 and Group 2b
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers at 1 month after first study vaccination was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: 1 month after Vaccination 1
Population: Evaluable immunogenicity population (EIP) included all eligible randomized participants who received 1st study intervention to which they were randomized (Groups 1, 2b), had valid determinate immunogenicity result from blood sample collected within 28-42 days after 1st study vaccination (Groups 1, 2b), have no other important protocol deviations as determined by clinician. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2b
Number analyzed (Participants) | 100 | 100
Titer | 5094.1 [4118.2 to 6301.2] | 1775.6 [1484.8 to 2123.4]
Statistical Analysis 1: Comparison: SSD: Cohort 1: Group 1 vs SSD: Cohort 1: Group 2b; [analysis description as in outcome 42, analysis 1]; Test type: Other; Geometric Mean Ration (GMR) = 2.87, 95% CI 2-sided [2.18 to 3.78]

45. Primary Outcome: SSD: GMR Based on Geometric Mean Titers of SARS-CoV-2 Omicron BA.1 Strain Neutralizing Titers: Comparison Between 1 Month After Second Study Vaccination for Cohort 1 Group 2 and 1 Month After First Study Vaccination for Cohort 1 Group 2b
Description: GMR was calculated based on GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers at 1 month after Vaccination 2 for Group 2 and 1 month after Vaccination 1 for Group 2b was reported. GMTs and corresponding 2-sided CIs were calculated by exponentiating mean logarithm of titers and corresponding CIs (based on Student's t distribution).
Time Frame: For Cohort 1 Group 2b:1 month after Vaccination 1; for Cohort 1 Group 2: 1 month after Vaccination 2
Population: EIP: all eligible participants received 1st study drug as randomized (Group 2b) or received 2 doses of study drug as randomized with Dose 2 received within 19-42 days after Dose1 (Group 2), had valid determinate immunogenicity result from blood sample collected within 28-42 days after 1st study vaccination (Group 2b) or 28-42 days after 2nd study vaccination (Group 2), had no other important protocol deviations as determined by clinician. Here 'N'=participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b
Number analyzed (Participants) | 100 | 100
Titer | 4684.3 [3937.4 to 5573.0] | 1775.6 [1484.8 to 2123.4]
Statistical Analysis 1: Comparison: SSD: Cohort 1: Group 2 vs SSD: Cohort 1: Group 2b; [analysis description as in outcome 42, analysis 1]; Test type: Other; Geometric Mean Ratio (GMR) = 2.64, 95% CI 2-sided [2.06 to 3.38]

46. Primary Outcome: Percentage of Participants With Seroresponse to the SARS-CoV-2 Omicron BA.1 Strain at 1 Month After First Study Vaccination: Comparison Between Cohort 1 Group 1 and Group 2b
Description: Seroresponse: achieving >= 4-fold rise from baseline (before study vaccination). If baseline measurement is below lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse 1 month after first study vaccination was reported in this outcome measure.
Time Frame: 1 month after Vaccination 1
Population: Evaluable immunogenicity population included all eligible randomized participants who received 1st study intervention to which they were randomized (Group 1, 2b), had valid determinate immunogenicity result from blood sample collected within 28-42 days after 1st study vaccination (Group 1, 2b), had no other important protocol deviations as determined by clinician. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2b
Number analyzed (Participants) | 100 | 100
Percentage of participants | 88.0 [80.0 to 93.6] | 59.0 [48.7 to 68.7]
Statistical Analysis 1: Comparison: SSD: Cohort 1: Group 1 vs SSD: Cohort 1: Group 2b; [analysis description as in outcome 43, analysis 1]; Test type: Other; Difference in Percentages = 29.0, 95% CI 2-sided [17.2 to 40.3]

47. Primary Outcome: SSD: Percentage of Participants With Seroresponse to SARS-CoV-2 Omicron BA.1 Strain at 1 Month After Vaccination 2: Comparison Between 1 Month After Vaccination 2 for Cohort 1 Group 2 and 1 Month After Vaccination 1 for Cohort 1 Group 2b
Description: Seroresponse: achieving >= 4-fold rise from baseline (before study vaccination). If baseline measurement is below LLOQ, postvaccination measure of >= 4 × LLOQ is considered seroresponse. Exact 2-sided CI, based on Clopper and Pearson method was used. Percentage of participants achieving seroresponse 1 month after second study vaccination for Group 2 and 1 month after study vaccination for Group 2b was reported in this outcome measure.
Time Frame: For Cohort 1 Group 2b:1 month after Vaccination 1; for Cohort 1 Group 2: 1 month after Vaccination 2
Population: as for outcome 45
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 1: Group 2 | SSD: Cohort 1: Group 2b
Number analyzed (Participants) | 100 | 100
Percentage of participants | 80.0 [70.8 to 87.3] | 59.0 [48.7 to 68.7]
Statistical Analysis 1: Comparison: SSD: Cohort 1: Group 2 vs SSD: Cohort 1: Group 2b; [analysis description as in outcome 43, analysis 1]; Test type: Other; Difference in Percentages = 21.0, 95% CI 2-sided [8.3 to 33.2]

48. Primary Outcome: SSD: GMR Based on Geometric Mean Titers of SARS-CoV-2 Omicron BA.1 Strain Neutralizing Titers 1 Month After Second Study Vaccination: Cohort 3
Description: GMR calculated based on GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMR comparison between GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers of participants of SSD Cohort 3: Group 5 to GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers of participants of study C4591001 (NCT04368728) Phase 3 BNT162b2 single arm 18-55 years of age, at 1 month after vaccination 2 was reported. GMTs and corresponding 2-sided CIs were calculated by exponentiating mean logarithm of titers and corresponding CIs (student's t distribution).
Time Frame: 1 month after Vaccination 2
Population: EIP:eligible participants received 2 doses of study drug as randomized with Dose2 received within 19-42 days after Dose1 (SSD Cohort 3:Group 5), had valid determinate immunogenicity result from blood sample collected within 28-42 days after 2nd study vaccination, had no other important protocol deviations as determined by clinician. Data of eligible participants from Study C4591001 Phase 3 BNT162b2 single arm 18-55 years was included for comparison.'N'=participants evaluable for outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- C4591001 Study Cohort: Data of evaluable participants from Study C4591001 (NCT04368728) Phase 3 BNT162b2 single arm 18-55 years of age who had received 2 doses of BNT162b2 30 mcg in study C4591001 was included for this comparison.
Arm/Group | SSD: Cohort 3: Group 5 | C4591001 Study Cohort
Number analyzed (Participants) | 152 | 157
Titer | 2892.2 [2522.3 to 3316.3] | 290.6 [241.2 to 350.1]
Statistical Analysis 1: Comparison: SSD: Cohort 3: Group 5 vs C4591001 Study Cohort; [analysis description as in outcome 42, analysis 1]; Test type: Other; Geometric Mean Ration (GMR) = 9.95, 95% CI 2-sided [7.90 to 12.53]

49. Primary Outcome: SSD: Percentage of Participants With Seroresponse to the SARS-CoV-2 Omicron BA.1 Strain at 1 Month After Second Study Vaccination: Cohort 3
Description: EIP:eligible participants received 2 doses of study drug as randomized with Dose2 received within 19-42 days after Dose1 (SSD Cohort 3:Group 5), had valid determinate immunogenicity result from blood sample collected within 28-42 days after 2nd study vaccination, had no other important protocol deviations as determined by clinician. Data of eligible participants from Study C4591001 Phase 3 BNT162b2 single arm 18-55 years was included for comparison.'N'=participants evaluable for outcome measure.
Time Frame: 1 month after Vaccination 2
Population: as for outcome 48
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSD: Cohort 3: Group 5 | C4591001 Study Cohort
Number analyzed (Participants) | 152 | 156
Percentage of participants | 86.2 [79.7 to 91.2] | 80.8 [73.7 to 86.6]
Statistical Analysis 1: Comparison: SSD: Cohort 3: Group 5 vs C4591001 Study Cohort; [analysis description as in outcome 43, analysis 1]; Test type: Other; Difference in Percentages = 5.4, 95% CI 2-sided [-3.0 to 13.8]

50. Primary Outcome: SSE: Percentage of Participants With Local Reactions Within 7 Days After Study Vaccination
Description: Local reactions were recorded by participants in e-diary. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu=0.5 centimeter (cm) and were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm),severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis/exfoliative dermatitis [redness]).Pain at injection site was graded as mild (did not interfere with activity),moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (emergency room [ER] visit/hospitalization for severe pain). Grade 4 were classified by investigator or medically qualified person. Percentage of participants reporting local reactions within 7 days after study vaccination and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented.
Time Frame: Day 1 up to Day 7 after study vaccination
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'Number of Participants Analyzed (N)' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg
Number analyzed (Participants) | 30 | 30 | 30 | 480 | 158 | 320 | 20 | 20 | 20 | 20 | 20 | 20 | 298 | 298 | 301 | 301 | 301 | 312
Percentage of participants
  Redness: Any | 6.7 [0.8 to 22.1] | 0 [0.0 to 11.6] | 6.7 [0.8 to 22.1] | 8.1 [5.8 to 10.9] | 6.3 [3.1 to 11.3] | 10.9 [7.7 to 14.9] | 0 [0.0 to 16.8] | 15.0 [3.2 to 37.9] | 20.0 [5.7 to 43.7] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.8] | 10.0 [1.2 to 31.7] | 6.4 [3.9 to 9.8] | 10.4 [7.2 to 14.4] | 6.3 [3.8 to 9.7] | 10.6 [7.4 to 14.7] | 7.0 [4.4 to 10.5] | 7.4 [4.7 to 10.9]
  Redness: Mild | 6.7 [0.8 to 22.1] | 0 [0.0 to 11.6] | 6.7 [0.8 to 22.1] | 3.8 [2.2 to 5.9] | 4.4 [1.8 to 8.9] | 6.3 [3.9 to 9.5] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 10.0 [1.2 to 31.7] | 4.0 [2.1 to 6.9] | 6.0 [3.6 to 9.4] | 3.3 [1.6 to 6.0] | 4.0 [2.1 to 6.9] | 4.3 [2.3 to 7.3] | 3.5 [1.8 to 6.2]
  Redness: Moderate | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 4.2 [2.6 to 6.4] | 1.9 [0.4 to 5.4] | 4.4 [2.4 to 7.2] | 0 [0.0 to 16.8] | 10.0 [1.2 to 31.7] | 15.0 [3.2 to 37.9] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 2.0 [0.7 to 4.3] | 4.0 [2.1 to 6.9] | 2.7 [1.2 to 5.2] | 6.6 [4.1 to 10.1] | 2.7 [1.2 to 5.2] | 3.2 [1.5 to 5.8]
  Redness: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0.2 [0.0 to 1.2] | 0 [0.0 to 2.3] | 0.3 [0.0 to 1.7] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0.3 [0.0 to 1.9] | 0.3 [0.0 to 1.9] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0.6 [0.1 to 2.3]
  Redness: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Swelling: Any | 0 [0.0 to 11.6] | 6.7 [0.8 to 22.1] | 20.0 [7.7 to 38.6] | 9.6 [7.1 to 12.6] | 7.0 [3.5 to 12.1] | 11.9 [8.5 to 15.9] | 0 [0.0 to 16.8] | 10.0 [1.2 to 31.7] | 15.0 [3.2 to 37.9] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 6.0 [3.6 to 9.4] | 13.1 [9.5 to 17.5] | 8.3 [5.4 to 12.0] | 10.0 [6.8 to 13.9] | 6.6 [4.1 to 10.1] | 5.4 [3.2 to 8.6]
  Swelling: Mild | 0 [0.0 to 11.6] | 6.7 [0.8 to 22.1] | 13.3 [3.8 to 30.7] | 5.0 [3.2 to 7.3] | 4.4 [1.8 to 8.9] | 6.3 [3.9 to 9.5] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 10.0 [1.2 to 31.7] | 3.4 [1.6 to 6.1] | 7.7 [5.0 to 11.4] | 5.0 [2.8 to 8.1] | 4.0 [2.1 to 6.9] | 4.7 [2.6 to 7.7] | 2.9 [1.3 to 5.4]
  Swelling: Moderate | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 6.7 [0.8 to 22.1] | 4.4 [2.7 to 6.6] | 2.5 [0.7 to 6.4] | 5.3 [3.1 to 8.4] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 2.7 [1.2 to 5.2] | 5.4 [3.1 to 8.6] | 3.3 [1.6 to 6.0] | 5.3 [3.1 to 8.5] | 2.0 [0.7 to 4.3] | 2.2 [0.9 to 4.6]
  Swelling: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0.2 [0.0 to 1.2] | 0 [0.0 to 2.3] | 0.3 [0.0 to 1.7] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0.7 [0.1 to 2.4] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.8]
  Swelling: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Pain at the injection site: Any | 90.0 [73.5 to 97.9] | 83.3 [65.3 to 94.4] | 96.7 [82.8 to 99.9] | 82.9 [79.2 to 86.2] | 81.0 [74.0 to 86.8] | 86.3 [82.0 to 89.8] | 70.0 [45.7 to 88.1] | 70.0 [45.7 to 88.1] | 65.0 [40.8 to 84.6] | 100.0 [83.2 to 100.0] | 65.0 [40.8 to 84.6] | 85.0 [62.1 to 96.8] | 60.1 [54.3 to 65.7] | 71.1 [65.6 to 76.2] | 66.1 [60.5 to 71.4] | 70.8 [65.3 to 75.8] | 58.1 [52.3 to 63.8] | 67.9 [62.5 to 73.1]
  Pain at the injection site: Mild | 60.0 [40.6 to 77.3] | 76.7 [57.7 to 90.1] | 33.3 [17.3 to 52.8] | 55.2 [50.6 to 59.7] | 67.7 [59.8 to 74.9] | 45.3 [39.8 to 50.9] | 55.0 [31.5 to 76.9] | 65.0 [40.8 to 84.6] | 55.0 [31.5 to 76.9] | 75.0 [50.9 to 91.3] | 60.0 [36.1 to 80.9] | 45.0 [23.1 to 68.5] | 51.7 [45.8 to 57.5] | 53.4 [47.5 to 59.1] | 52.8 [47.0 to 58.6] | 44.9 [39.1 to 50.7] | 52.8 [47.0 to 58.6] | 55.4 [49.7 to 61.0]
  Pain at the injection site: Moderate | 30.0 [14.7 to 49.4] | 6.7 [0.8 to 22.1] | 60.0 [40.6 to 77.3] | 26.0 [22.2 to 30.2] | 13.3 [8.4 to 19.6] | 39.4 [34.0 to 45.0] | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 25.0 [8.7 to 49.1] | 5.0 [0.1 to 24.9] | 40.0 [19.1 to 63.9] | 8.1 [5.2 to 11.7] | 17.4 [13.3 to 22.2] | 13.3 [9.7 to 17.7] | 25.2 [20.4 to 30.6] | 5.0 [2.8 to 8.1] | 12.2 [8.8 to 16.3]
  Pain at the injection site: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 3.3 [0.1 to 17.2] | 1.7 [0.7 to 3.3] | 0 [0.0 to 2.3] | 1.6 [0.5 to 3.6] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0.3 [0.0 to 1.9] | 0.3 [0.0 to 1.9] | 0 [0.0 to 1.2] | 0.7 [0.1 to 2.4] | 0.3 [0.0 to 1.8] | 0.3 [0.0 to 1.8]
  Pain at the injection site: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]

51. Primary Outcome: SSE: Percentage of Participants With Systemic Events Within 7 Days After Study Vaccination
Description: Systemic events were recorded in e-diary. Fever: oral temperature greater than or equal to 38.0 deg C and categorized as >=38.0-38.4 deg C, >38.4-38.9 deg C, >38.9-40.0 deg C & >40.0 deg C. Fatigue, headache, chills, muscle pain and joint pain: mild (did not interfere with activity), moderate (some interference with activity), severe (prevented daily routine activity) and Grade 4 (ER visit or hospitalization). Vomiting: mild: 1-2 times in 24 h, moderate: > 2 times in 24h, severe: required intravenous hydration and Grade 4: ER or hospitalization for hypotensive shock. Diarrhea: mild: 2-3 loose stools in 24h, moderate: 4-5 loose stools in 24h, severe: 6 or more loose stools in 24h and Grade 4: ER visit or hospitalization for severe diarrhea. Grade 4 were classified by investigator or medically qualified person. Exact 95% CI was based on Clopper and Pearson method.
Time Frame: Day 1 up to Day 7 after study vaccination
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg
Number analyzed (Participants) | 30 | 30 | 30 | 480 | 158 | 320 | 20 | 20 | 20 | 20 | 20 | 20 | 298 | 298 | 301 | 301 | 301 | 312
Percentage of participants
  Fever: >= 38.0 deg C | 13.3 [3.8 to 30.7] | 0 [0.0 to 11.6] | 10.0 [2.1 to 26.5] | 10.0 [7.5 to 13.0] | 10.8 [6.4 to 16.7] | 19.4 [15.2 to 24.1] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 20.0 [5.7 to 43.7] | 20.0 [5.7 to 43.7] | 3.7 [1.9 to 6.5] | 7.4 [4.7 to 11.0] | 8.3 [5.4 to 12.0] | 9.0 [6.0 to 12.8] | 5.0 [2.8 to 8.1] | 7.7 [5.0 to 11.2]
  Fever: >= 38.0 deg C to 38.4 deg C | 3.3 [0.1 to 17.2] | 0 [0.0 to 11.6] | 10.0 [2.1 to 26.5] | 4.2 [2.6 to 6.4] | 6.3 [3.1 to 11.3] | 6.9 [4.4 to 10.2] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 15.0 [3.2 to 37.9] | 5.0 [0.1 to 24.9] | 2.0 [0.7 to 4.3] | 3.7 [1.9 to 6.5] | 3.7 [1.8 to 6.4] | 4.7 [2.6 to 7.7] | 3.7 [1.8 to 6.4] | 5.4 [3.2 to 8.6]
  Fever: >38.4 deg C to 38.9 deg C | 10.0 [2.1 to 26.5] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 3.8 [2.2 to 5.9] | 3.8 [1.4 to 8.1] | 8.1 [5.4 to 11.7] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 1.7 [0.5 to 3.9] | 3.7 [1.9 to 6.5] | 3.7 [1.8 to 6.4] | 2.7 [1.2 to 5.2] | 0 [0.0 to 1.2] | 1.6 [0.5 to 3.7]
  Fever: >38.9 deg C to 40.0 deg C | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 2.1 [1.0 to 3.8] | 0.6 [0.0 to 3.5] | 4.4 [2.4 to 7.2] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 1.0 [0.2 to 2.9] | 1.3 [0.4 to 3.4] | 1.3 [0.4 to 3.4] | 0.6 [0.1 to 2.3]
  Fever: >40 deg C | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Fatigue: Any | 66.7 [47.2 to 82.7] | 63.3 [43.9 to 80.1] | 70.0 [50.6 to 85.3] | 73.8 [69.6 to 77.6] | 68.4 [60.5 to 75.5] | 77.5 [72.5 to 82.0] | 45.0 [23.1 to 68.5] | 55.0 [31.5 to 76.9] | 45.0 [23.1 to 68.5] | 65.0 [40.8 to 84.6] | 40.0 [19.1 to 63.9] | 70.0 [45.7 to 88.1] | 45.3 [39.6 to 51.1] | 52.3 [46.5 to 58.1] | 52.5 [46.7 to 58.3] | 58.8 [53.0 to 64.4] | 49.2 [43.4 to 55.0] | 57.4 [51.7 to 62.9]
  Fatigue: Mild | 20.0 [7.7 to 38.6] | 26.7 [12.3 to 45.9] | 23.3 [9.9 to 42.3] | 25.2 [21.4 to 29.3] | 32.3 [25.1 to 40.2] | 25.9 [21.2 to 31.1] | 30.0 [11.9 to 54.3] | 15.0 [3.2 to 37.9] | 10.0 [1.2 to 31.7] | 35.0 [15.4 to 59.2] | 15.0 [3.2 to 37.9] | 45.0 [23.1 to 68.5] | 23.5 [18.8 to 28.7] | 22.5 [17.9 to 27.7] | 20.3 [15.9 to 25.3] | 24.6 [19.8 to 29.9] | 29.2 [24.2 to 34.7] | 27.2 [22.4 to 32.5]
  Fatigue: Moderate | 43.3 [25.5 to 62.6] | 33.3 [17.3 to 52.8] | 40.0 [22.7 to 59.4] | 44.0 [39.5 to 48.5] | 34.8 [27.4 to 42.8] | 46.9 [41.3 to 52.5] | 10.0 [1.2 to 31.7] | 40.0 [19.1 to 63.9] | 35.0 [15.4 to 59.2] | 30.0 [11.9 to 54.3] | 25.0 [8.7 to 49.1] | 25.0 [8.7 to 49.1] | 21.5 [17.0 to 26.6] | 26.8 [21.9 to 32.3] | 29.6 [24.5 to 35.1] | 30.6 [25.4 to 36.1] | 18.3 [14.1 to 23.1] | 28.2 [23.3 to 33.5]
  Fatigue: Severe | 3.3 [0.1 to 17.2] | 3.3 [0.1 to 17.2] | 6.7 [0.8 to 22.1] | 4.6 [2.9 to 6.9] | 1.3 [0.2 to 4.5] | 4.7 [2.6 to 7.6] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0.3 [0.0 to 1.9] | 3.0 [1.4 to 5.7] | 2.7 [1.2 to 5.2] | 3.7 [1.8 to 6.4] | 1.7 [0.5 to 3.8] | 1.9 [0.7 to 4.1]
  Fatigue: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Headache: Any | 46.7 [28.3 to 65.7] | 30.0 [14.7 to 49.4] | 60.0 [40.6 to 77.3] | 53.5 [49.0 to 58.1] | 50.0 [42.0 to 58.0] | 57.5 [51.9 to 63.0] | 20.0 [5.7 to 43.7] | 30.0 [11.9 to 54.3] | 35.0 [15.4 to 59.2] | 15.0 [3.2 to 37.9] | 30.0 [11.9 to 54.3] | 50.0 [27.2 to 72.8] | 26.5 [21.6 to 31.9] | 38.9 [33.4 to 44.7] | 36.5 [31.1 to 42.3] | 36.5 [31.1 to 42.3] | 33.6 [28.2 to 39.2] | 36.5 [31.2 to 42.1]
  Headache: Mild | 40.0 [22.7 to 59.4] | 23.3 [9.9 to 42.3] | 26.7 [12.3 to 45.9] | 27.7 [23.7 to 31.9] | 29.1 [22.2 to 36.9] | 27.5 [22.7 to 32.7] | 10.0 [1.2 to 31.7] | 30.0 [11.9 to 54.3] | 30.0 [11.9 to 54.3] | 10.0 [1.2 to 31.7] | 20.0 [5.7 to 43.7] | 25.0 [8.7 to 49.1] | 15.8 [11.8 to 20.4] | 23.5 [18.8 to 28.7] | 22.3 [17.7 to 27.4] | 20.6 [16.2 to 25.6] | 23.6 [18.9 to 28.8] | 24.4 [19.7 to 29.5]
  Headache: Moderate | 6.7 [0.8 to 22.1] | 6.7 [0.8 to 22.1] | 30.0 [14.7 to 49.4] | 24.2 [20.4 to 28.3] | 19.0 [13.2 to 26.0] | 27.2 [22.4 to 32.4] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 25.0 [8.7 to 49.1] | 10.4 [7.2 to 14.4] | 14.4 [10.6 to 18.9] | 13.3 [9.7 to 17.7] | 14.6 [10.8 to 19.1] | 9.6 [6.5 to 13.5] | 10.9 [7.7 to 14.9]
  Headache: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 3.3 [0.1 to 17.2] | 1.7 [0.7 to 3.3] | 1.9 [0.4 to 5.4] | 2.8 [1.3 to 5.3] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0.3 [0.0 to 1.9] | 1.0 [0.2 to 2.9] | 1.0 [0.2 to 2.9] | 1.3 [0.4 to 3.4] | 0.3 [0.0 to 1.8] | 1.3 [0.4 to 3.2]
  Headache: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Chills: Any | 23.3 [9.9 to 42.3] | 23.3 [9.9 to 42.3] | 40.0 [22.7 to 59.4] | 35.6 [31.3 to 40.1] | 27.8 [21.0 to 35.5] | 38.4 [33.1 to 44.0] | 5.0 [0.1 to 24.9] | 20.0 [5.7 to 43.7] | 15.0 [3.2 to 37.9] | 35.0 [15.4 to 59.2] | 25.0 [8.7 to 49.1] | 30.0 [11.9 to 54.3] | 16.4 [12.4 to 21.1] | 24.2 [19.4 to 29.4] | 25.6 [20.7 to 30.9] | 25.6 [20.7 to 30.9] | 13.0 [9.4 to 17.3] | 23.7 [19.1 to 28.8]
  Chills: Mild | 13.3 [3.8 to 30.7] | 13.3 [3.8 to 30.7] | 13.3 [3.8 to 30.7] | 20.4 [16.9 to 24.3] | 15.8 [10.5 to 22.5] | 18.8 [14.6 to 23.5] | 0 [0.0 to 16.8] | 15.0 [3.2 to 37.9] | 5.0 [0.1 to 24.9] | 30.0 [11.9 to 54.3] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 10.7 [7.5 to 14.8] | 13.1 [9.5 to 17.5] | 13.0 [9.4 to 17.3] | 11.3 [8.0 to 15.4] | 8.3 [5.4 to 12.0] | 13.5 [9.9 to 17.8]
  Chills: Moderate | 10.0 [2.1 to 26.5] | 10.0 [2.1 to 26.5] | 20.0 [7.7 to 38.6] | 14.6 [11.5 to 18.1] | 11.4 [6.9 to 17.4] | 17.8 [13.8 to 22.5] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 20.0 [5.7 to 43.7] | 15.0 [3.2 to 37.9] | 5.7 [3.4 to 9.0] | 10.4 [7.2 to 14.4] | 12.0 [8.5 to 16.2] | 12.0 [8.5 to 16.2] | 4.7 [2.6 to 7.7] | 10.3 [7.1 to 14.2]
  Chills: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 6.7 [0.8 to 22.1] | 0.6 [0.1 to 1.8] | 0.6 [0.0 to 3.5] | 1.9 [0.7 to 4.0] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 1.2] | 0.7 [0.1 to 2.4] | 0.7 [0.1 to 2.4] | 2.3 [0.9 to 4.7] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Chills: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Vomiting: Any | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 3.1 [1.8 to 5.1] | 0.6 [0.0 to 3.5] | 3.8 [2.0 to 6.5] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 1.3 [0.4 to 3.4] | 1.7 [0.5 to 3.9] | 3.0 [1.4 to 5.6] | 2.7 [1.2 to 5.2] | 1.7 [0.5 to 3.8] | 1.3 [0.4 to 3.2]
  Vomiting: Mild | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 2.7 [1.4 to 4.6] | 0.6 [0.0 to 3.5] | 3.4 [1.7 to 6.1] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0.7 [0.1 to 2.4] | 1.3 [0.4 to 3.4] | 2.3 [0.9 to 4.7] | 2.3 [0.9 to 4.7] | 1.7 [0.5 to 3.8] | 1.3 [0.4 to 3.2]
  Vomiting: Moderate | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0.4 [0.1 to 1.5] | 0 [0.0 to 2.3] | 0.3 [0.0 to 1.7] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0.7 [0.1 to 2.4] | 0.3 [0.0 to 1.9] | 0.7 [0.1 to 2.4] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Vomiting: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Vomiting: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  Diarrhea: Any | 20.0 [7.7 to 38.6] | 3.3 [0.1 to 17.2] | 13.3 [3.8 to 30.7] | 12.7 [9.9 to 16.0] | 10.8 [6.4 to 16.7] | 12.2 [8.8 to 16.3] | 15.0 [3.2 to 37.9] | 15.0 [3.2 to 37.9] | 15.0 [3.2 to 37.9] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 4.4 [2.3 to 7.3] | 5.7 [3.4 to 9.0] | 8.0 [5.2 to 11.6] | 10.3 [7.1 to 14.3] | 9.0 [6.0 to 12.8] | 6.4 [4.0 to 9.7]
  Diarrhea: Mild | 16.7 [5.6 to 34.7] | 3.3 [0.1 to 17.2] | 13.3 [3.8 to 30.7] | 9.6 [7.1 to 12.6] | 9.5 [5.4 to 15.2] | 10.0 [6.9 to 13.8] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 3.4 [1.6 to 6.1] | 3.7 [1.9 to 6.5] | 6.6 [4.1 to 10.1] | 9.0 [6.0 to 12.8] | 6.0 [3.6 to 9.3] | 5.8 [3.5 to 9.0]
  Diarrhea: Moderate | 3.3 [0.1 to 17.2] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 3.1 [1.8 to 5.1] | 1.3 [0.2 to 4.5] | 2.2 [0.9 to 4.5] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 1.0 [0.2 to 2.9] | 2.0 [0.7 to 4.3] | 0.7 [0.1 to 2.4] | 1.3 [0.4 to 3.4] | 1.7 [0.5 to 3.8] | 0.6 [0.1 to 2.3]
  Diarrhea: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0.7 [0.1 to 2.4] | 0 [0.0 to 1.2] | 1.3 [0.4 to 3.4] | 0 [0.0 to 1.2]
  Diarrhea: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  New or worsened muscle pain: Any | 30.0 [14.7 to 49.4] | 30.0 [14.7 to 49.4] | 46.7 [28.3 to 65.7] | 39.8 [35.4 to 44.3] | 36.7 [29.2 to 44.7] | 42.2 [36.7 to 47.8] | 25.0 [8.7 to 49.1] | 20.0 [5.7 to 43.7] | 25.0 [8.7 to 49.1] | 35.0 [15.4 to 59.2] | 20.0 [5.7 to 43.7] | 35.0 [15.4 to 59.2] | 19.8 [15.4 to 24.8] | 25.5 [20.7 to 30.8] | 23.9 [19.2 to 29.1] | 30.6 [25.4 to 36.1] | 22.3 [17.7 to 27.4] | 27.2 [22.4 to 32.5]
  New or worsened muscle pain: Mild | 6.7 [0.8 to 22.1] | 10.0 [2.1 to 26.5] | 23.3 [9.9 to 42.3] | 18.3 [15.0 to 22.1] | 20.3 [14.3 to 27.4] | 17.8 [13.8 to 22.5] | 10.0 [1.2 to 31.7] | 15.0 [3.2 to 37.9] | 10.0 [1.2 to 31.7] | 25.0 [8.7 to 49.1] | 5.0 [0.1 to 24.9] | 25.0 [8.7 to 49.1] | 11.7 [8.3 to 16.0] | 10.1 [6.9 to 14.1] | 11.6 [8.2 to 15.8] | 12.6 [9.1 to 16.9] | 13.3 [9.7 to 17.7] | 14.1 [10.4 to 18.5]
  New or worsened muscle pain: Moderate | 23.3 [9.9 to 42.3] | 20.0 [7.7 to 38.6] | 23.3 [9.9 to 42.3] | 21.3 [17.7 to 25.2] | 15.8 [10.5 to 22.5] | 22.2 [17.8 to 27.1] | 15.0 [3.2 to 37.9] | 5.0 [0.1 to 24.9] | 15.0 [3.2 to 37.9] | 10.0 [1.2 to 31.7] | 15.0 [3.2 to 37.9] | 10.0 [1.2 to 31.7] | 8.1 [5.2 to 11.7] | 14.4 [10.6 to 18.9] | 12.0 [8.5 to 16.2] | 15.9 [12.0 to 20.6] | 9.0 [6.0 to 12.8] | 12.8 [9.3 to 17.0]
  New or worsened muscle pain: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0.2 [0.0 to 1.2] | 0.6 [0.0 to 3.5] | 2.2 [0.9 to 4.5] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 1.0 [0.2 to 2.9] | 0.3 [0.0 to 1.8] | 2.0 [0.7 to 4.3] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.8]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]
  New or worsened joint pain: Any | 20.0 [7.7 to 38.6] | 16.7 [5.6 to 34.7] | 23.3 [9.9 to 42.3] | 25.4 [21.6 to 29.6] | 20.9 [14.8 to 28.1] | 24.1 [19.5 to 29.1] | 20.0 [5.7 to 43.7] | 25.0 [8.7 to 49.1] | 15.0 [3.2 to 37.9] | 20.0 [5.7 to 43.7] | 15.0 [3.2 to 37.9] | 35.0 [15.4 to 59.2] | 9.1 [6.1 to 12.9] | 16.1 [12.1 to 20.8] | 16.6 [12.6 to 21.3] | 19.6 [15.3 to 24.5] | 11.3 [8.0 to 15.4] | 18.6 [14.4 to 23.4]
  New or worsened joint pain: Mild | 10.0 [2.1 to 26.5] | 13.3 [3.8 to 30.7] | 10.0 [2.1 to 26.5] | 12.5 [9.7 to 15.8] | 10.1 [5.9 to 15.9] | 9.1 [6.2 to 12.8] | 10.0 [1.2 to 31.7] | 15.0 [3.2 to 37.9] | 5.0 [0.1 to 24.9] | 20.0 [5.7 to 43.7] | 5.0 [0.1 to 24.9] | 15.0 [3.2 to 37.9] | 5.4 [3.1 to 8.6] | 9.7 [6.6 to 13.7] | 9.3 [6.3 to 13.2] | 8.3 [5.4 to 12.0] | 7.6 [4.9 to 11.2] | 10.3 [7.1 to 14.2]
  New or worsened joint pain: Moderate | 10.0 [2.1 to 26.5] | 3.3 [0.1 to 17.2] | 13.3 [3.8 to 30.7] | 12.5 [9.7 to 15.8] | 10.8 [6.4 to 16.7] | 14.1 [10.4 to 18.4] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.8] | 10.0 [1.2 to 31.7] | 20.0 [5.7 to 43.7] | 3.7 [1.9 to 6.5] | 6.0 [3.6 to 9.4] | 7.3 [4.6 to 10.9] | 11.0 [7.7 to 15.1] | 3.7 [1.8 to 6.4] | 8.0 [5.3 to 11.6]
  New or worsened joint pain: Severe | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0.4 [0.1 to 1.5] | 0 [0.0 to 2.3] | 0.9 [0.2 to 2.7] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.9] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.8] | 0 [0.0 to 1.2] | 0.3 [0.0 to 1.8]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 0.8] | 0 [0.0 to 2.3] | 0 [0.0 to 1.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2] | 0 [0.0 to 1.2]

52. Primary Outcome: SSE: Percentage of Participants Reporting Adverse Events (AEs) Within 1 Month After Study Vaccination
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants reporting AEs within 1 month after study vaccination were reported in this outcome measure. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e., excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From study vaccination up to 1 Month after study vaccination
Population: Safety population included all participants who received at least 1 dose of the study intervention. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg
Number analyzed (Participants) | 30 | 30 | 30 | 482 | 159 | 321 | 20 | 20 | 20 | 20 | 20 | 20 | 305 | 302 | 307 | 306 | 305 | 313
Percentage of participants | 13.3 [3.8 to 30.7] | 6.7 [0.8 to 22.1] | 13.3 [3.8 to 30.7] | 7.7 [5.5 to 10.4] | 6.3 [3.1 to 11.3] | 9.3 [6.4 to 13.1] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.8] | 15.0 [3.2 to 37.9] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 5.9 [3.5 to 9.2] | 6.6 [4.1 to 10.0] | 8.5 [5.6 to 12.2] | 3.6 [1.8 to 6.3] | 6.2 [3.8 to 9.6] | 10.4 [7.3 to 14.4]

53. Primary Outcome: SSE: Percentage of Participants Reporting Serious Adverse Events (SAEs) Within 6 Month After Study Vaccination
Description: as for outcome 18
Time Frame: From study vaccination up to 6 Months after study vaccination
Population: as for outcome 52
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg
Number analyzed (Participants) | 30 | 30 | 30 | 482 | 159 | 321 | 20 | 20 | 20 | 20 | 20 | 20 | 305 | 302 | 307 | 307 | 304 | 313
Percentage of participants | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0.6 [0.1 to 1.8] | 1.3 [0.2 to 4.5] | 0.9 [0.2 to 2.7] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 2.0 [0.7 to 4.2] | 0.7 [0.1 to 2.4] | 3.9 [2.0 to 6.7] | 1.3 [0.4 to 3.3] | 1.3 [0.4 to 3.3] | 1.9 [0.7 to 4.1]

54. Primary Outcome: SSE: Percentage of Participants With Elevated Troponin I Levels Before the Study Vaccination- 18 to 55 Years of Age
Description: Percentage of participants with elevated troponin I levels before study vaccination were reported in this outcome measure.
Time Frame: Before study vaccination (pre-dose)
Population: Safety population included all participants who received at least 1 dose of the study intervention. As pre-specified in the protocol, this outcome measure was planned to be analyzed only in the Sentinel Cohort in participants of 18 to 55 years of age.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg
Number analyzed (Participants) | 30 | 30 | 30
Percentage of participants | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6]

55. Primary Outcome: SSE: Percentage of Participants With Elevated Troponin I Levels 3 Days After Study Vaccination- 18 to 55 Years of Age
Description: as for outcome 54
Time Frame: 3 days after study vaccination
Population: as for outcome 54
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg
Number analyzed (Participants) | 30 | 30 | 30
Percentage of participants | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6]

56. Primary Outcome: SSE: Geometric Mean Ratio (GMR) Based on Geometric Mean Titers of SARS-CoV-2 Omicron BA.1 Strain Neutralizing Titers 1 Month After Study Vaccination
Description: GMR calculated based on GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers at 1 month after the study vaccination was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: 1 month after study vaccination
Population: EIP: all eligible randomized participants who received study intervention to which they were randomized, had valid and determinate immunogenicity result within 28-42 days after study vaccination, had no other important protocol deviations as determined by the clinician. 'N' = participants evaluable for this outcome measure. As pre-specified in the protocol, this outcome measure was not planned to be analyzed in ''SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg''.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg
Number analyzed (Participants) | 163 | 169 | 174 | 178 | 175
Titer | 455.8 [365.9 to 567.6] | 1014.5 [825.6 to 1246.7] | 1435.2 [1208.1 to 1704.8] | 711.0 [588.3 to 859.2] | 900.1 [726.3 to 1115.6]
Statistical Analysis 1: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the mean difference of the logarithms of the titers (BNT162b2 OMI [30 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on the student t distribution; Test type: Other; Geometric mean ratio (GMR) = 2.23, 95% CI 2-sided [1.65 to 3.00]
Statistical Analysis 2: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the mean difference of the logarithms of the titers (BNT162b2 OMI [60 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on the student t distribution; Test type: Other; Geometric mean ratio (GMR) = 3.15, 95% CI 2-sided [2.38 to 4.16]
Statistical Analysis 3: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the mean difference of the logarithms of the titers (BNT162b2 [15 mcg] + BNT162b2 OMI [15 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on the student t distribution; Test type: Other; Geometric mean ratio (GMR) = 1.56, 95% CI 2-sided [1.17 to 2.08]
Statistical Analysis 4: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the mean difference of the logarithms of the titers (BNT162b2 [30 mcg] + BNT162b2 OMI [30 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on the student t distribution; Test type: Other; Geometric mean ratio (GMR) = 1.97, 95% CI 2-sided [1.45 to 2.68]

57. Primary Outcome: SSE: Percentage of Participants With Seroresponse to the SARS-CoV-2 Omicron BA.1 Strain at 1 Month After Study Vaccination
Description: Seroresponse was defined as achieving >= 4-fold rise from baseline (before study vaccination). If baseline measurement is below lower limit of quantification (LLOQ), postvaccination measure of >= 4 × LLOQ is considered seroresponse. Exact 2-sided CI, based on Clopper and Pearson method was used. Percentage of participants achieving seroresponse at 1 month was reported in this outcome measure.
Time Frame: 1 month after study vaccination
Population: as for outcome 56
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg
Number analyzed (Participants) | 149 | 163 | 166 | 169 | 162
Percentage of participants | 57.0 [48.7 to 65.1] | 76.7 [69.4 to 82.9] | 86.1 [79.9 to 91.0] | 71.6 [64.2 to 78.3] | 67.9 [60.1 to 75.0]
Statistical Analysis 1: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg; Difference in proportions, expressed as a percentage (BNT162b2 OMI [30 mcg] - BNT162b2 [30 μg]). 2-Sided CI based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Other; Difference in percentages = 19.6, 95% CI 2-sided [9.3 to 29.7]
Statistical Analysis 2: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg; Difference in proportions, expressed as a percentage (BNT162b2 OMI [60 mcg] - BNT162b2 [30 μg]). 2-Sided CI based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Other; Difference in Percentages = 29.1, 95% CI 2-sided [19.4 to 38.5]
Statistical Analysis 3: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg; Difference in proportions, expressed as a percentage (BNT162b2 [15 mcg] + BNT162b2 OMI [15 mcg] - BNT162b2 [30 μg]). 2-Sided CI based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Other; Difference in percentages = 14.6, 95% CI 2-sided [4.0 to 24.9]
Statistical Analysis 4: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg; Difference in proportions, expressed as a percentage (BNT162b2 [30 mcg] + BNT162b2 OMI [30 mcg] - BNT162b2 [30 μg]). 2-Sided CI based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Other; Difference in Percentages = 10.9, 95% CI 2-sided [0.1 to 21.4]

58. Primary Outcome: SSF: Geometric Mean Titer (GMTs) of SARS-CoV-2 Omicron BA.1 Strain Neutralizing Titers Before Vaccination
Description: GMT of SARS-CoV-2 Omicron BA.1 strain neutralizing titers before vaccination was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: Before vaccination (pre-dose)
Population: All-available immunogenicity population included all randomized participants who received the study intervention with a valid and determinate immunogenicity result after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 21
Titer | 41.7 [22.4 to 77.4] | 33.2 [17.6 to 62.6] | 32.0 [17.0 to 60.1] | 36.8 [17.5 to 77.1] | 78.8 [29.3 to 211.6] | 21.5 [14.2 to 32.7]

59. Primary Outcome: SSF: Percentage of Participants With Local Reactions Within 7 Days After Study Vaccination
Description: Local reactions were recorded by participants in e-diary. Redness and swelling were measured and recorded in measuring device units (mdu) where, 1 mdu =0.5 centimeter (cm) and were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and Grade 4 (necrosis [swelling] or necrosis/exfoliative dermatitis [redness]). Grade 4 were classified by investigator or medically qualified person. Percentage of participants reporting local reactions after study vaccination and associated 2-sided 95% confidence interval (CI) based on Clopper and Pearson method was presented.
Time Frame: Day 1 up to Day 7 after the study vaccination
Population: Safety population included all participants receiving at least 1 dose of study intervention. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 21
Percentage of participants
  Redness: Any | 19.0 [5.4 to 41.9] | 21.1 [6.1 to 45.6] | 23.8 [8.2 to 47.2] | 20.0 [5.7 to 43.7] | 10.0 [1.2 to 31.7] | 28.6 [11.3 to 52.2]
  Redness: Mild | 4.8 [0.1 to 23.8] | 10.5 [1.3 to 33.1] | 14.3 [3.0 to 36.3] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 23.8 [8.2 to 47.2]
  Redness: Moderate | 14.3 [3.0 to 36.3] | 10.5 [1.3 to 33.1] | 9.5 [1.2 to 30.4] | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 4.8 [0.1 to 23.8]
  Redness: Severe | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Redness: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Swelling: Any | 14.3 [3.0 to 36.3] | 15.8 [3.4 to 39.6] | 14.3 [3.0 to 36.3] | 15.0 [3.2 to 37.9] | 15.0 [3.2 to 37.9] | 28.6 [11.3 to 52.2]
  Swelling: Mild | 4.8 [0.1 to 23.8] | 5.3 [0.1 to 26.0] | 4.8 [0.1 to 23.8] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 23.8 [8.2 to 47.2]
  Swelling: Moderate | 9.5 [1.2 to 30.4] | 10.5 [1.3 to 33.1] | 9.5 [1.2 to 30.4] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 4.8 [0.1 to 23.8]
  Swelling: Severe | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Swelling: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Pain at the injection site: Any | 71.4 [47.8 to 88.7] | 94.7 [74.0 to 99.9] | 90.5 [69.6 to 98.8] | 80.0 [56.3 to 94.3] | 75.0 [50.9 to 91.3] | 90.5 [69.6 to 98.8]
  Pain at the injection site: Mild | 52.4 [29.8 to 74.3] | 52.6 [28.9 to 75.6] | 66.7 [43.0 to 85.4] | 45.0 [23.1 to 68.5] | 55.0 [31.5 to 76.9] | 57.1 [34.0 to 78.2]
  Pain at the injection site: Moderate | 19.0 [5.4 to 41.9] | 36.8 [16.3 to 61.6] | 19.0 [5.4 to 41.9] | 35.0 [15.4 to 59.2] | 20.0 [5.7 to 43.7] | 33.3 [14.6 to 57.0]
  Pain at the injection site: Severe | 0 [0.0 to 16.1] | 5.3 [0.1 to 26.0] | 4.8 [0.1 to 23.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Pain at the injection site: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]

60. Primary Outcome: SSF: Percentage of Participants With Systemic Events Within 7 Days After Study Vaccination
Description: as for outcome 51
Time Frame: Day 1 up to Day 7 after the study vaccination
Population: as for outcome 51
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 21
Percentage of participants
  Fever: >= 38.0 deg C | 9.5 [1.2 to 30.4] | 10.5 [1.3 to 33.1] | 9.5 [1.2 to 30.4] | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 4.8 [0.1 to 23.8]
  Fever: >= 38.0 deg C to 38.4 deg C | 9.5 [1.2 to 30.4] | 5.3 [0.1 to 26.0] | 4.8 [0.1 to 23.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 4.8 [0.1 to 23.8]
  Fever: >38.4 deg C to 38.9 deg C | 0 [0.0 to 16.1] | 5.3 [0.1 to 26.0] | 0 [0.0 to 16.1] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.1]
  Fever: >38.9 deg C to 40.0 deg C | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 4.8 [0.1 to 23.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Fever: >40.0 deg C | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Fatigue: Any | 47.6 [25.7 to 70.2] | 36.8 [16.3 to 61.6] | 42.9 [21.8 to 66.0] | 55.0 [31.5 to 76.9] | 50.0 [27.2 to 72.8] | 57.1 [34.0 to 78.2]
  Fatigue: Mild | 9.5 [1.2 to 30.4] | 10.5 [1.3 to 33.1] | 9.5 [1.2 to 30.4] | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 23.8 [8.5 to 47.2]
  Fatigue: Moderate | 23.8 [8.2 to 47.2] | 21.1 [6.1 to 45.6] | 28.6 [11.3 to 52.2] | 35.0 [15.4 to 59.2] | 40.0 [19.1 to 63.9] | 33.3 [14.6 to 57.0]
  Fatigue: Severe | 14.3 [3.0 to 36.3] | 5.3 [0.1 to 26.0] | 4.8 [0.1 to 23.8] | 10.0 [1.2 to 31.7] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.1]
  Fatigue: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Headache: Any | 28.6 [11.3 to 52.2] | 26.3 [9.1 to 51.2] | 23.8 [8.2 to 47.2] | 55.0 [31.5 to 76.9] | 35.0 [15.4 to 59.2] | 38.1 [18.1 to 61.6]
  Headache: Mild | 19.0 [5.4 to 41.9] | 15.8 [3.4 to 39.6] | 4.8 [0.1 to 23.8] | 15.0 [3.2 to 37.9] | 20.0 [5.7 to 43.7] | 19.0 [5.4 to 41.9]
  Headache: Moderate | 9.5 [1.2 to 30.4] | 10.5 [1.3 to 33.1] | 14.3 [3.0 to 36.3] | 40.0 [19.1 to 63.9] | 15.0 [3.2 to 37.9] | 19.0 [5.4 to 41.9]
  Headache: Severe | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 4.8 [0.1 to 23.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.7] | 0 [0.0 to 16.1]
  Headache: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Chills: Any | 14.3 [3.0 to 36.3] | 15.8 [3.4 to 39.6] | 23.8 [8.2 to 47.2] | 25.0 [8.7 to 49.1] | 5.0 [0.1 to 24.9] | 14.3 [3.0 to 36.3]
  Chills: Mild | 4.8 [0.1 to 23.8] | 10.5 [1.3 to 33.1] | 14.3 [3.0 to 36.3] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.8] | 9.5 [1.2 to 30.4]
  Chills: Moderate | 9.5 [1.2 to 30.4] | 5.3 [0.1 to 26.0] | 4.8 [0.1 to 23.8] | 5.0 [0.1 to 24.9] | 5.0 [0.1 to 24.9] | 4.8 [0.1 to 23.8]
  Chills: Severe | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 4.8 [0.1 to 23.8] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Chills: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Vomiting: Any | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Vomiting: Mild | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Vomiting: Moderate | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Vomiting: Severe | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Vomiting: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Diarrhea: Any | 14.3 [3.0 to 36.3] | 5.3 [0.1 to 26.0] | 9.5 [1.2 to 30.4] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Diarrhea: Mild | 9.5 [1.2 to 30.4] | 5.3 [0.1 to 26.0] | 4.8 [0.1 to 23.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Diarrhea: Moderate | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 4.8 [0.1 to 23.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Diarrhea: Severe | 4.8 [0.1 to 23.8] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  Diarrhea: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  New or worsened muscle pain: Any | 19.0 [5.4 to 41.9] | 42.1 [20.3 to 66.5] | 23.8 [8.2 to 47.2] | 30.0 [11.9 to 54.3] | 25.0 [8.7 to 49.1] | 28.6 [11.3 to 52.2]
  New or worsened muscle pain: Mild | 4.8 [0.1 to 23.8] | 10.5 [1.3 to 33.1] | 14.3 [3.0 to 36.3] | 10.0 [1.2 to 31.9] | 15.0 [3.2 to 37.9] | 23.8 [8.2 to 47.2]
  New or worsened muscle pain: Moderate | 14.3 [3.0 to 36.3] | 31.6 [12.6 to 56.6] | 4.8 [0.1 to 23.8] | 20.0 [5.7 to 43.7] | 10.0 [1.2 to 31.7] | 4.8 [0.1 to 23.8]
  New or worsened muscle pain: Severe | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 4.8 [0.1 to 23.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  New or worsened joint pain: Any | 14.3 [3.0 to 36.3] | 15.8 [3.4 to 39.6] | 14.3 [3.0 to 36.3] | 20.0 [5.7 to 43.7] | 10.0 [1.2 to 31.7] | 9.5 [1.2 to 30.4]
  New or worsened joint pain: Mild | 4.8 [0.1 to 23.8] | 10.5 [1.3 to 33.1] | 9.5 [1.2 to 30.4] | 10.0 [1.2 to 31.7] | 10.0 [1.2 to 31.7] | 4.8 [0.1 to 23.8]
  New or worsened joint pain: Moderate | 9.5 [1.2 to 30.4] | 5.3 [0.1 to 26.0] | 4.8 [0.1 to 23.8] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.8] | 4.8 [0.1 to 23.8]
  New or worsened joint pain: Severe | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 16.1] | 0 [0.0 to 17.6] | 0 [0.0 to 16.1] | 0 [0.0 to 16.8] | 0 [0.0 to 16.8] | 0 [0.0 to 16.1]

61. Primary Outcome: SSF: Percentage of Participants Reporting Adverse Events (AEs) Within 1 Month After Study Vaccination
Description: as for outcome 52
Time Frame: From study vaccination up to 1 Month after study vaccination
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 21
Percentage of participants | 0 [0.0 to 16.1] | 10.5 [1.3 to 33.1] | 9.5 [1.2 to 30.4] | 5.0 [0.1 to 24.9] | 10.0 [1.2 to 31.7] | 0 [0.0 to 16.1]

62. Primary Outcome: SSF: Percentage of Participants Reporting Serious Adverse Events (SAEs) Within 6 Months After Study Vaccination
Description: as for outcome 18
Time Frame: From study vaccination up to 6 Months after study vaccination
Population: Safety population included all participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 21
Percentage of participants | 0 [0.0 to 16.1] | 5.3 [0.1 to 26.0] | 4.8 [0.1 to 23.8] | 0 [0.0 to 16.8] | 5.0 [0.1 to 24.9] | 0 [0.0 to 16.1]

63. Primary Outcome: SSF: GMTs of SARS-CoV-2 Reference-Strain-Neutralizing Titers Before Vaccination
Description: GMT of SARS-CoV-2 reference-strain-neutralizing titers before vaccination was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: Before vaccination (pre-dose)
Population: as for outcome 58
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 21
Titer | 541.1 [345.1 to 848.3] | 382.4 [176.3 to 829.3] | 437.5 [244.0 to 784.2] | 315.2 [188.0 to 528.4] | 803.4 [347.8 to 1855.8] | 256.0 [135.1 to 485.0]

64. Primary Outcome: SSF: GMTs of SARS-CoV-2 Omicron BA.4/BA.5 Strain Neutralizing Titers Before Vaccination
Description: GMT of SARS-CoV-2 Omicron BA.4/BA.5 strain neutralizing titers before vaccination was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: Before vaccination (pre-dose)
Population: All-available immunogenicity population included all randomized participants who received the study intervention with a valid and determinate immunogenicity result after vaccination. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 21
Titer | 27.1 [16.8 to 43.7] | 18.0 [12.1 to 26.7] | 20.2 [12.6 to 32.3] | 23.4 [13.9 to 39.4] | 42.2 [19.6 to 91.1] | 15.0 [11.8 to 19.1]

65. Primary Outcome: SSF: Geometric Mean Ratio (GMR) Based on GMT of SARS-CoV-2 Omicron BA.1 Strain-Neutralizing Titers at Day 7
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 Omicron BA.1 strain neutralizing titers at Day 7 were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Day 7 (7 days after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 20
Titer | 146.1 [102.5 to 208.2] | 101.6 [48.6 to 212.6] | 217.1 [97.8 to 481.9] | 315.2 [164.6 to 603.5] | 337.8 [133.8 to 852.7] | 222.9 [125.7 to 395.1]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the difference in LS means (BNT162b2 [60 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of baseline assay results (log scale) and vaccine group; Test type: Other; Geometric mean ratio (GMR) = 0.79, 95% CI 2-sided [0.40 to 1.56]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the difference in LS means (BNT162b2 OMI [30 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of baseline assay results (log scale) and vaccine group; Test type: Other; Geometric mean ratio (GMR) = 1.78, 95% CI 2-sided [0.93 to 3.43]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the difference in LS means (BNT162b2 OMI [60 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of baseline assay results (log scale) and vaccine group; Test type: Other; Geometric mean ratio (GMR) = 2.35, 95% CI 2-sided [1.22 to 4.55]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the difference in LS means (BNT162b2 [15 mcg] + BNT162b2 OMI [15 mcg]- BNT162b2 [30 mcg]) and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of baseline assay results (log scale) and vaccine group; Test type: Other; Geometric mean ratio (GMR) = 1.49, 95% CI 2-sided [0.76 to 2.89]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the difference in LS means (BNT162b2 [30 mcg] + BNT162b2 OMI [30 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of baseline assay results (log scale) and vaccine group; Test type: Other; Geometric mean ratio (GMR) = 2.33, 95% CI 2-sided [1.20 to 4.53]

66. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Reference-Strain-Neutralizing Titers at Day 7
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron reference strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 reference strain neutralizing titers at Day 7 were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Day 7 (7 days after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 20
Titer | 1917.2 [1153.8 to 3185.7] | 1241.4 [624.3 to 2468.6] | 1472.3 [855.4 to 2534.0] | 1499.2 [838.6 to 2680.4] | 2702.4 [1419.7 to 5143.8] | 1845.8 [1087.4 to 3133.1]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.76, 95% CI 2-sided [0.40 to 1.42]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 0.86, 95% CI 2-sided [0.47 to 1.58]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 1.06, 95% CI 2-sided [0.57 to 1.95]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the difference in LS means BNT162b2 [15 mcg] + BNT162b2 OMI [15 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of baseline assay results (log scale) and vaccine group; Test type: Other; Geometric mean ratio (GMR) = 1.13, 95% CI 2-sided [0.61 to 2.09]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 1.35, 95% CI 2-sided [0.73 to 2.50]

67. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Omicron BA.4/BA.5 Strain Neutralizing Titers at Day 7
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.4/BA.5 strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 Omicron BA.4/BA.5 strain neutralizing titers at Day 7 were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Day 7 (7 days after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 17 | 21 | 20 | 20 | 21
Titer | 75.5 [52.7 to 108.0] | 56.6 [32.1 to 99.8] | 73.0 [38.7 to 137.9] | 76.1 [46.0 to 125.9] | 123.6 [63.8 to 239.5] | 70.7 [48.5 to 103.0]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.95, 95% CI 2-sided [0.58 to 1.56]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 1.22, 95% CI 2-sided [0.77 to 1.93]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 1.13, 95% CI 2-sided [0.71 to 1.80]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; GMRs and 2-sided 95% CIs were calculated by exponentiating the difference in LS means (BNT162b2 [15 mcg] + BNT162b2 OMI [15 mcg] - BNT162b2 [30 mcg]) and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of baseline assay results (log scale) and vaccine group; Test type: Other; Geometric mean ratio (GMR) = 1.16, 95% CI 2-sided [0.73 to 1.84]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 1.49, 95% CI 2-sided [0.94 to 2.37]

68. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Omicron BA.1 Strain-Neutralizing Titers at Month 1
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 Omicron BA.1 strain neutralizing titers at 1 month were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 1 (1 month after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 20 | 20 | 20 | 20
Titer | 420.0 [252.2 to 699.5] | 188.1 [88.9 to 398.2] | 699.4 [398.9 to 1226.4] | 675.6 [343.2 to 1329.8] | 1024.0 [509.4 to 2058.3] | 477.7 [236.0 to 967.1]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.49, 95% CI 2-sided [0.24 to 1.03]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 1.84, 95% CI 2-sided [0.90 to 3.76]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 1.72, 95% CI 2-sided [0.84 to 3.50]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 1.75, 95% CI 2-sided [0.85 to 3.59]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 1.56, 95% CI 2-sided [0.76 to 3.20]

69. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Reference-Strain-Neutralizing Titers at Month 1
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron reference strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 reference strain neutralizing titers at 1 month were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 1 (1 month after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 20 | 20 | 20 | 20
Titer | 4674.1 [3112.1 to 7020.2] | 2048.4 [1007.8 to 4163.7] | 3327.0 [1867.6 to 5926.9] | 3565.8 [1992.1 to 6382.7] | 5404.7 [3359.8 to 8694.1] | 2521.4 [1388.9 to 4577.4]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.50, 95% CI 2-sided [0.26 to 0.95]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 0.76, 95% CI 2-sided [0.41 to 1.43]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 0.98, 95% CI 2-sided [0.52 to 1.84]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 0.96, 95% CI 2-sided [0.51 to 1.80]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 0.71, 95% CI 2-sided [0.38 to 1.34]

70. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Omicron BA.4/BA.5 Strain-Neutralizing Titers at Month 1
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron reference strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 Omicron BA.4/BA.5 strain neutralizing titers at 1 month were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 1 (1 month after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 19 | 21 | 20 | 20 | 20
Titer | 157.6 [94.0 to 264.2] | 85.7 [52.5 to 139.8] | 151.0 [72.6 to 314.1] | 230.7 [140.0 to 379.2] | 284.0 [134.7 to 599.1] | 147.0 [86.3 to 250.4]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.72, 95% CI 2-sided [0.38 to 1.37]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 1.19, 95% CI 2-sided [0.65 to 2.21]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 1.63, 95% CI 2-sided [0.88 to 3.02]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 1.28, 95% CI 2-sided [0.68 to 2.39]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 1.42, 95% CI 2-sided [0.76 to 2.67]

71. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Omicron BA.1 Strain-Neutralizing Titers at Month 3
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 Omicron BA.1 strain neutralizing titers at 3 months were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 3 (3 month after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 20 | 19 | 20 | 19
Titer | 247.3 [119.7 to 510.7] | 118.5 [54.6 to 257.1] | 461.4 [203.8 to 1044.7] | 711.0 [388.8 to 1300.1] | 512.0 [246.9 to 1061.6] | 285.6 [132.8 to 614.1]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.52, 95% CI 2-sided [0.21 to 1.25]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 2.07, 95% CI 2-sided [0.88 to 4.88]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 2.96, 95% CI 2-sided [1.24 to 7.06]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 1.52, 95% CI 2-sided [0.64 to 3.62]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio = 1.53, 95% CI 2-sided [0.64 to 3.67]

72. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Reference-Strain-Neutralizing Titers at Month 3
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron reference strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 reference strain neutralizing titers at 3 months were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 3 (3 month after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 20 | 19 | 20 | 19
Titer | 2896.3 [1738.8 to 4824.3] | 1290.2 [675.2 to 2465.3] | 2610.3 [1265.9 to 5382.4] | 2949.6 [1550.2 to 5612.3] | 2610.3 [1506.5 to 4522.8] | 1474.8 [815.0 to 2668.9]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.52, 95% CI 2-sided [0.25 to 1.09]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 1.00, 95% CI 2-sided [0.49 to 2.04]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 1.29, 95% CI 2-sided [0.63 to 2.68]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 0.78, 95% CI 2-sided [0.38 to 1.59]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 0.66, 95% CI 2-sided [0.32 to 1.36]

73. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Omicron BA.4/BA.5 Strain-Neutralizing Titers at Month 3
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.4/BA.5 strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 Omicron BA.4/BA.5 strain neutralizing titers at 3 months were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 3 (3 month after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 19 | 21 | 19 | 19 | 21
Titer | 222.9 [123.3 to 402.7] | 132.8 [63.7 to 276.7] | 322.5 [147.6 to 704.6] | 458.9 [206.8 to 1018.6] | 296.2 [143.2 to 612.6] | 141.3 [86.4 to 231.1]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.75, 95% CI 2-sided [0.32 to 1.76]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 1.69, 95% CI 2-sided [0.74 to 3.85]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 2.12, 95% CI 2-sided [0.92 to 4.91]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 1.00, 95% CI 2-sided [0.43 to 2.33]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 0.89, 95% CI 2-sided [0.39 to 2.04]

74. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Omicron BA.1 Strain-Neutralizing Titers at Month 6
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 Omicron BA.1 strain neutralizing titers at 6 months were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 6 (6 month after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 20
Titer | 239.6 [98.8 to 581.4] | 229.5 [68.7 to 766.4] | 1058.4 [490.3 to 2284.6] | 1722.2 [844.3 to 3512.9] | 588.1 [280.3 to 1234.2] | 284.0 [131.8 to 612.4]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 0.99, 95% CI 2-sided [0.31 to 3.12]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 4.57, 95% CI 2-sided [1.49 to 14.07]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 7.30, 95% CI 2-sided [2.34 to 22.76]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 2.26, 95% CI 2-sided [0.72 to 7.10]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 1.28, 95% CI 2-sided [0.41 to 4.03]

75. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Reference-Strain-Neutralizing Titers at Month 6
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 reference strain neutralizing titers at 6 months were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 6 (6 months after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 20
Titer | 1424.5 [667.9 to 3037.9] | 1371.0 [508.5 to 3696.4] | 2756.4 [1328.0 to 5721.4] | 3956.5 [2256.3 to 6937.8] | 2702.4 [1457.6 to 5010.0] | 1097.5 [555.3 to 2169.1]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 1.01, 95% CI 2-sided [0.38 to 2.70]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 1.99, 95% CI 2-sided [0.76 to 5.20]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 2.99, 95% CI 2-sided [1.13 to 7.94]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 1.80, 95% CI 2-sided [0.68 to 4.75]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 0.84, 95% CI 2-sided [0.32 to 2.24]

76. Primary Outcome: SSF: GMR Based on GMT of SARS-CoV-2 Omicron BA.4/BA.5 Strain-Neutralizing Titers at Month 6
Description: GMR was calculated based on the GMT of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers and reported in statistical analysis. GMTs of SARS-CoV-2 Omicron BA.4/BA.5 strain neutralizing titers at 6 months were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Month 6 (6 months after vaccination)
Population: as for outcome 64
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 20
Titer | 203.2 [85.5 to 483.1] | 265.5 [75.9 to 928.9] | 645.1 [281.1 to 1480.5] | 1305.2 [601.1 to 2834.1] | 430.5 [204.7 to 905.4] | 187.4 [80.5 to 436.3]
Statistical Analysis 1: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 60 mcg; [analysis description as in outcome 65, analysis 1]; Test type: Other; Geometric mean ratio (GMR) = 1.50, 95% CI 2-sided [0.44 to 5.12]
Statistical Analysis 2: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 2]; Test type: Other; Geometric mean ratio (GMR) = 3.22, 95% CI 2-sided [0.99 to 10.46]
Statistical Analysis 3: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 OMI 60 mcg; [analysis description as in outcome 65, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 6.46, 95% CI 2-sided [1.96 to 21.27]
Statistical Analysis 4: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg; [analysis description as in outcome 67, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 2.08, 95% CI 2-sided [0.63 to 6.89]
Statistical Analysis 5: Comparison: SSF: BNT162b2 30 mcg vs SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg; [analysis description as in outcome 65, analysis 5]; Test type: Other; Geometric mean ratio (GMR) = 0.95, 95% CI 2-sided [0.28 to 3.17]

77. Primary Outcome: SSF: Geometric Mean Fold-Rise (GMFR) of SARS-CoV-2 Omicron BA.1 Strain-Neutralizing Titers From Before the Study Vaccination to 7 Days After Vaccination
Description: GMFR of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers before vaccination to Day 7 was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to Day 7 (7 days after vaccination)
Population: All-available immunogenicity population included all randomized or assigned participants who received the study intervention with a valid and determinate immunogenicity result after vaccination. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 20
Fold rise | 3.5 [2.1 to 5.8] | 2.9 [1.6 to 5.4] | 6.8 [4.3 to 10.7] | 8.6 [5.1 to 14.3] | 4.3 [2.0 to 9.1] | 9.8 [6.9 to 14.0]

78. Primary Outcome: SSF: GMFR of SARS-CoV-2 Reference-Strain-Neutralizing Titers From Before the Study Vaccination to 7 Days After Vaccination
Description: GMFR of SARS-CoV-2 reference-strain-neutralizing titers before vaccination to Day 7 was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to Day 7 (7 days after vaccination)
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 20
Fold rise | 3.5 [2.5 to 5.0] | 3.1 [1.8 to 5.2] | 3.4 [2.2 to 5.1] | 4.8 [3.0 to 7.5] | 3.4 [1.4 to 8.1] | 6.3 [3.9 to 10.2]

79. Primary Outcome: SSF: GMFR of SARS-CoV-2 Omicron BA.4/BA.5 Strain-Neutralizing Titers From Before the Study Vaccination to 7 Days After Vaccination
Description: GMFR of SARS-CoV-2 Omicron BA.4/BA.5 strain-neutralizing titers before vaccination to Day 7 was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to Day 7 (7 days after vaccination)
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 16 | 21 | 20 | 20 | 21
Fold rise | 2.8 [2.1 to 3.7] | 2.8 [1.8 to 4.4] | 3.6 [2.5 to 5.2] | 3.2 [2.2 to 4.8] | 2.9 [1.9 to 4.4] | 4.7 [3.4 to 6.5]

80. Primary Outcome: SSF: GMFR of SARS-CoV-2 Omicron BA.1 Strain-Neutralizing Titers From Before the Study Vaccination to 1 Month After Vaccination
Description: GMFR of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers before vaccination to 1 month was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 1 month after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 20 | 20 | 20 | 20
Fold rise | 10.1 [5.5 to 18.4] | 5.4 [2.6 to 11.4] | 20.4 [11.8 to 35.3] | 18.4 [9.5 to 35.6] | 13.0 [6.7 to 25.1] | 21.1 [11.5 to 38.8]

81. Primary Outcome: SSF: GMFR of SARS-CoV-2 Reference-Strain-Neutralizing Titers From Before the Study Vaccination to 1 Month After Vaccination
Description: GMFR of SARS-CoV-2 reference-strain-neutralizing titers before vaccination to 1 month was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 1 month after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 20 | 20 | 20 | 20
Fold rise | 8.6 [5.5 to 13.6] | 5.0 [2.5 to 10.0] | 7.2 [4.7 to 10.9] | 11.3 [6.2 to 20.8] | 6.7 [3.7 to 12.1] | 8.6 [4.1 to 17.8]

82. Primary Outcome: SSF: GMFR of SARS-CoV-2 Omicron BA.4/BA.5 Strain-Neutralizing Titers From Before the Study Vaccination to 1 Month After Vaccination
Description: GMFR of SARS-CoV-2 Omicron BA.4/BA.5 strain-neutralizing titers before vaccination to 1 month was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 1 month after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 21 | 20 | 20 | 20
Fold rise | 5.9 [3.8 to 9.1] | 4.7 [3.1 to 7.1] | 7.5 [4.6 to 12.3] | 9.8 [7.3 to 13.3] | 6.7 [3.5 to 13.0] | 9.5 [6.0 to 15.2]

83. Primary Outcome: SSF: GMFR of SARS-CoV-2 Omicron BA.1 Strain-Neutralizing Titers From Before the Study Vaccination to 3 Months After Vaccination
Description: GMFR of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers before vaccination to 3 months was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 3 months after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 20 | 19 | 20 | 19
Fold rise | 5.9 [2.7 to 12.8] | 3.3 [1.4 to 7.5] | 13.5 [6.0 to 30.0] | 17.9 [8.7 to 36.5] | 6.5 [3.2 to 13.1] | 12.0 [6.4 to 22.3]

84. Primary Outcome: SSF: GMFR of SARS-CoV-2 Reference-Strain-Neutralizing Titers From Before the Study Vaccination to 3 Months After Vaccination
Description: GMFR of SARS-CoV-2 reference-strain-neutralizing titers before vaccination to 3 months was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 3 months after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 20 | 19 | 20 | 19
Fold rise | 5.0 [2.9 to 8.5] | 3.2 [1.6 to 6.3] | 5.6 [2.6 to 11.9] | 8.6 [4.3 to 17.2] | 3.2 [1.8 to 5.8] | 4.5 [2.4 to 8.2]

85. Primary Outcome: SSF: GMFR of SARS-CoV-2 Omicron BA.4/BA.5 Strain-Neutralizing Titers From Before the Study Vaccination to 3 Months After Vaccination
Description: GMFR of SARS-CoV-2 Omicron BA.4/BA.5 strain-neutralizing titers before vaccination to 3 months was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 3 months after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 21 | 19 | 19 | 21
Fold rise | 8.6 [4.3 to 16.9] | 7.4 [3.7 to 14.9] | 16.0 [7.5 to 34.0] | 18.5 [9.2 to 37.3] | 7.2 [4.1 to 12.7] | 9.4 [5.9 to 15.2]

86. Primary Outcome: SSF: GMFR of SARS-CoV-2 Omicron BA.1 Strain-Neutralizing Titers From Before the Study Vaccination to 6 Months After Vaccination
Description: GMFR of SARS-CoV-2 Omicron BA.1 strain-neutralizing titers before vaccination to 6 months was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 6 months after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 20
Fold rise | 5.8 [2.2 to 15.0] | 6.9 [1.6 to 30.4] | 33.1 [13.7 to 79.6] | 46.9 [17.6 to 124.7] | 7.5 [2.4 to 22.8] | 12.6 [5.8 to 27.3]

87. Primary Outcome: SSF: GMFR of SARS-CoV-2 Reference-Strain-Neutralizing Titers From Before the Study Vaccination to 6 Months After Vaccination
Description: GMFR of SARS-CoV-2 reference-strain-neutralizing titers before vaccination to 6 months was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 6 months after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 20
Fold rise | 2.6 [1.1 to 6.1] | 3.6 [1.0 to 12.7] | 6.3 [2.6 to 15.2] | 12.6 [6.0 to 26.1] | 3.4 [1.3 to 8.9] | 3.9 [1.8 to 8.2]

88. Primary Outcome: SSF: GMFR of SARS-CoV-2 Omicron BA.4/BA.5 Strain-Neutralizing Titers From Before the Study Vaccination to 6 Months After Vaccination
Description: GMFR of SARS-CoV-2 Omicron BA.4/BA.5 strain-neutralizing titers before vaccination to 6 months was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From before the study vaccination to 6 months after vaccination
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 20
Fold rise | 7.5 [2.8 to 20.2] | 16.6 [4.1 to 66.8] | 32.0 [12.7 to 80.7] | 55.7 [22.2 to 140.0] | 10.2 [3.7 to 28.0] | 13.0 [5.4 to 31.4]

89. Primary Outcome: SSF: Percentage of Participants With Seroresponse to Omicron BA.1 Strain-Neutralizing Titers at Day 7
Description: Seroresponse was defined as achieving >= 4-fold rise from baseline (before the study vaccination). If the baseline measurement is below the lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse on Day 7 was reported in this outcome measure.
Time Frame: Day 7 (7 days after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 20
Percentage of participants | 52.4 [29.8 to 74.3] | 44.4 [21.5 to 69.2] | 71.4 [47.8 to 88.7] | 85.0 [62.1 to 96.8] | 55.0 [31.5 to 76.9] | 90.0 [68.3 to 98.8]

90. Primary Outcome: SSF: Percentage of Participants With Seroresponse to the Reference-Strain-Neutralizing Titers at Day 7
Description: as for outcome 89
Time Frame: Day 7 (7 days after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 20
Percentage of participants | 52.4 [29.8 to 74.3] | 55.6 [30.8 to 78.5] | 61.9 [38.4 to 81.9] | 80.0 [56.3 to 94.3] | 55.0 [31.5 to 76.9] | 80.0 [56.3 to 94.3]

91. Primary Outcome: SSF: Percentage of Participants With Seroresponse to Omicron BA.4/BA.5 Strain-Neutralizing Titers at Day 7
Description: as for outcome 89
Time Frame: Day 7 (7 days after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 16 | 21 | 20 | 20 | 21
Percentage of participants | 33.3 [14.6 to 57.0] | 43.8 [19.8 to 70.1] | 42.9 [21.8 to 66.0] | 40.0 [19.1 to 63.9] | 40.0 [19.1 to 63.9] | 61.9 [38.4 to 81.9]

92. Primary Outcome: SSF: Percentage of Participants With Seroresponse to Omicron BA.1 Strain-Neutralizing Titers at Month 1
Description: Seroresponse was defined as achieving >= 4-fold rise from baseline (before the study vaccination). If the baseline measurement is below the lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse at 1 month was reported in this outcome measure.
Time Frame: Month 1 (1 month after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 20 | 20 | 20 | 20
Percentage of participants | 85.7 [63.7 to 97.0] | 61.1 [35.7 to 82.7] | 90.0 [68.3 to 98.8] | 85.0 [62.1 to 96.8] | 90.0 [68.3 to 98.8] | 85.0 [62.1 to 96.8]

93. Primary Outcome: SSF: Percentage of Participants With Seroresponse to the Reference-Strain-Neutralizing Titers at Month 1
Description: as for outcome 92
Time Frame: Month 1 (1 month after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 20 | 20 | 20 | 20
Percentage of participants | 81.0 [58.1 to 94.6] | 61.1 [35.7 to 82.7] | 85.0 [62.1 to 96.8] | 85.0 [62.1 to 96.8] | 70.0 [45.7 to 88.1] | 75.0 [50.9 to 91.3]

94. Primary Outcome: SSF: Percentage of Participants With Seroresponse to Omicron BA.4/BA.5 Strain-Neutralizing Titers at Month 1
Description: as for outcome 92
Time Frame: Month 1 (1 month after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 21 | 20 | 20 | 20
Percentage of participants | 75.0 [50.9 to 91.3] | 61.1 [35.7 to 82.7] | 66.7 [43.0 to 85.4] | 95.0 [75.1 to 99.9] | 80.0 [56.3 to 94.3] | 85.0 [62.1 to 96.8]

95. Primary Outcome: SSF: Percentage of Participants With Seroresponse to Omicron BA.1 Strain-Neutralizing Titers at Month 3
Description: Seroresponse was defined as achieving >= 4-fold rise from baseline (before the study vaccination). If the baseline measurement is below the lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse at 3 months was reported in this outcome measure.
Time Frame: Month 3 (3 months after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 20 | 19 | 20 | 19
Percentage of participants | 65.0 [40.8 to 84.6] | 50.0 [26.0 to 74.0] | 75.0 [50.9 to 91.3] | 84.2 [60.4 to 96.6] | 70.0 [45.7 to 88.1] | 89.5 [66.9 to 98.7]

96. Primary Outcome: SSF: Percentage of Participants With Seroresponse to the Reference-Strain-Neutralizing Titers at Month 3
Description: as for outcome 95
Time Frame: Month 3 (3 months after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg: Edit Participants received a total of 30 mcg bivalent BNT162b2 (15 mcg BNT162b2 and 15 mcg BNT162b2 OMI) as a single dose intramuscularly in the deltoid muscle of the non-dominant arm.
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 20 | 19 | 20 | 19
Percentage of participants | 65.0 [40.8 to 84.6] | 55.6 [30.8 to 78.5] | 65.0 [40.8 to 84.6] | 78.9 [54.4 to 93.9] | 55.0 [31.5 to 76.9] | 63.2 [38.4 to 83.7]

97. Primary Outcome: SSF: Percentage of Participants With Seroresponse to Omicron BA.4/BA.5 Strain-Neutralizing Titers at Month 3
Description: as for outcome 95
Time Frame: Month 3 (3 months after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 20 | 18 | 21 | 19 | 19 | 21
Percentage of participants | 75.0 [50.9 to 91.3] | 61.1 [35.7 to 82.7] | 85.7 [63.7 to 97.0] | 84.2 [60.4 to 96.6] | 63.2 [38.4 to 83.7] | 85.7 [63.7 to 97.0]

98. Primary Outcome: SSF: Percentage of Participants With Seroresponse to Omicron BA.1 Strain-Neutralizing Titers at Month 6
Description: Seroresponse was defined as achieving >= 4-fold rise from baseline (before the study vaccination). If the baseline measurement is below the lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse at 6 months was reported in this outcome measure.
Time Frame: Month 6 (6 months after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 20
Percentage of participants | 42.9 [21.8 to 66.0] | 47.4 [24.4 to 71.1] | 85.7 [63.7 to 97.0] | 90.0 [68.3 to 98.8] | 65.0 [40.8 to 84.6] | 85.0 [62.1 to 96.8]

99. Primary Outcome: SSF: Percentage of Participants With Seroresponse to the Reference-Strain-Neutralizing Titers at Month 6
Description: as for outcome 98
Time Frame: Month 6 (6 months after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 20 | 20
Percentage of participants | 42.9 [21.8 to 66.0] | 42.1 [20.3 to 66.5] | 61.9 [38.4 to 81.9] | 85.0 [62.1 to 96.8] | 55.0 [31.5 to 76.9] | 50.0 [27.2 to 72.8]

100. Primary Outcome: SSF: Percentage of Participants With Seroresponse to Omicron BA.4/BA.5 Strain-Neutralizing Titers at Month 6
Description: as for outcome 98
Time Frame: Month 6 (6 months after vaccination)
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg
Number analyzed (Participants) | 21 | 18 | 21 | 20 | 20 | 20
Percentage of participants | 52.4 [29.8 to 74.3] | 50.0 [26.0 to 74.0] | 85.7 [63.7 to 97.0] | 90.0 [68.3 to 98.8] | 70.0 [45.7 to 88.1] | 75.0 [50.9 to 91.3]

101. Secondary Outcome: SSA: Occurrence of First Severe COVID-19 Infection (FDA Definition) Per 1000 Person-Years of Blinded Follow-up Without Evidence of Past SARS-CoV-2 Infection: Evaluable Efficacy Population
Description: Occurrence (number of cases) of first severe COVID-19 infection based on FDA definition after booster dose without past SARS-CoV-2 infection is reported. FDA definition: confirmed COVID-19 and presence of at least 1 of the following: 1) clinical signs at rest indicative of severe systemic illness (respiratory rate greater than or equal to [>=]30 breaths per minute, heart rate >= 125 beats per minute, oxygen saturation less than or equal to [<=]93% on room air at sea level, or Horovitz quotient <300 mmHg); 2) respiratory failure (needing high-flow oxygen, noninvasive ventilation, mechanical ventilation, or extracorporeal membrane oxygenation); 3) evidence of shock (systolic blood pressure [BP] <90 mmHg, diastolic BP <60 mmHg, or requiring vasopressors); 4) significant acute renal, hepatic, or neurologic dysfunction; 5) admission to an intensive care unit; 6) death.
Time Frame: From 7 Days after booster vaccination to end of surveillance period, total surveillance time (in 1000 person-year) for BNT162b2 was 1.105 and for Placebo was 0.951
Population: SSA evaluable efficacy population included all eligible randomized participants who received the booster vaccination as randomized and had no other important protocol deviations as determined by the clinician. HIV positive participants were excluded from this analysis. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Number of 1st severe Covid19cases/1000PY
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 4639 | 4601
Number of 1st severe Covid19cases/1000PY | 0 | 2.103
Statistical Analysis 1: Comparison: SSA: BNT162b2 30 mcg: Blinded and Open Label Period vs SSA: Placebo: Blinded Period; Test type: Other; Adjusted Surveillance Time = 100.0, 95% CI 2-sided [-358.6 to 100.0]

102. Secondary Outcome: SSA: Occurrence of First Severe COVID-19 Infection (FDA Definition) Per 1000 Person-Years of Blinded Follow-up With and Without Evidence of Past SARS-CoV-2 Infection: Evaluable Efficacy Population
Description: Occurrence (number of cases) of first severe COVID-19 infection based on FDA definition after booster dose with and without past SARS-CoV-2 infection is reported. FDA definition: confirmed COVID-19 and presence of at least 1 of the following: 1) clinical signs at rest indicative of severe systemic illness (respiratory rate >= 30 breaths per minute, heart rate >= 125 beats per minute, oxygen saturation <= 93% on room air at sea level, or Horovitz quotient <300 mm Hg); 2) respiratory failure (defined as needing high-flow oxygen, noninvasive ventilation, mechanical ventilation, or extracorporeal membrane oxygenation); 3) evidence of shock (systolic BP <90 mm Hg, diastolic BP <60 mm Hg, or requiring vasopressors); 4) significant acute renal, hepatic, or neurologic dysfunction; 5) admission to an intensive care unit; 6) death.
Time Frame: From 7 Days after booster vaccination to end of surveillance period, total surveillance time (in 1000 person-year) for BNT162b2 was 1.182 and for Placebo was 1.011
Population: Evaluable efficacy population included all eligible randomized participants who received the booster vaccination as randomized and had no other important protocol deviations as determined by the clinician. HIV positive participants were excluded from this analysis. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Number of 1st severe Covid19cases/1000PY
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 4911 | 4861
Number of 1st severe Covid19cases/1000PY | 0 | 1.978
Statistical Analysis 1: Comparison: SSA: BNT162b2 30 mcg: Blinded and Open Label Period vs SSA: Placebo: Blinded Period; 2-Sided CI for RVE is derived based on the Clopper and Pearson method adjusted for surveillance time; Test type: Other; Adjusted Surveillance Time = 100.0, 95% CI 2-sided [-355.5 to 100.0]

103. Secondary Outcome: SSA: Occurrence of First Severe COVID-19 Infection (CDC Definition) Per 1000 Person-Years of Blinded Follow-up Without Evidence of Past SARS-CoV-2 Infection
Description: Occurrence (number of cases) of first severe COVID-19 infection based on CDC definition after booster dose without past SARS-CoV-2 infection is reported. CDC definition: confirmed COVID-19 and presence of at least 1 of the following: 1) hospitalization; 2) admission to an intensive care unit; 3) intubation or mechanical ventilation; 4) death.
Time Frame: From 7 Days after booster vaccination
Population: Evaluable efficacy population included eligible randomized participants who received the booster vaccination as randomized and had no other important protocol deviations as determined by the clinician. HIV positive participants were excluded from this analysis. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Number of 1st severe Covid19cases/1000PY
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 4689 | 4664
Number of 1st severe Covid19cases/1000PY | 0 | 0

104. Secondary Outcome: SSA: Occurrence of First Severe COVID-19 Infection (CDC Definition) Per 1000 Person-Years of Blinded Follow-up With and Without Evidence of Past SARS-CoV-2 Infection
Description: Occurrence (number of cases) of first severe COVID-19 infection based on CDC definition after booster dose with and without past SARS-CoV-2 infection is reported. CDC definition: confirmed COVID-19 AND presence of at least 1 of the following: 1) hospitalization; 2) admission to an intensive care unit; 3) intubation or mechanical ventilation; 4) death.
Time Frame: From 7 Days after booster vaccination
Population: as for outcome 103
Measure: Number; unit: Number of 1st severe Covid19cases/1000PY
Arm/Group | SSA: BNT162b2 30 mcg: Blinded and Open Label Period | SSA: Placebo: Blinded Period
Number analyzed (Participants) | 4977 | 4942
Number of 1st severe Covid19cases/1000PY | 0 | 0

105. Secondary Outcome: SSC: GMTs of SARS-CoV-2 Reference-Strain Neutralizing Titers at Baseline and 7 Days After the Booster Dose
Description: GMT of SARS-CoV-2 reference-strain neutralizing titers at baseline and 7 days after the booster dose was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: At baseline and 7 days after the booster dose
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 52 | 47
Titer
  Baseline | 1846.7 [1232.1 to 2767.9] | 2230.4 [1451.8 to 3426.7]
  Day 7 | 15193.4 [12335.9 to 18712.8] | 22689.7 [18949.8 to 27167.7]

106. Secondary Outcome: SSC: GMTs of SARS-CoV-2 Omicron BA.1- Neutralizing Titers at Baseline and 7 Days After the Booster Dose
Description: GMT of SARS-CoV-2 Omicron BA.1- neutralizing titers at baseline and 7 days after the booster dose was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: At baseline and 7 days after booster dose
Population: All-available immunogenicity population included all randomized or assigned participants who received the study intervention with a valid and determinate immunogenicity result after vaccination. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'n' signifies participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 52 | 47
Titer
  Baseline | 68.2 [39.1 to 119.1] | 131.1 [68.7 to 250.7]
  Day 7: number analyzed (Participants) | 49 | 47
  Day 7 | 1356.4 [970.1 to 1896.4] | 2655.7 [2046.7 to 3445.9]

107. Secondary Outcome: SSC: GMFRs of SARS-CoV-2 Reference-Strain-Neutralizing Titers From Baseline to 7 Days After the Booster Dose
Description: GMFR of SARS-CoV-2 reference-strain-neutralizing titers from baseline (before the booster dose) to 7 days after the booster dose was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From baseline (before booster dose) to 7 days after the booster dose
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 52 | 47
Fold rise | 8.2 [5.9 to 11.5] | 10.2 [6.8 to 15.2]

108. Secondary Outcome: SSC: GMFRs of SARS-CoV-2 Omicron BA.1-Neutralizing Titers From Baseline to 7 Days After the Booster Dose
Description: GMFR of SARS-CoV-2 Omicron BA.1-strain-neutralizing titers from baseline (before the booster dose) to 7 days after the booster dose was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises from before vaccination and the corresponding CIs (based on the student's t distribution).
Time Frame: From baseline (before booster dose) to 7 days after the booster dose
Population: as for outcome 77
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 49 | 47
Fold rise | 19.7 [12.3 to 31.6] | 20.2 [11.7 to 35.0]

109. Secondary Outcome: SSC: Percentages of Participants With Seroresponse to Reference Strain at 7 Days After the Booster Dose
Description: Seroresponse was defined as achieving >= 4-fold rise from before booster dose. If the baseline measurement is below the lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse to reference strain at 7 days after the booster dose was reported in this outcome measure.
Time Frame: 7 days after the booster dose
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 52 | 47
Percentage of participants | 71.2 [56.9 to 82.9] | 68.1 [52.9 to 80.9]

110. Secondary Outcome: SSC: Percentages of Participants With Seroresponse to Omicron BA.1 at 7 Days After the Booster Dose
Description: Seroresponse was defined as achieving >= 4-fold rise from before booster dose. If the baseline measurement is below the lower limit of quantification (LLOQ), the postvaccination measure of >= 4 × LLOQ is considered a seroresponse. Exact 2-sided CI, based on the Clopper and Pearson method was used. Percentage of participants achieving seroresponse to Omicron BA.1 strain at 7 days after the booster dose was reported in this outcome measure.
Time Frame: 7 days after the booster dose
Population: as for outcome 77
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg
Number analyzed (Participants) | 49 | 47
Percentage of participants | 77.6 [63.4 to 88.2] | 74.5 [59.7 to 86.1]

111. Secondary Outcome: SSE: GMR Based on Geometric Mean Titers of SARS-CoV-2 Reference Strain Neutralizing Titers at 1 Month After the Study Vaccination- >55 Years of Age
Description: GMR based on GMT of SARS-CoV-2 reference strain neutralizing titers was calculated and reported in statistical analysis section. GMT of SARS-CoV-2 Reference strain-neutralizing titers at 1 month after the study vaccination was reported in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: 1 month after study vaccination
Population: Evaluable immunogenicity population was analyzed. Participants without evidence of prior infection were included in the analysis. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Participants were analyzed only in Expanded cohort >55 years BNT162b2 30 mcg, BNT162b2 15 mcg + BNT162b2 OMI 15 mcg and BNT162b2 30 mcg + BNT162b2 OMI 30 mcg, as pre-specified in protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg
Number analyzed (Participants) | 182 | 186 | 180
Titer | 5998.1 [5223.6 to 6887.4] | 5933.2 [5188.2 to 6785.2] | 7816.9 [6820.7 to 8958.6]
Statistical Analysis 1: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg; [analysis description as in outcome 56, analysis 3]; Test type: Other; Geometric mean ratio (GMR) = 0.99, 95% CI 2-sided [0.82 to 1.20]
Statistical Analysis 2: Comparison: SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg vs SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg; [analysis description as in outcome 56, analysis 4]; Test type: Other; Geometric mean ratio (GMR) = 1.30, 95% CI 2-sided [1.07 to 1.58]

ADVERSE EVENTS:
Time Frame: Death/SAEs: 6 months after last dose (or 1 month after each dose for SSB, or 6 months after BNT162b2 for SSA original placebo). Non-SAEs: 1 month after each booster dose (or after Dose 2 for SSD naïve group, or after BNT162b2 for SSA original placebo)
Description: Same event may appear as both AE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both AE and non-SAE. For SSB, SSC, SSE and SSF, MedDRA version used is v25.1. For SSD, MedDRA version used is v26.0.
Groups:
- SSA: BNT162b2 30 mcg- Blinded and Open Label Period; SSB: BNT162b2: Subjects received one dose (30 microgram) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
- SSA: Original Placebo/BNT162b2 (30 mcg)- Open Label Period: Subjects received placebo (normal saline solution of 0.9 percent [%] sodium chloride) intramuscularly and then one dose (30 microgram) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
- SSB: Placebo: Subjects received placebo (normal saline solution of 0.9 percent [%] sodium chloride) intramuscularly.
- SSC: BNT162b2 30 mcg: Subjects received one dose (30 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm.
- SSD: Cohort 1: Group 2a: Subjects received two doses (30 mcg) of BNT162b2 Omicron (OMI) intramuscularly 4 weeks apart in the deltoid muscle of the non-dominant arm.
- SSD: Cohort 2: Group 3a: Subjects received one dose (30 mcg) of BNT162b2 Omicron (OMI) intramuscularly in the deltoid muscle of the non-dominant arm (Vaccination 1).
- SSD: Cohort 2: Group 3 b; SSD: Cohort 2: Group 4b: After 3 months of Vaccination 1, subjects upon their consent received optional additional one dose (30 mcg) of BNT162b2 OMI (Vaccination 2).
- SSD: Cohort 2: Group 4a: Subjects received one dose (30 mcg) of BNT162b2 intramuscularly in the deltoid muscle of the non-dominant arm (Vaccination 1).
- SSD: Cohort 3: Group 5a: Subjects received two doses (30 mcg) of BNT162b2 Omicron (OMI) 3 weeks apart intramuscularly in the deltoid muscle of the non-dominant arm (Vaccination 1 and 2).
- SSD: Cohort 3: Group 5b: Subjects upon their consent received one dose (30 mcg) of BNT162b2 5 months after second dose of BNT162b2 OMI vaccination (Vaccination 3).
Arm/Group | SSA: BNT162b2 30 mcg- Blinded and Open Label Period | SSA: Placebo: Blinded Period | SSA: Original Placebo/BNT162b2 (30 mcg)- Open Label Period | SSB: BNT162b2 | SSB: Placebo | SSF: BNT162b2 30 mcg | SSF: BNT162b2 60 mcg | SSF: BNT162b2 OMI 30 mcg | SSF: BNT162b2 OMI 60 mcg | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg | SSC: BNT162b2 10 mcg | SSC: BNT162b2 30 mcg | SSD: Cohort 1: Group 1 | SSD: Cohort 1: Group 2a | SSD: Cohort 1: Group 2b | SSD: Cohort 2: Group 3a | SSD: Cohort 2: Group 3 b | SSD: Cohort 2: Group 4a | SSD: Cohort 2: Group 4b | SSD: Cohort 3: Group 5a | SSD: Cohort 3: Group 5b | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg
All-Cause Mortality (participants affected / at risk) | 5/5080 | 2/5041 | 5/4429 | 0/1453 | 0/1463 | 0/21 | 0/19 | 0/21 | 0/20 | 0/20 | 0/21 | 0/75 | 0/65 | 0/216 | 2/197 | 1/204 | 1/315 | 0/213 | 0/323 | 0/238 | 1/210 | 1/172 | 0/30 | 0/30 | 0/30 | 0/482 | 0/159 | 0/321 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 1/20 | 0/305 | 0/302 | 1/307 | 1/307 | 0/308 | 1/313
Serious Adverse Events (participants affected / at risk) | 73/5080 | 42/5041 | 45/4429 | 2/1453 | 2/1463 | 0/21 | 1/19 | 1/21 | 0/20 | 1/20 | 0/21 | 0/75 | 1/65 | 2/216 | 3/197 | 2/204 | 5/315 | 1/213 | 2/323 | 3/238 | 7/210 | 1/172 | 0/30 | 0/30 | 0/30 | 3/482 | 2/159 | 3/321 | 1/20 | 0/20 | 0/20 | 0/20 | 0/20 | 1/20 | 6/305 | 2/302 | 12/307 | 4/307 | 4/308 | 6/313
Other Adverse Events (participants affected / at risk) | 1201/5080 | 202/5041 | 771/4429 | 1180/1453 | 615/1463 | 17/21 | 19/19 | 20/21 | 18/20 | 18/20 | 20/21 | 49/75 | 57/65 | 124/216 | 131/197 | 109/204 | 260/315 | 167/213 | 270/323 | 175/238 | 135/210 | 69/172 | 29/30 | 27/30 | 29/30 | 431/482 | 143/159 | 297/321 | 15/20 | 15/20 | 15/20 | 20/20 | 16/20 | 17/20 | 220/305 | 243/302 | 241/307 | 248/307 | 226/308 | 247/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | SSA: BNT162b2 30 mcg- Blinded and Open Label Period (N=5080) | SSA: Placebo: Blinded Period (N=5041) | SSA: Original Placebo/BNT162b2 (30 mcg)- Open Label Period (N=4429) | SSB: BNT162b2 (N=1453) | SSB: Placebo (N=1463) | SSF: BNT162b2 30 mcg (N=21) | SSF: BNT162b2 60 mcg (N=19) | SSF: BNT162b2 OMI 30 mcg (N=21) | SSF: BNT162b2 OMI 60 mcg (N=20) | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg (N=20) | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg (N=21) | SSC: BNT162b2 10 mcg (N=75) | SSC: BNT162b2 30 mcg (N=65) | SSD: Cohort 1: Group 1 (N=216) | SSD: Cohort 1: Group 2a (N=197) | SSD: Cohort 1: Group 2b (N=204) | SSD: Cohort 2: Group 3a (N=315) | SSD: Cohort 2: Group 3 b (N=213) | SSD: Cohort 2: Group 4a (N=323) | SSD: Cohort 2: Group 4b (N=238) | SSD: Cohort 3: Group 5a (N=210) | SSD: Cohort 3: Group 5b (N=172) | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg (N=30) | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg (N=30) | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg (N=30) | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg (N=482) | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg (N=159) | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg (N=321) | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg (N=20) | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg (N=305) | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg (N=302) | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg (N=307) | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg (N=307) | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg (N=308) | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg (N=313)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired immunodeficiency syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/302 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/302 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penetrating aortic ulcer (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyosarcomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral myocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/64 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSA: BNT162b2 30 mcg- Blinded and Open Label Period (N=5080) | SSA: Placebo: Blinded Period (N=5041) | SSA: Original Placebo/BNT162b2 (30 mcg)- Open Label Period (N=4429) | SSB: BNT162b2 (N=1453) | SSB: Placebo (N=1463) | SSF: BNT162b2 30 mcg (N=21) | SSF: BNT162b2 60 mcg (N=19) | SSF: BNT162b2 OMI 30 mcg (N=21) | SSF: BNT162b2 OMI 60 mcg (N=20) | SSF: BNT162b2 15 mcg + BNT162b2 OMI 15 mcg (N=20) | SSF: BNT162b2 30 mcg + BNT162b2 OMI 30 mcg (N=21) | SSC: BNT162b2 10 mcg (N=75) | SSC: BNT162b2 30 mcg (N=65) | SSD: Cohort 1: Group 1 (N=216) | SSD: Cohort 1: Group 2a (N=197) | SSD: Cohort 1: Group 2b (N=204) | SSD: Cohort 2: Group 3a (N=315) | SSD: Cohort 2: Group 3 b (N=213) | SSD: Cohort 2: Group 4a (N=323) | SSD: Cohort 2: Group 4b (N=238) | SSD: Cohort 3: Group 5a (N=210) | SSD: Cohort 3: Group 5b (N=172) | SSE: Sentinel Cohort (18-55 Years): BNT 30mcg + BNT OMI 30 mcg (N=30) | SSE: Sentinel Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg (N=30) | SSE: Sentinel Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg (N=30) | SSE: Expanded Cohort (18-55 Years): BNT 30 mcg +BNT OMI 30 mcg (N=482) | SSE: Expanded Cohort (18-55 Years): BNT 15 mcg +BNT OMI 15 mcg (N=159) | SSE: Expanded Cohort (18 to 55 Years): BNT162b2 OMI 60 mcg (N=321) | SSE: Sentinel Cohort (> 55 Years): BNT162b2 30 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT162b2 60 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 30 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT162b2 OMI 60 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg (N=20) | SSE: Sentinel Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg (N=20) | SSE: Expanded Cohort (> 55 Years): BNT162b2 30 mcg (N=305) | SSE: Expanded Cohort (> 55 Years): BNT162b2 60 mcg (N=302) | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 30 mcg (N=307) | SSE: Expanded Cohort (> 55 Years): BNT162b2 OMI 60 mcg (N=307) | SSE: Expanded Cohort (> 55 Years): BNT 15 mcg + BNT OMI 15 mcg (N=308) | SSE: Expanded Cohort (> 55 Years): BNT 30 mcg +BNT OMI 30 mcg (N=313)
Lymphadenopathy (Blood and lymphatic system disorders) | 141 (147) | 3 (3) | 59 (59) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 7 (7) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 54 (54) | 16 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 243 (243) | 11 (11) | 107 (107) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 383 (383) | 66 (66) | 228 (228) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 673 (675) | 83 (83) | 412 (412) | 17 (17) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 139 (140) | 16 (16) | 122 (122) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 258 (258) | 8 (8) | 142 (143) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 248 (248) | 21 (21) | 118 (119) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 58 (58) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 267 (269) | 54 (54) | 144 (144) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 109 (109) | 77 (77) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 19 (19) | 20 (24) | 13 (13) | 25 (25) | 18 (18) | 35 (35) | 13 (13) | 20 (24) | 3 (3) | 6 (6) | 1 (1) | 4 (4) | 61 (61) | 17 (17) | 39 (39) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 13 (13) | 17 (17) | 24 (24) | 31 (31) | 26 (26) | 21 (21)
Vomiting (VOMITING) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 37 (37) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 8 (8) | 7 (7) | 8 (8) | 1 (1) | 5 (5) | 4 (4) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 15 (15) | 1 (1) | 12 (12) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 5 (5) | 9 (9) | 8 (8) | 4 (4) | 4 (4)
Chills (CHILLS) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 278 (278) | 69 (69) | 3 (3) | 3 (3) | 5 (5) | 5 (5) | 1 (1) | 3 (3) | 10 (10) | 15 (15) | 31 (31) | 35 (39) | 21 (21) | 93 (93) | 39 (39) | 80 (80) | 41 (41) | 32 (36) | 14 (14) | 7 (7) | 7 (7) | 12 (12) | 171 (171) | 44 (44) | 123 (123) | 1 (1) | 4 (4) | 3 (3) | 7 (7) | 5 (5) | 6 (6) | 49 (49) | 72 (72) | 77 (77) | 78 (78) | 38 (38) | 74 (74)
Fatigue (FATIGUE) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 723 (723) | 356 (356) | 10 (10) | 7 (7) | 9 (9) | 11 (11) | 10 (10) | 12 (12) | 37 (37) | 35 (35) | 67 (67) | 61 (79) | 57 (57) | 189 (189) | 119 (119) | 184 (184) | 117 (117) | 87 (109) | 35 (35) | 20 (20) | 19 (19) | 21 (21) | 354 (354) | 108 (108) | 248 (248) | 9 (9) | 11 (11) | 9 (9) | 13 (13) | 8 (8) | 14 (14) | 135 (135) | 156 (156) | 158 (158) | 177 (177) | 147 (147) | 177 (177)
Injection site erythema (REDNESS) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 74 (74) | 9 (9) | 4 (4) | 4 (4) | 5 (5) | 4 (4) | 2 (2) | 6 (6) | 1 (1) | 4 (4) | 7 (7) | 18 (20) | 5 (5) | 21 (21) | 10 (10) | 13 (13) | 9 (9) | 14 (16) | 7 (7) | 2 (2) | 0 (0) | 2 (2) | 39 (39) | 10 (10) | 35 (35) | 0 (0) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 19 (19) | 31 (31) | 19 (19) | 33 (33) | 22 (22) | 22 (22)
Injection site pain (PAIN) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1038 (1038) | 163 (163) | 15 (15) | 18 (18) | 19 (19) | 16 (16) | 15 (15) | 19 (19) | 42 (42) | 50 (50) | 96 (96) | 110 (145) | 85 (85) | 229 (229) | 145 (145) | 239 (239) | 153 (153) | 109 (146) | 60 (60) | 27 (27) | 25 (25) | 29 (29) | 398 (398) | 128 (128) | 276 (276) | 14 (14) | 14 (14) | 13 (13) | 20 (20) | 13 (131) | 17 (17) | 179 (179) | 212 (212) | 199 (199) | 214 (214) | 177 (177) | 208 (208)
Injection site swelling (SWELLING) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 86 (86) | 7 (7) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 6 (6) | 2 (2) | 6 (6) | 17 (17) | 23 (28) | 11 (11) | 25 (25) | 8 (8) | 27 (27) | 14 (14) | 27 (32) | 16 (16) | 0 (0) | 2 (2) | 6 (6) | 46 (46) | 11 (11) | 38 (38) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 18 (18) | 39 (39) | 25 (25) | 31 (31) | 20 (20) | 17 (17)
Pyrexia (FEVER) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 74 (74) | 17 (17) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 12 (12) | 7 (7) | 10 (10) | 25 (25) | 9 (9) | 22 (22) | 13 (13) | 11 (12) | 4 (4) | 4 (4) | 0 (0) | 3 (3) | 48 (48) | 17 (17) | 62 (62) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 4 (4) | 11 (11) | 22 (22) | 25 (25) | 27 (27) | 15 (15) | 24 (24)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 18 (18) | 26 (26) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 178 (178) | 55 (55) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 23 (23) | 33 (38) | 20 (20) | 69 (69) | 28 (28) | 46 (46) | 26 (26) | 29 (30) | 14 (14) | 6 (6) | 5 (5) | 7 (7) | 122 (122) | 33 (33) | 77 (77) | 4 (4) | 5 (5) | 3 (3) | 4 (4) | 3 (3) | 7 (7) | 27 (27) | 48 (48) | 50 (50) | 59 (59) | 34 (34) | 57 (57)
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 402 (402) | 88 (88) | 4 (4) | 8 (8) | 5 (5) | 6 (6) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 32 (32) | 41 (48) | 28 (28) | 99 (99) | 51 (51) | 86 (86) | 58 (58) | 45 (48) | 23 (23) | 9 (9) | 9 (9) | 14 (14) | 191 (191) | 58 (58) | 135 (135) | 5 (5) | 4 (4) | 5 (5) | 7 (7) | 4 (4) | 7 (7) | 59 (59) | 76 (76) | 72 (72) | 92 (92) | 70 (70) | 82 (82)
Headache (HEADACHE) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 585 (585) | 332 (332) | 6 (6) | 5 (5) | 5 (5) | 11 (11) | 7 (7) | 8 (8) | 31 (31) | 34 (34) | 64 (64) | 70 (89) | 55 (55) | 140 (140) | 78 (78) | 137 (137) | 81 (81) | 67 (77) | 39 (39) | 14 (14) | 9 (9) | 18 (18) | 257 (257) | 79 (79) | 184 (184) | 4 (4) | 6 (6) | 7 (7) | 3 (3) | 6 (6) | 10 (10) | 79 (79) | 116 (116) | 110 (110) | 110 (110) | 99 (99) | 114 (114)
Eye pruritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infections (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit-hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (7):
  • Study Protocol (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04955626/Prot_000.pdf
  • Statistical Analysis Plan: substudy A (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT04955626/SAP_001.pdf
  • Statistical Analysis Plan: substudy B (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT04955626/SAP_002.pdf
  • Statistical Analysis Plan: substudy C (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT04955626/SAP_003.pdf
  • Statistical Analysis Plan: substudy D (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04955626/SAP_004.pdf
  • Statistical Analysis Plan: substudy E (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04955626/SAP_005.pdf
  • Statistical Analysis Plan: substudy F (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04955626/SAP_006.pdf